CLINICAL TRIAL: NCT00583362
Title: A Multi-Center, Open-Label, Continuation Trial LymphoStat-B™ Antibody (Monoclonal Anti-BLyS Antibody) in Subjects With Systemic Lupus Erythematosus (SLE) Who Completed the Phase 2 Protocol LBSL02
Brief Title: A Continuation Trial for Subjects With Systemic Lupus Erythematosus That Have Completed Protocol LBSL02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112626
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belimumab 10 mg/kg (Experimental): Belimumab 10 mg/kg IV over one hour every 28 days.
  Interventions: Biological: Belimumab

INTERVENTIONS:
Biological: Belimumab — Belimumab 10mg/kg IV over one hour every 28 days
  Other Names: LymphoStat-B™; HGS1006; BENLYSTA

SUMMARY:
This is a continuation study to evaluate the long-term safety and efficacy of LymphoStat-B™ in subjects with SLE disease, that completed study LBSL02 and benefitted from treatment.

DETAILED DESCRIPTION:
The purpose of this continuation study to evaluate the long-term safety and efficacy of LymphoStat-B™ in subjects with Systemic Lupus Erythematosus (SLE), that completed study LBSL02 and benefitted from treatment.

ELIGIBILITY:
Primary Inclusion Criteria

1. Have completed the LBSL02 trial and achieved a satisfactory response.

Primary Exclusion Criteria

1. Required more than 2 courses of corticosteroids for treatment of severe SLE flares in the last 5 months of LBSL02.
2. Had an SLE flare during the last 30 days of LBSL02 and through the 1st dose in LBSL99.
3. Used any of the following prohibited medications during their participation in LBSL02:

   * Other investigational agents.
   * Biologic therapeutic agents: adalimumab (Humira™), etanercept (Enbrel™), infliximab (Remicade™), and rituximab (Rituxan™).
   * Intravenous cyclophosphamide.
   * Corticosteroids >100 mg/day prednisone equivalent for reasons other than severe SLE flare.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2005-05-04 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (52):
- United States (51):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Munster, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Cumberland, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Concord, New Hampshire
  - GSK Investigational Site, Dover, New Hampshire
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Willow Grove, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Onalaska, Wisconsin
- GSK Investigational Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=bel112626

REFERENCES:
- [Derived] Ginzler EM, Wallace DJ, Merrill JT, Furie RA, Stohl W, Chatham WW, Weinstein A, McKay JD, McCune WJ, Zhong ZJ, Freimuth WW, Petri MA; LBSL02/99 Study Group. Disease control and safety of belimumab plus standard therapy over 7 years in patients with systemic lupus erythematosus. J Rheumatol. 2014 Feb;41(2):300-9. doi: 10.3899/jrheum.121368. Epub 2013 Nov 1. PMID 24187095
- [Derived] Merrill JT, Ginzler EM, Wallace DJ, McKay JD, Lisse JR, Aranow C, Wellborne FR, Burnette M, Condemi J, Zhong ZJ, Pineda L, Klein J, Freimuth WW; LBSL02/99 Study Group. Long-term safety profile of belimumab plus standard therapy in patients with systemic lupus erythematosus. Arthritis Rheum. 2012 Oct;64(10):3364-73. doi: 10.1002/art.34564. PMID 22674457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the parent study LBSL02 (NCT00071487) through the 24-week extension period, who received belimumab 1 milligram (mg)/kilogram (kg), 4 mg/kg, 10 mg/kg or placebo in the parent study and achieved a satisfactory response were enrolled in the study.
Groups:
- Belimumab 10 mg/kg IV: Participants received 10 mg/kg of belimumab every 28 days as an intravenous (IV) infusion over a period of 1 to 2 hours. The first dose of belimumab was given 4 weeks after the last (Day 532) dose in LBSL02. Treatment continued for 10 years from the time the last participant was enrolled in the present study or until there were 100 or fewer participants continuing in the study, whichever came first. All participants received standard of care for systemic lupus erythematosus (SLE) during study participation.
Period: Overall Study
Arm/Group | Belimumab 10 mg/kg IV
Started | 298
Completed | 96
Not Completed | 202
Not completed — Adverse Event | 44
Not completed — Lack of Efficacy | 22
Not completed — Lost to Follow-up | 4
Not completed — Non-compliance with study drug | 28
Not completed — Pregnancy | 7
Not completed — Miscommunication of visit window | 5
Not completed — Current site closed | 7
Not completed — Subject not dosed in LBSL99 | 1
Not completed — Subject moved out of the country/state | 2
Not completed — Missed visits due to staff changes | 1
Not completed — Misunderstanding of protocol | 1
Not completed — Behavioral problems and non-compliance | 1
Not completed — Sponsor request due to missed doses | 1
Not completed — Physician Decision | 19
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 57

BASELINE CHARACTERISTICS:
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] — Modified Intent to Treat (MITT) Population: All participants who were enrolled in the study and were treated with at least one dose of belimumab in the study.
  Years | 43 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants] — MITT Population
  Participants
    Female | 276
    Male | 20
Race/Ethnicity, Customized [Number; unit: Participants] — MITT Population
  Participants
    American Indian or Alaska Native | 6
    Asian | 6
    Black or African American | 68
    Native Hawaiian or Other Pacific Islander | 1
    White | 215

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Type of Adverse Event (AEs) and Serious Adverse Event (SAEs)
Description: An AE is defined as any unfavorable or unintended sign, symptom, or disease that is temporally associated with the use of a study agent but is not necessarily caused by the study agent. This includes worsening (example [eg], increase in frequency or severity) of pre-existing conditions. An SAE is defined as an AE resulting in any of the following outcomes: death, is life threatening (that is, an immediate threat to life), inpatient hospitalization, prolongation of an existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, and is medically important.
Time Frame: Approximately up to 13 years
Population: MITT Population. Only those participants available at the specified time points (represented by n=X, in the category titles) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Participants
  AE, Any time post baseline, n=296 | 294
  AE, Year 0-1, n=296 | 291
  AE, Year 1-2, n=294 | 283
  AE, Year 2-3, n=276 | 260
  AE, Year 3-4, n=250 | 239
  AE, Year 4-5, n=223 | 203
  AE, Year 5-6, n=209 | 190
  AE, Year 6-7, n=192 | 182
  AE, Year 7-8, n=178 | 162
  AE, Year 8-9, n=169 | 157
  AE, Year 9-10, n=152 | 137
  AE, Year 10-11, n=131 | 105
  AE, Year 11 plus, n=88 | 45
  SAE, Any time post baseline, n=296 | 182
  SAE, Year 0-1, n=296 | 41
  SAE, Year 1-2, n=294 | 43
  SAE, Year 2-3, n=276 | 50
  SAE, Year 3-4, n=250 | 30
  SAE, Year 4-5, n=223 | 40
  SAE, Year 5-6, n=209 | 33
  SAE, Year 6-7, n=192 | 35
  SAE, Year 7-8, n=178 | 34
  SAE, Year 8-9, n=169 | 28
  SAE, Year 9-10, n=152 | 25
  SAE, Year 10-11, n=131 | 14
  SAE, Year 11 plus, n=88 | 7

2. Primary Outcome: Adverse Event (AE) Rates by System Organ Class (SOC) During the Study
Description: AE rates by SOC adjusting for participant-years on study drug anytime post Baseline are summarized, which included the follow up visits. Only treatmentemergent AEs are summarized. The Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. The event rate of an AE was calculated as the number of events per 100 participant years: Event Rate=100* number of events divided by participant years. Participant years were calculated as sum across all participants ([last visit of interval day minus first visit of interval day plus 1] divided by 365).
Time Frame: Approximately up to 13 years
Population: MITT Population
Measure: Number; unit: Events per 100 participant years
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Events per 100 participant years
  Infections and infestations | 285
  Musculoskeletal and connective tissue disorders | 276
  Gastrointestinal disorders | 257
  Skin and subcutaneous tissue disorders | 256
  General disorders, administration site conditions | 247
  Nervous system disorders | 244
  Respiratory, thoracic and mediastinal disorders | 241
  Investigations | 227
  Injury, poisoning and procedural complications | 221
  Psychiatric disorders | 180
  Metabolism and nutrition disorders | 144
  Vascular disorders | 134
  Eye disorders | 133
  Blood and lymphatic system disorders | 127
  Reproductive system and breast disorders | 114
  Renal and urinary disorders | 109
  Immune system disorders | 101
  Neoplasms benign, malignant and unspecified | 100
  Cardiac disorders | 86
  Ear and labyrinth disorders | 69
  Endocrine disorders | 40
  Hepatobiliary disorders | 27
  Social circumstances | 15
  Congenital, familial and genetic disorders | 7
  Pregnancy, puerperium and perinatal conditions | 5

3. Primary Outcome: SAE Rates by System Organ Class (SOC) During the Study
Description: SAE rates by SOC adjusting for participant-years on study drug anytime post Baseline are summarized, which included the follow up visits. Only treatmentemergent SAEs are summarized. The Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pretreatment value in the parent study for participants treated with belimumab in the parent study. The event rate of an SAE was calculated as the number of events per 100 participant years: Event Rate=100* number of events divided by participant years. Participant years were calculated as sum across all participants ([last visit of interval day minus first visit of interval day plus 1] divided by 365).
Time Frame: Approximately up to 13 years
Population: MITT population
Measure: Number; unit: Events per 100 participant years
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Events per 100 participant years
  Infections and infestations | 69
  Musculoskeletal and connective tissue disorders | 44
  Gastrointestinal disorders | 38
  Nervous system disorders | 35
  General disorders, administration site conditions | 31
  Injury, poisoning and procedural complications | 29
  Respiratory, thoracic and mediastinal disorders | 25
  Cardiac disorders | 23
  Neoplasms benign, malignant and unspecified | 23
  Renal and urinary disorders | 20
  Vascular disorders | 19
  Reproductive system and breast disorders | 18
  Metabolism and nutrition disorders | 14
  Hepatobiliary disorders | 10
  Blood and lymphatic system disorders | 8
  Skin and subcutaneous tissue disorders | 8
  Investigations | 7
  Psychiatric disorders | 6
  Immune system disorders | 2
  Pregnancy, puerperium and perinatal conditions | 2
  Congenital, familial and genetic disorders | 1
  Eye disorders | 1
  Social circumstances | 1

4. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (APTT) and Prothrombin Time (PT) at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 8, 16, 24, 40, and 48 during Year 1 to 8; Week 8, 16, 24, and 40 during Year 9; Week 24 and 40 during Year 10; Week 48 during Year 11; Week 32 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in APTT and PT is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: MITT Population. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Seconds
  APTT, Year 1, Week 8, n=274 | 0.3 (12.60)
  APTT, Year 1, Week 16, n=276 | -1.3 (7.46)
  APTT, Year 1, Week 24, n=222 | -1.6 (13.61)
  APTT, Year 1, Week 32, n=221 | -1.9 (7.24)
  APTT, Year 1, Week 40, n=219 | -1.6 (7.00)
  APTT, Year 1, Week 48, n=218 | -1.0 (7.29)
  APTT, Year 2, Week 8, n=220 | -0.3 (6.73)
  APTT, Year 2, Week 16, n=214 | -0.2 (8.79)
  APTT, Year 2, Week 24, n=212 | 0.6 (13.81)
  APTT, Year 2, Week 32, n=35 | 1.5 (9.20)
  APTT, Year 2, Week 40, n=28 | 2.6 (7.53)
  APTT, Year 2, Week 48, n=21 | 3.0 (8.69)
  APTT, Year 3, Week 8, n=25 | 2.4 (10.70)
  APTT, Year 3, Week 16, n=23 | 2.3 (7.77)
  APTT, Year 3, Week 24, n=23 | 1.7 (6.30)
  APTT, Year 3, Week 32, n=22 | 5.4 (10.01)
  APTT, Year 3, Week 40, n=18 | 2.1 (9.62)
  APTT, Year 3, Week 48, n=18 | 3.9 (17.23)
  APTT, Year 4, Week 8, n=14 | 2.9 (11.42)
  APTT, Year 4, Week 16, n=16 | 3.1 (8.97)
  APTT, Year 4, Week 24, n=10 | 1.1 (10.29)
  APTT, Year 4, Week 32, n=18 | 2.1 (11.37)
  APTT, Year 4, Week 40, n=13 | -2.1 (10.02)
  APTT, Year 4, Week 48, n=11 | 2.2 (11.83)
  APTT, Year 5, Week 8, n=4 | 3.0 (14.76)
  APTT, Year 5, Week 16, n=11 | 1.3 (5.62)
  APTT, Year 5, Week 24, n=3 | 13.0 (11.53)
  APTT, Year 5, Week 32, n=12 | 3.1 (6.64)
  APTT, Year 5, Week 40, n=10 | -0.5 (8.03)
  APTT, Year 5, Week 48, n=3 | 12.3 (5.51)
  APTT, Year 6, Week 8, n=3 | -2.3 (19.50)
  APTT, Year 6, Week 16, n=3 | 9.0 (12.12)
  APTT, Year 6, Week 24, n=3 | 14.0 (16.52)
  APTT, Year 6, Week 32, n=2 | 6.5 (17.68)
  APTT, Year 6, Week 40, n=8 | 9.9 (9.11)
  APTT, Year 6, Week 48, n=4 | 18.3 (4.99)
  APTT, Year 7, Week 8, n=1 | 27.0 (NA) — No value as only one participant was analyzed.
  APTT, Year 7, Week 16, n=2 | 24.5 (14.85)
  APTT, Year 7, Week 24, n=2 | 19.5 (6.36)
  APTT, Year 7, Week 32, n=1 | 7.0 (NA) — No value as only one participant was analyzed.
  APTT, Year 7, Week 40, n=2 | 16.5 (16.26)
  APTT, Year 7, Week 48, n=2 | 18.5 (2.12)
  APTT, Year 8, Week 8, n=3 | 11.7 (18.04)
  APTT, Year 8, Week 16, n=3 | 15.7 (10.07)
  APTT, Year 8, Week 24, n=3 | 21.3 (22.50)
  APTT, Year 8, Week 32, n=3 | 8.7 (14.36)
  APTT, Year 8, Week 40, n=2 | 25.0 (5.66)
  APTT, Year 8, Week 48, n=3 | 13.3 (15.01)
  APTT, Year 9, Week 8, n=3 | 10.3 (9.07)
  APTT, Year 9, Week 16, n=3 | 11.0 (9.85)
  APTT, Year 9, Week 24, n=2 | 24.0 (25.46)
  APTT, Year 9, Week 32, n=4 | -11.0 (21.91)
  APTT, Year 9, Week 40, n=1 | 20.0 (NA) — No value as only one participant was analyzed
  APTT, Year 10, Week 24, n=1 | 10.0 (NA) — No value as only one participant was analyzed
  APTT, Year 10, Week 40, n=1 | -9 (NA) — No value as only one participant was analyzed
  APTT, Year 11, Week 48, n=1 | -27.0 (NA) — No value as only one participant was analyzed
  APTT, Year 13, Week 32, n=1 | 26 (NA) — No value as only one participant was analyzed
  APTT, Exit, n=10 | 2.3 (9.66)
  APTT, 8-Week Follow-up, n=6 | 3.8 (6.24)
  APTT, 24-Week Follow-up, n=3 | -12.3 (16.56)
  PT, Year 1, Week 8, n=278 | -0.67 (12.222)
  PT, Year 1, Week 16, n=276 | -0.98 (12.134)
  PT, Year 1, Week 24, n=222 | -1.00 (13.859)
  PT, Year 1, Week 32, n=223 | -0.89 (13.887)
  PT, Year 1, Week 40, n=221 | -0.67 (14.262)
  PT, Year 1, Week 48, n=219 | -0.95 (13.496)
  PT, Year 2, Week 8, n=221 | -0.87 (13.364)
  PT, Year 2, Week 16, n=215 | -0.84 (13.682)
  PT, Year 2, Week 24, n=214 | -0.66 (14.156)
  PT, Year 2, Week 32, n=35 | 0.85 (6.887)
  PT, Year 2, Week 40, n=28 | 3.28 (11.046)
  PT, Year 2, Week 48, n=22 | 1.75 (8.747)
  PT, Year 3, Week 8, n=25 | 1.75 (12.409)
  PT, Year 3, Week 16, n=23 | 0.39 (5.469)
  PT, Year 3, Week 24, n=23 | 0.98 (3.120)
  PT, Year 3, Week 32, n=22 | 4.29 (10.640)
  PT, Year 3, Week 40, n=18 | 2.02 (8.833)
  PT, Year 3, Week 48, n=18 | 3.23 (15.863)
  PT, Year 4, Week 8, n=14 | 4.14 (9.948)
  PT, Year 4, Week 16, n=16 | 0.69 (8.188)
  PT, Year 4, Week 24, n=10 | 2.10 (8.506)
  PT, Year 4, Week 32, n=18 | 1.87 (11.251)
  PT, Year 4, Week 40, n=13 | -2.70 (6.698)
  PT, Year 4, Week 48, n=11 | 0.60 (9.651)
  PT, Year 5, Week 8, n=4 | -0.43 (12.189)
  PT, Year 5, Week 16, n=11 | 2.52 (6.118)
  PT, Year 5, Week 24, n=3 | 9.90 (8.347)
  PT, Year 5, Week 32, n=12 | 0.67 (3.731)
  PT, Year 5, Week 40, n=10 | -0.33 (5.443)
  PT, Year 5, Week 48, n=3 | 13.23 (9.064)
  PT, Year 6, Week 8, n=3 | -2.93 (7.859)
  PT, Year 6, Week 16, n=3 | 2.10 (5.336)
  PT, Year 6, Week 24, n=3 | 7.60 (11.623)
  PT, Year 6, Week 32, n=2 | 4.55 (21.425)
  PT, Year 6, Week 40, n=8 | 2.30 (5.865)
  PT, Year 6, Week 48, n=4 | 6.18 (10.637)
  PT, Year 7, Week 8, n=1 | 19.90 (NA) — No value as only one participant was analyzed
  PT, Year 7, Week 16, n=2 | 18.20 (14.425)
  PT, Year 7, Week 24, n=2 | 7.35 (0.636)
  PT, Year 7, Week 32, n=1 | 4.00 (NA) — No value as only one participant was analyzed
  PT, Year 7, Week 40, n=2 | 11.15 (19.587)
  PT, Year 7, Week 48, n=2 | 11.50 (4.808)
  PT, Year 8, Week 8, n=3 | 12.47 (15.546)
  PT, Year 8, Week 16, n=3 | 7.57 (6.799)
  PT, Year 8, Week 24, n=3 | 12.87 (13.787)
  PT, Year 8, Week 32, n=3 | 5.63 (9.850)
  PT, Year 8, Week 40, n=2 | 26.60 (13.435)
  PT, Year 8, Week 48, n=3 | 11.07 (9.845)
  PT, Year 9, Week 8, n=3 | 8.23 (7.976)
  PT, Year 9, Week 16, n=3 | 4.60 (6.773)
  PT, Year 9, Week 24, n=2 | 25.75 (36.416)
  PT, Year 9, Week 32, n=4 | -10.08 (8.139)
  PT, Year 9, Week 40, n=1 | 21.40 (NA) — No value as only one participant was analyzed
  PT, Year 10, Week 24, n=1 | 1.30 (NA) — No value as only one participant was analyzed
  PT, Year 10, Week 40, n=1 | -8.00 (NA) — No value as only one participant was analyzed
  PT, Year 11, Week 48, n=1 | -22.80 (NA) — No value as only one participant was analyzed
  PT, Year 13, Week 32, n=1 | 14.80 (NA) — No value as only one participant was analyzed
  PT, Exit, n=10 | 0.64 (5.559)
  PT, 8-Week Follow-up, n=6 | -0.95 (4.561)
  PT, 24-Week Follow-up, n=3 | -10.23 (11.657)

5. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils Segmented and Platelets at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in basophils, eosinophils, lymphocytes, monocytes, neutrophils segmented and platelets is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9 per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
10^9 per liter
  Basophils, Year 1, Week 8, n=287 | 0.001 (0.0163)
  Basophils, Year 1, Week 16, n=288 | 0.000 (0.0181)
  Basophils, Year 1, Week 24, n=293 | 0.000 (0.0171)
  Basophils, Year 1, Week 32, n=290 | 0.002 (0.0166)
  Basophils, Year 1, Week 40, n=287 | 0.001 (0.0159)
  Basophils, Year 1, Week 48, n=287 | 0.001 (0.0178)
  Basophils, Year 2, Week 8, n=288 | 0.001 (0.0164)
  Basophils, Year 2, Week 16, n=279 | 0.002 (0.0172)
  Basophils, Year 2, Week 24, n=276 | 0.001 (0.0168)
  Basophils, Year 2, Week 32, n=281 | 0.003 (0.0179)
  Basophils, Year 2, Week 40, n=262 | 0.002 (0.0162)
  Basophils, Year 2, Week 48, n=260 | 0.003 (0.0174)
  Basophils, Year 3, Week 8, n=260 | 0.003 (0.0167)
  Basophils, Year 3, Week 16, n=258 | 0.004 (0.0177)
  Basophils, Year 3, Week 24, n=242 | 0.002 (0.0160)
  Basophils, Year 3, Week 32, n=248 | 0.004 (0.0204)
  Basophils, Year 3, Week 40, n=242 | 0.004 (0.0178)
  Basophils, Year 3, Week 48, n=240 | 0.002 (0.0172)
  Basophils, Year 4, Week 8, n=234 | 0.001 (0.0189)
  Basophils, Year 4, Week 16, n=238 | 0.003 (0.0183)
  Basophils, Year 4, Week 24, n=227 | 0.003 (0.0160)
  Basophils, Year 4, Week 32, n=229 | 0.003 (0.0174)
  Basophils, Year 4, Week 40, n=216 | 0.004 (0.0174)
  Basophils, Year 4, Week 48, n=220 | 0.002 (0.0181)
  Basophils, Year 5, Week 8, n=215 | 0.004 (0.0173)
  Basophils, Year 5, Week 16, n=214 | 0.003 (0.0182)
  Basophils, Year 5, Week 24, n=207 | 0.003 (0.0174)
  Basophils, Year 5, Week 32, n=207 | 0.002 (0.0159)
  Basophils, Year 5, Week 40, n=196 | 0.003 (0.0184)
  Basophils, Year 5, Week 48, n=209 | 0.004 (0.0177)
  Basophils, Year 6, Week 8, n=206 | 0.004 (0.0183)
  Basophils, Year 6, Week 16, n=195 | 0.004 (0.0203)
  Basophils, Year 6, Week 24, n=192 | 0.003 (0.0212)
  Basophils, Year 6, Week 32, n=197 | 0.004 (0.0177)
  Basophils, Year 6, Week 40, n=183 | 0.003 (0.0157)
  Basophils, Year 6, Week 48, n=188 | 0.002 (0.0174)
  Basophils, Year 7, Week 8, n=180 | 0.002 (0.0194)
  Basophils, Year 7, Week 16, n=181 | 0.001 (0.0186)
  Basophils, Year 7, Week 24, n=176 | 0.003 (0.0178)
  Basophils, Year 7, Week 32, n=179 | 0.004 (0.0173)
  Basophils, Year 7, Week 40, n=177 | 0.004 (0.0172)
  Basophils, Year 7, Week 48, n=173 | 0.004 (0.0171)
  Basophils, Year 8, Week 8, n=172 | 0.003 (0.0184)
  Basophils, Year 8, Week 16, n=173 | 0.005 (0.0167)
  Basophils, Year 8, Week 24, n=170 | 0.005 (0.0160)
  Basophils, Year 8, Week 32, n=169 | 0.003 (0.0165)
  Basophils, Year 8, Week 40, n=162 | 0.005 (0.0177)
  Basophils, Year 8, Week 48, n=161 | 0.004 (0.0187)
  Basophils, Year 9, Week 8, n=164 | 0.006 (0.0227)
  Basophils, Year 9, Week 16, n=161 | 0.005 (0.0194)
  Basophils, Year 9, Week 24, n=163 | 0.004 (0.0170)
  Basophils, Year 9, Week 32, n=159 | 0.004 (0.0167)
  Basophils, Year 9, Week 40, n=156 | 0.004 (0.0180)
  Basophils, Year 9, Week 48, n=151 | 0.003 (0.0153)
  Basophils, Year 10, Week 8, n=149 | 0.002 (0.0183)
  Basophils, Year 10, Week 16, n=145 | 0.006 (0.0205)
  Basophils, Year 10, Week 24, n=147 | 0.003 (0.0186)
  Basophils, Year 10, Week 32, n=142 | 0.005 (0.0214)
  Basophils, Year 10, Week 40, n=137 | 0.004 (0.0192)
  Basophils, Year 10, Week 48, n=137 | 0.006 (0.0185)
  Basophils, Year 11, Week 8, n=137 | 0.004 (0.0200)
  Basophils, Year 11, Week 16, n=130 | 0.004 (0.0188)
  Basophils, Year 11, Week 24, n=130 | 0.005 (0.0176)
  Basophils, Year 11, Week 32, n=128 | 0.006 (0.0187)
  Basophils, Year 11, Week 40, n=122 | 0.006 (0.0232)
  Basophils, Year 11, Week 48, n=106 | 0.005 (0.0189)
  Basophils, Year 12, Week 8, n=109 | 0.007 (0.0209)
  Basophils, Year 12, Week 16, n=97 | 0.004 (0.0197)
  Basophils, Year 12, Week 24, n=86 | 0.007 (0.0204)
  Basophils, Year 12, Week 32, n=88 | 0.004 (0.0213)
  Basophils, Year 12, Week 40, n=83 | 0.007 (0.0201)
  Basophils, Year 12, Week 48, n=72 | 0.006 (0.0172)
  Basophils, Year 13, Week 8, n=53 | 0.005 (0.0173)
  Basophils, Year 13, Week 16, n=42 | 0.006 (0.0178)
  Basophils, Year 13, Week 24, n=20 | 0.008 (0.0170)
  Basophils, Year 13, Week 32, n=7 | 0.014 (0.0151)
  Basophils, Year 13, Week 40, n=1 | 0.020 (NA) — No value as only one participant was analyzed
  Basophils, Exit, n=241 | 0.005 (0.0171)
  Basophils, 8-Week Follow-up, n=219 | 0.006 (0.0205)
  Basophils, 24-Week Follow-up, n=198 | 0.006 (0.0213)
  Eosinophils, Year 1, Week 8, n=287 | 0.003 (0.0999)
  Eosinophils, Year 1, Week 16, n=288 | 0.007 (0.1213)
  Eosinophils, Year 1, Week 24, n=293 | 0.008 (0.1222)
  Eosinophils, Year 1, Week 32, n=290 | 0.011 (0.1219)
  Eosinophils, Year 1, Week 40, n=287 | 0.007 (0.1070)
  Eosinophils, Year 1, Week 48, n=287 | 0.006 (0.1130)
  Eosinophils, Year 2, Week 8, n=288 | 0.003 (0.1135)
  Eosinophils, Year 2, Week 16, n=279 | 0.034 (0.1312)
  Eosinophils, Year 2, Week 24, n=276 | 0.023 (0.1375)
  Eosinophils, Year 2, Week 32, n=281 | 0.028 (0.1423)
  Eosinophils, Year 2, Week 40, n=262 | 0.028 (0.1280)
  Eosinophils, Year 2, Week 48, n=260 | 0.042 (0.1635)
  Eosinophils, Year 3, Week 8, n=260 | 0.033 (0.1353)
  Eosinophils, Year 3, Week 16, n=258 | 0.038 (0.1391)
  Eosinophils, Year 3, Week 24, n=242 | 0.038 (0.1610)
  Eosinophils, Year 3, Week 32, n=248 | 0.029 (0.1427)
  Eosinophils, Year 3, Week 40, n=242 | 0.035 (0.1539)
  Eosinophils, Year 3, Week 48, n=240 | 0.033 (0.1369)
  Eosinophils, Year 4, Week 8, n=234 | 0.035 (0.1331)
  Eosinophils, Year 4, Week 16, n=238 | 0.034 (0.1273)
  Eosinophils, Year 4, Week 24, n=227 | 0.033 (0.1384)
  Eosinophils, Year 4, Week 32, n=229 | 0.039 (0.1381)
  Eosinophils, Year 4, Week 40, n=216 | 0.038 (0.1284)
  Eosinophils, Year 4, Week 48, n=220 | 0.030 (0.1261)
  Eosinophils, Year 5, Week 8, n=215 | 0.035 (0.1242)
  Eosinophils, Year 5, Week 16, n=214 | 0.019 (0.1294)
  Eosinophils, Year 5, Week 24, n=207 | 0.023 (0.1078)
  Eosinophils, Year 5, Week 32, n=207 | 0.027 (0.1201)
  Eosinophils, Year 5, Week 40, n=196 | 0.019 (0.1224)
  Eosinophils, Year 5, Week 48, n=209 | 0.022 (0.1224)
  Eosinophils, Year 6, Week 8, n=206 | 0.020 (0.1288)
  Eosinophils, Year 6, Week 16, n=195 | 0.021 (0.1103)
  Eosinophils, Year 6, Week 24, n=192 | 0.034 (0.1335)
  Eosinophils, Year 6, Week 32, n=197 | 0.026 (0.1171)
  Eosinophils, Year 6, Week 40, n=183 | 0.044 (0.1580)
  Eosinophils, Year 6, Week 48, n=188 | 0.026 (0.1299)
  Eosinophils, Year 7, Week 8, n=180 | 0.021 (0.1317)
  Eosinophils, Year 7, Week 16, n=181 | 0.015 (0.1170)
  Eosinophils, Year 7, Week 24, n=176 | 0.014 (0.1239)
  Eosinophils, Year 7, Week 32, n=179 | 0.010 (0.1149)
  Eosinophils, Year 7, Week 40, n=177 | 0.009 (0.1167)
  Eosinophils, Year 7, Week 48, n=173 | -0.008 (0.1176)
  Eosinophils, Year 8, Week 8, n=172 | -0.003 (0.1389)
  Eosinophils, Year 8, Week 16, n=173 | -0.009 (0.1234)
  Eosinophils, Year 8, Week 24, n=170 | -0.007 (0.1309)
  Eosinophils, Year 8, Week 32, n=169 | -0.023 (0.1136)
  Eosinophils, Year 8, Week 40, n=162 | -0.009 (0.1263)
  Eosinophils, Year 8, Week 48, n=161 | -0.011 (0.1341)
  Eosinophils, Year 9, Week 8, n=164 | -0.004 (0.1373)
  Eosinophils, Year 9, Week 16, n=161 | -0.020 (0.1204)
  Eosinophils, Year 9, Week 24, n=163 | -0.020 (0.1134)
  Eosinophils, Year 9, Week 32, n=159 | -0.012 (0.1154)
  Eosinophils, Year 9, Week 40, n=156 | -0.029 (0.1200)
  Eosinophils, Year 9, Week 48, n=151 | -0.018 (0.1307)
  Eosinophils, Year 10, Week 8, n=149 | -0.020 (0.1343)
  Eosinophils, Year 10, Week 16, n=145 | -0.010 (0.1438)
  Eosinophils, Year 10, Week 24, n=147 | -0.019 (0.1237)
  Eosinophils, Year 10, Week 32, n=142 | -0.002 (0.1332)
  Eosinophils, Year 10, Week 40, n=137 | -0.021 (0.1184)
  Eosinophils, Year 10, Week 48, n=137 | -0.021 (0.1274)
  Eosinophils, Year 11, Week 8, n=137 | -0.018 (0.1167)
  Eosinophils, Year 11, Week 16, n=130 | -0.004 (0.1336)
  Eosinophils, Year 11, Week 24, n=130 | 0.004 (0.1445)
  Eosinophils, Year 11, Week 32, n=128 | 0.003 (0.1360)
  Eosinophils, Year 11, Week 40, n=122 | -0.013 (0.1298)
  Eosinophils, Year 11, Week 48, n=106 | -0.021 (0.1435)
  Eosinophils, Year 12, Week 8, n=109 | -0.021 (0.1242)
  Eosinophils, Year 12, Week 16, n=97 | -0.020 (0.1349)
  Eosinophils, Year 12, Week 24, n=86 | -0.000 (0.1535)
  Eosinophils, Year 12, Week 32, n=88 | -0.008 (0.1356)
  Eosinophils, Year 12, Week 40, n=83 | -0.020 (0.1242)
  Eosinophils, Year 12, Week 48, n=72 | -0.016 (0.1319)
  Eosinophils, Year 13, Week 8, n=53 | -0.001 (0.1436)
  Eosinophils, Year 13, Week 16, n=42 | -0.009 (0.1244)
  Eosinophils, Year 13, Week 24, n=20 | 0.035 (0.1810)
  Eosinophils, Year 13, Week 32, n=7 | 0.081 (0.0722)
  Eosinophils, Year 13, Week 40, n=1 | 0.080 (NA) — No value as only one participant was analyzed
  Eosinophils, Exit, n=241 | 0.006 (0.1430)
  Eosinophils, 8-Week Follow-up, n=219 | -0.002 (0.1436)
  Eosinophils, 24-Week Follow-up, n=198 | 0.013 (0.2255)
  Lymphocytes, Year 1, Week 8, n=287 | 0.006 (0.4143)
  Lymphocytes, Year 1, Week 16, n=288 | -0.046 (0.4612)
  Lymphocytes, Year 1, Week 24, n=293 | -0.035 (0.4725)
  Lymphocytes, Year 1, Week 32, n=290 | -0.057 (0.4425)
  Lymphocytes, Year 1, Week 40, n=287 | -0.074 (0.5084)
  Lymphocytes, Year 1, Week 48, n=287 | -0.075 (0.4832)
  Lymphocytes, Year 2, Week 8, n=288 | -0.049 (0.4324)
  Lymphocytes, Year 2, Week 16, n=279 | -0.025 (0.4774)
  Lymphocytes, Year 2, Week 24, n=276 | -0.053 (0.4949)
  Lymphocytes, Year 2, Week 32, n=281 | -0.038 (0.5080)
  Lymphocytes, Year 2, Week 40, n=262 | -0.025 (0.5046)
  Lymphocytes, Year 2, Week 48, n=260 | 0.006 (0.4874)
  Lymphocytes, Year 3, Week 8, n=260 | -0.037 (0.5202)
  Lymphocytes, Year 3, Week 16, n=258 | -0.019 (0.5004)
  Lymphocytes, Year 3, Week 24, n=242 | -0.045 (0.5131)
  Lymphocytes, Year 3, Week 32, n=248 | -0.008 (0.4702)
  Lymphocytes, Year 3, Week 40, n=242 | -0.015 (0.5407)
  Lymphocytes, Year 3, Week 48, n=240 | -0.016 (0.5858)
  Lymphocytes, Year 4, Week 8, n=234 | -0.041 (0.4933)
  Lymphocytes, Year 4, Week 16, n=238 | -0.012 (0.4974)
  Lymphocytes, Year 4, Week 24, n=227 | 0.034 (0.5406)
  Lymphocytes, Year 4, Week 32, n=229 | 0.017 (0.5270)
  Lymphocytes, Year 4, Week 40, n=216 | 0.003 (0.4347)
  Lymphocytes, Year 4, Week 48, n=220 | 0.017 (0.4826)
  Lymphocytes, Year 5, Week 8, n=215 | 0.012 (0.4654)
  Lymphocytes, Year 5, Week 16, n=214 | 0.050 (0.5205)
  Lymphocytes, Year 5, Week 24, n=207 | 0.052 (0.5355)
  Lymphocytes, Year 5, Week 32, n=207 | 0.031 (0.5323)
  Lymphocytes, Year 5, Week 40, n=196 | 0.057 (0.5482)
  Lymphocytes, Year 5, Week 48, n=209 | 0.031 (0.5125)
  Lymphocytes, Year 6, Week 8, n=206 | 0.059 (0.5734)
  Lymphocytes, Year 6, Week 16, n=195 | 0.045 (0.5931)
  Lymphocytes, Year 6, Week 24, n=192 | 0.087 (0.5757)
  Lymphocytes, Year 6, Week 32, n=197 | 0.066 (0.5970)
  Lymphocytes, Year 6, Week 40, n=183 | 0.075 (0.5984)
  Lymphocytes, Year 6, Week 48, n=188 | 0.043 (0.5839)
  Lymphocytes, Year 7, Week 8, n=180 | 0.110 (0.6114)
  Lymphocytes, Year 7, Week 16, n=181 | 0.077 (0.6114)
  Lymphocytes, Year 7, Week 24, n=176 | 0.091 (0.5944)
  Lymphocytes, Year 7, Week 32, n=179 | 0.104 (0.5944)
  Lymphocytes, Year 7, Week 40, n=177 | 0.075 (0.5385)
  Lymphocytes, Year 7, Week 48, n=173 | 0.060 (0.6039)
  Lymphocytes, Year 8, Week 8, n=172 | 0.036 (0.5942)
  Lymphocytes, Year 8, Week 16, n=173 | -0.005 (0.5480)
  Lymphocytes, Year 8, Week 24, n=170 | 0.030 (0.6126)
  Lymphocytes, Year 8, Week 32, n=169 | -0.020 (0.5269)
  Lymphocytes, Year 8, Week 40, n=162 | 0.065 (0.6260)
  Lymphocytes, Year 8, Week 48, n=161 | 0.087 (0.7204)
  Lymphocytes, Year 9, Week 8, n=164 | 0.090 (0.6612)
  Lymphocytes, Year 9, Week 16, n=161 | 0.022 (0.5664)
  Lymphocytes, Year 9, Week 24, n=163 | 0.062 (0.5704)
  Lymphocytes, Year 9, Week 32, n=159 | 0.017 (0.5326)
  Lymphocytes, Year 9, Week 40, n=156 | 0.069 (0.6410)
  Lymphocytes, Year 9, Week 48, n=151 | 0.064 (0.5979)
  Lymphocytes, Year 10, Week 8, n=149 | 0.046 (0.5547)
  Lymphocytes, Year 10, Week 16, n=145 | 0.089 (0.6336)
  Lymphocytes, Year 10, Week 24, n=147 | 0.033 (0.5811)
  Lymphocytes, Year 10, Week 32, n=142 | 0.076 (0.5914)
  Lymphocytes, Year 10, Week 40, n=137 | 0.071 (0.5621)
  Lymphocytes, Year 10, Week 48, n=137 | 0.073 (0.5807)
  Lymphocytes, Year 11, Week 8, n=137 | 0.112 (0.5764)
  Lymphocytes, Year 11, Week 16, n=130 | 0.112 (0.6926)
  Lymphocytes, Year 11, Week 24, n=130 | 0.129 (0.7026)
  Lymphocytes, Year 11, Week 32, n=128 | 0.139 (0.6249)
  Lymphocytes, Year 11, Week 40, n=122 | 0.143 (0.6927)
  Lymphocytes, Year 11, Week 48, n=106 | 0.133 (0.5942)
  Lymphocytes, Year 12, Week 8, n=109 | 0.145 (0.5976)
  Lymphocytes, Year 12, Week 16, n=97 | 0.179 (0.5839)
  Lymphocytes, Year 12, Week 24, n=86 | 0.150 (0.5857)
  Lymphocytes, Year 12, Week 32, n=88 | 0.135 (0.6319)
  Lymphocytes, Year 12, Week 40, n=83 | 0.150 (0.6512)
  Lymphocytes, Year 12, Week 48, n=72 | 0.106 (0.5855)
  Lymphocytes, Year 13, Week 8, n=53 | 0.133 (0.6269)
  Lymphocytes, Year 13, Week 16, n=42 | 0.078 (0.6783)
  Lymphocytes, Year 13, Week 24, n=20 | 0.131 (0.6760)
  Lymphocytes, Year 13, Week 32, n=7 | 0.293 (0.8019)
  Lymphocytes, Year 13, Week 40, n=1 | 0.160 (NA) — No value as only one participant was analyzed.
  Lymphocytes, Exit, n=241 | 0.088 (0.6208)
  Lymphocytes, 8-Week Follow-up, n=219 | 0.119 (0.6554)
  Lymphocytes, 24-Week Follow-up, n=198 | 0.054 (0.6847)
  Monocytes, Year 1, Week 8, n=287 | 0.014 (0.1795)
  Monocytes, Year 1, Week 16, n=288 | 0.018 (0.1903)
  Monocytes, Year 1, Week 24, n=293 | 0.007 (0.1834)
  Monocytes, Year 1, Week 32, n=290 | 0.016 (0.1666)
  Monocytes, Year 1, Week 40, n=287 | 0.020 (0.1750)
  Monocytes, Year 1, Week 48, n=287 | 0.018 (0.1739)
  Monocytes, Year 2, Week 8, n=288 | 0.009 (0.1718)
  Monocytes, Year 2, Week 16, n=279 | 0.016 (0.1783)
  Monocytes, Year 2, Week 24, n=276 | 0.029 (0.1764)
  Monocytes, Year 2, Week 32, n=281 | 0.018 (0.1842)
  Monocytes, Year 2, Week 40, n=262 | 0.014 (0.1848)
  Monocytes, Year 2, Week 48, n=260 | 0.030 (0.1594)
  Monocytes, Year 3, Week 8, n=260 | 0.024 (0.1677)
  Monocytes, Year 3, Week 16, n=258 | 0.038 (0.1705)
  Monocytes, Year 3, Week 24, n=242 | 0.034 (0.1632)
  Monocytes, Year 3, Week 32, n=248 | 0.022 (0.1776)
  Monocytes, Year 3, Week 40, n=242 | 0.044 (0.1650)
  Monocytes, Year 3, Week 48, n=240 | 0.039 (0.1855)
  Monocytes, Year 4, Week 8, n=234 | 0.035 (0.1687)
  Monocytes, Year 4, Week 16, n=238 | 0.039 (0.1665)
  Monocytes, Year 4, Week 24, n=227 | 0.032 (0.1667)
  Monocytes, Year 4, Week 32, n=229 | 0.027 (0.1566)
  Monocytes, Year 4, Week 40, n=216 | 0.035 (0.1688)
  Monocytes, Year 4, Week 48, n=220 | 0.015 (0.1771)
  Monocytes, Year 5, Week 8, n=215 | 0.018 (0.1824)
  Monocytes, Year 5, Week 16, n=214 | 0.036 (0.1527)
  Monocytes, Year 5, Week 24, n=207 | 0.041 (0.1632)
  Monocytes, Year 5, Week 32, n=207 | 0.039 (0.1625)
  Monocytes, Year 5, Week 40, n=196 | 0.049 (0.1510)
  Monocytes, Year 5, Week 48, n=209 | 0.050 (0.1628)
  Monocytes, Year 6, Week 8, n=206 | 0.045 (0.1670)
  Monocytes, Year 6, Week 16, n=195 | 0.033 (0.1700)
  Monocytes, Year 6, Week 24, n=192 | 0.030 (0.1556)
  Monocytes, Year 6, Week 32, n=197 | 0.048 (0.1635)
  Monocytes, Year 6, Week 40, n=183 | 0.051 (0.1342)
  Monocytes, Year 6, Week 48, n=188 | 0.038 (0.1665)
  Monocytes, Year 7, Week 8, n=180 | 0.028 (0.1507)
  Monocytes, Year 7, Week 16, n=181 | 0.030 (0.1482)
  Monocytes, Year 7, Week 24, n=176 | 0.033 (0.1583)
  Monocytes, Year 7, Week 32, n=179 | 0.039 (0.1534)
  Monocytes, Year 7, Week 40, n=177 | 0.047 (0.1391)
  Monocytes, Year 7, Week 48, n=173 | 0.055 (0.1508)
  Monocytes, Year 8, Week 8, n=172 | 0.071 (0.1536)
  Monocytes, Year 8, Week 16, n=173 | 0.072 (0.1464)
  Monocytes, Year 8, Week 24, n=170 | 0.075 (0.1545)
  Monocytes, Year 8, Week 32, n=169 | 0.049 (0.1414)
  Monocytes, Year 8, Week 40, n=162 | 0.070 (0.1480)
  Monocytes, Year 8, Week 48, n=161 | 0.072 (0.1744)
  Monocytes, Year 9, Week 8, n=164 | 0.069 (0.1513)
  Monocytes, Year 9, Week 16, n=161 | 0.063 (0.1462)
  Monocytes, Year 9, Week 24, n=163 | 0.077 (0.1603)
  Monocytes, Year 9, Week 32, n=159 | 0.074 (0.1393)
  Monocytes, Year 9, Week 40, n=156 | 0.075 (0.1440)
  Monocytes, Year 9, Week 48, n=151 | 0.063 (0.1576)
  Monocytes, Year 10, Week 8, n=149 | 0.084 (0.1511)
  Monocytes, Year 10, Week 16, n=145 | 0.083 (0.1439)
  Monocytes, Year 10, Week 24, n=147 | 0.087 (0.1874)
  Monocytes, Year 10, Week 32, n=142 | 0.077 (0.1517)
  Monocytes, Year 10, Week 40, n=137 | 0.064 (0.1522)
  Monocytes, Year 10, Week 48, n=137 | 0.070 (0.1454)
  Monocytes, Year 11, Week 8, n=137 | 0.077 (0.1622)
  Monocytes, Year 11, Week 16, n=130 | 0.077 (0.1484)
  Monocytes, Year 11, Week 24, n=130 | 0.079 (0.1775)
  Monocytes, Year 11, Week 32, n=128 | 0.080 (0.1849)
  Monocytes, Year 11, Week 40, n=122 | 0.075 (0.1435)
  Monocytes, Year 11, Week 48, n=106 | 0.075 (0.1854)
  Monocytes, Year 12, Week 8, n=109 | 0.088 (0.2166)
  Monocytes, Year 12, Week 16, n=97 | 0.104 (0.1829)
  Monocytes, Year 12, Week 24, n=86 | 0.073 (0.1616)
  Monocytes, Year 12, Week 32, n=88 | 0.065 (0.1682)
  Monocytes, Year 12, Week 40, n=83 | 0.078 (0.1734)
  Monocytes, Year 12, Week 48, n=72 | 0.060 (0.1635)
  Monocytes, Year 13, Week 8, n=53 | 0.013 (0.1453)
  Monocytes, Year 13, Week 16, n=42 | 0.061 (0.1882)
  Monocytes, Year 13, Week 24, n=20 | 0.074 (0.1471)
  Monocytes, Year 13, Week 32, n=7 | 0.097 (0.1452)
  Monocytes, Year 13, Week 40, n=1 | 0.120 (NA) — No value as only one participant was analyzed.
  Monocytes, Exit, n=241 | 0.062 (0.1813)
  Monocytes, 8-Week Follow-up, n=219 | 0.061 (0.2153)
  Monocytes, 24-Week Follow-up , n=198 | 0.049 (0.2118)
  Neutrophils segmented, Year 1, Week 8, n=287 | 0.003 (1.7881)
  Neutrophils segmented, Year 1, Week 16, n=288 | -0.107 (1.7909)
  Neutrophils segmented, Year 1, Week 24, n=293 | -0.166 (1.9241)
  Neutrophils segmented, Year 1, Week 32, n=290 | -0.129 (2.0814)
  Neutrophils segmented, Year 1, Week 40, n=287 | -0.140 (1.7884)
  Neutrophils segmented, Year 1, Week 48, n=287 | -0.223 (1.7187)
  Neutrophils segmented, Year 2, Week 8, n=288 | -0.301 (2.0434)
  Neutrophils segmented, Year 2, Week 16, n=279 | -0.392 (2.0076)
  Neutrophils segmented, Year 2, Week 24, n=276 | -0.250 (2.2163)
  Neutrophils segmented, Year 2, Week 32, n=281 | -0.129 (2.1622)
  Neutrophils segmented, Year 2, Week 40, n=262 | -0.236 (2.1413)
  Neutrophils segmented, Year 2, Week 48, n=260 | -0.148 (2.1176)
  Neutrophils segmented, Year 3, Week 8, n=260 | -0.333 (2.1308)
  Neutrophils segmented, Year 3, Week 16, n=258 | -0.308 (2.2022)
  Neutrophils segmented, Year 3, Week 24, n=242 | -0.129 (1.9829)
  Neutrophils segmented, Year 3, Week 32, n=248 | -0.211 (2.2333)
  Neutrophils segmented, Year 3, Week 40, n=242 | -0.161 (1.9939)
  Neutrophils segmented, Year 3, Week 48, n=240 | -0.159 (2.1315)
  Neutrophils segmented, Year 4, Week 8, n=234 | -0.119 (2.0635)
  Neutrophils segmented, Year 4, Week 16, n=238 | -0.177 (2.1063)
  Neutrophils segmented, Year 4, Week 24, n=227 | -0.136 (1.9402)
  Neutrophils segmented, Year 4, Week 32, n=229 | -0.123 (2.2231)
  Neutrophils segmented, Year 4, Week 40, n=216 | -0.119 (1.9639)
  Neutrophils segmented, Year 4, Week 48, n=220 | -0.024 (2.2228)
  Neutrophils segmented, Year 5, Week 8, n=215 | -0.169 (2.2107)
  Neutrophils segmented, Year 5, Week 16, n=214 | -0.189 (2.0362)
  Neutrophils segmented, Year 5, Week 24, n=207 | -0.120 (2.0997)
  Neutrophils segmented, Year 5, Week 32, n=207 | -0.088 (2.1895)
  Neutrophils segmented, Year 5, Week 40, n=196 | -0.064 (2.1536)
  Neutrophils segmented, Year 5, Week 48, n=209 | 0.014 (2.0473)
  Neutrophils segmented, Year 6, Week 8, n=206 | -0.097 (1.9542)
  Neutrophils segmented, Year 6, Week 16, n=195 | -0.218 (2.2682)
  Neutrophils segmented, Year 6, Week 24, n=192 | -0.226 (2.1749)
  Neutrophils segmented, Year 6, Week 32, n=197 | -0.144 (2.0689)
  Neutrophils segmented, Year 6, Week 40, n=183 | -0.359 (2.2241)
  Neutrophils segmented, Year 6, Week 48, n=188 | -0.306 (2.1609)
  Neutrophils segmented, Year 7, Week 8, n=180 | -0.371 (2.1016)
  Neutrophils segmented, Year 7, Week 16, n=181 | -0.410 (2.0287)
  Neutrophils segmented, Year 7, Week 24, n=176 | -0.363 (2.2018)
  Neutrophils segmented, Year 7, Week 32, n=179 | -0.214 (2.2148)
  Neutrophils segmented, Year 7, Week 40, n=177 | -0.360 (2.2393)
  Neutrophils segmented, Year 7, Week 48, n=173 | -0.423 (2.1389)
  Neutrophils segmented, Year 8, Week 8, n=172 | -0.387 (2.1621)
  Neutrophils segmented, Year 8, Week 16, n=173 | -0.310 (2.1373)
  Neutrophils segmented, Year 8, Week 24, n=170 | -0.152 (2.3134)
  Neutrophils segmented, Year 8, Week 32, n=169 | -0.218 (2.1233)
  Neutrophils segmented, Year 8, Week 40, n=162 | -0.281 (2.2042)
  Neutrophils segmented, Year 8, Week 48, n=161 | -0.407 (2.2558)
  Neutrophils segmented, Year 9, Week 8, n=164 | -0.161 (2.1968)
  Neutrophils segmented, Year 9, Week 16, n=161 | -0.332 (2.0436)
  Neutrophils segmented, Year 9, Week 24, n=163 | -0.240 (2.1439)
  Neutrophils segmented, Year 9, Week 32, n=159 | -0.114 (2.3286)
  Neutrophils segmented, Year 9, Week 40, n=156 | -0.252 (2.2301)
  Neutrophils segmented, Year 9, Week 48, n=151 | -0.268 (2.4153)
  Neutrophils segmented, Year 10, Week 8, n=149 | 0.049 (2.4409)
  Neutrophils segmented, Year 10, Week 16, n=145 | 0.008 (2.7611)
  Neutrophils segmented, Year 10, Week 24, n=147 | -0.166 (2.2970)
  Neutrophils segmented, Year 10, Week 32, n=142 | -0.299 (2.1597)
  Neutrophils segmented, Year 10, Week 40, n=137 | -0.051 (2.1023)
  Neutrophils segmented, Year 10, Week 48, n=137 | -0.176 (2.0628)
  Neutrophils segmented, Year 11, Week 8, n=137 | -0.077 (2.4456)
  Neutrophils segmented, Year 11, Week 16, n=130 | -0.035 (2.3922)
  Neutrophils segmented, Year 11, Week 24, n=130 | -0.031 (2.2826)
  Neutrophils segmented, Year 11, Week 32, n=128 | 0.145 (2.4689)
  Neutrophils segmented, Year 11, Week 40, n=122 | -0.043 (2.2994)
  Neutrophils segmented, Year 11, Week 48, n=106 | -0.004 (2.5913)
  Neutrophils segmented, Year 12, Week 8, n=109 | -0.011 (2.5216)
  Neutrophils segmented, Year 12, Week 16, n=97 | -0.032 (2.6750)
  Neutrophils segmented, Year 12, Week 24, n=86 | -0.126 (2.2583)
  Neutrophils segmented, Year 12, Week 32, n=88 | -0.081 (2.5744)
  Neutrophils segmented, Year 12, Week 40, n=83 | -0.293 (2.2448)
  Neutrophils segmented, Year 12, Week 48, n=72 | -0.126 (2.9212)
  Neutrophils segmented, Year 13, Week 8, n=53 | -0.747 (2.7599)
  Neutrophils segmented, Year 13, Week 16, n=42 | 0.169 (2.5731)
  Neutrophils segmented, Year 13, Week 24, n=20 | -0.121 (2.8499)
  Neutrophils segmented, Year 13, Week 32, n=7 | -0.927 (2.9565)
  Neutrophils segmented, Year 13, Week 40, n=1 | -0.680 (NA) — No value as only one participant was analyzed.
  Neutrophils segmented, Exit, n=241 | 0.436 (2.6133)
  Neutrophils segmented, 8-Week Follow-up, n=219 | 0.514 (3.6918)
  Neutrophils segmented, 24-Week Follow-up, n=198 | 0.369 (2.6988)
  Platelets, Year 1, Week ,8 n=279 | 3.7 (34.73)
  Platelets, Year 1, Week 16, n=279 | 4.5 (34.48)
  Platelets, Year 1, Week 24, n=286 | 7.9 (36.76)
  Platelets, Year 1, Week 32, n=285 | 10.3 (41.03)
  Platelets, Year 1, Week 40, n=283 | 13.1 (39.75)
  Platelets, Year 1, Week 48, n=282 | 13.2 (46.13)
  Platelets, Year 2, Week 8, n=280 | 18.1 (48.14)
  Platelets, Year 2, Week 16, n=276 | 15.4 (45.99)
  Platelets, Year 2, Week 24, n=273 | 16.7 (49.67)
  Platelets, Year 2, Week 32, n=277 | 24.0 (50.04)
  Platelets, Year 2, Week 40, n=259 | 21.9 (46.95)
  Platelets, Year 2, Week 48, n=255 | 21.2 (50.63)
  Platelets, Year 3, Week 8, n=256 | 22.0 (53.16)
  Platelets, Year 3, Week 16, n=253 | 22.7 (55.76)
  Platelets, Year 3, Week 24, n=239 | 18.4 (50.97)
  Platelets, Year 3, Week 32, n=243 | 14.1 (50.03)
  Platelets, Year 3, Week 40, n=240 | 14.3 (55.47)
  Platelets, Year 3, Week 48, n=235 | 12.6 (56.20)
  Platelets, Year 4, Week 8, n=230 | 11.5 (48.78)
  Platelets, Year 4, Week 16, n=234 | 11.7 (54.46)
  Platelets, Year 4, Week 24, n=226 | 11.7 (51.12)
  Platelets, Year 4, Week 32, n=220 | 9.6 (55.85)
  Platelets, Year 4, Week 40, n=214 | 5.6 (54.44)
  Platelets, Year 4, Week 48, n=216 | 6.7 (56.74)
  Platelets, Year 5, Week 8, n=211 | 4.6 (62.04)
  Platelets, Year 5, Week 16, n=212 | -2.1 (54.06)
  Platelets, Year 5, Week 24, n=206 | -3.0 (52.05)
  Platelets, Year 5, Week 32, n=203 | -4.8 (53.16)
  Platelets, Year 5, Week 40, n=194 | -7.7 (51.97)
  Platelets, Year 5, Week 48, n=206 | -3.4 (54.93)
  Platelets, Year 6, Week 8, n=203 | -10.8 (56.67)
  Platelets, Year 6, Week 16, n=193 | -12.7 (56.99)
  Platelets, Year 6, Week 24, n=190 | -15.6 (51.76)
  Platelets, Year 6, Week 32, n=194 | -12.2 (52.69)
  Platelets, Year 6, Week 40, n=182 | -15.8 (56.24)
  Platelets, Year 6, Week 48, n=186 | -19.5 (52.68)
  Platelets, Year 7, Week 8, n=179 | -17.3 (53.81)
  Platelets, Year 7, Week 16, n=179 | -24.2 (49.52)
  Platelets, Year 7, Week 24, n=175 | -22.0 (52.19)
  Platelets, Year 7, Week 32, n=178 | -19.4 (59.77)
  Platelets, Year 7, Week 40, n=176 | -16.6 (63.50)
  Platelets, Year 7, Week 48, n=171 | -14.3 (60.69)
  Platelets, Year 8, Week 8, n=168 | -11.5 (54.16)
  Platelets, Year 8, Week 16, n=172 | -15.0 (58.24)
  Platelets, Year 8, Week 24, n=169 | -11.0 (56.12)
  Platelets, Year 8, Week 32, n=168 | -13.9 (55.53)
  Platelets, Year 8, Week 40, n=161 | -12.0 (62.73)
  Platelets, Year 8, Week 48, n=161 | -8.9 (80.44)
  Platelets, Year 9, Week 8, n=162 | -8.4 (64.02)
  Platelets, Year 9, Week 16, n=160 | -11.7 (68.06)
  Platelets, Year 9, Week 24, n=162 | -13.6 (60.20)
  Platelets, Year 9, Week 32, n=158 | -16.8 (62.14)
  Platelets, Year 9, Week 40, n=156 | -13.4 (63.09)
  Platelets, Year 9, Week 48, n=150 | -13.0 (65.20)
  Platelets, Year 10, Week 8, n=149 | -10.9 (60.24)
  Platelets, Year 10, Week 16, n=144 | -9.7 (62.61)
  Platelets, Year 10, Week 24, n=146 | -9.7 (60.67)
  Platelets, Year 10, Week 32, n=141 | -10.6 (62.35)
  Platelets, Year 10, Week 40, n=136 | -9.5 (61.80)
  Platelets, Year 10, Week 48, n=136 | -11.7 (61.81)
  Platelets, Year 11, Week 8, n=136 | -8.4 (69.58)
  Platelets, Year 11, Week 16, n=129 | -6.4 (63.81)
  Platelets, Year 11, Week 24, n=129 | -6.7 (61.75)
  Platelets, Year 11, Week 32, n=127 | -3.0 (65.54)
  Platelets, Year 11, Week 40, n=121 | -5.8 (68.01)
  Platelets, Year 11, Week 48, n=105 | -7.8 (62.13)
  Platelets, Year 12, Week 8, n=108 | -4.1 (73.02)
  Platelets, Year 12, Week 16, n=96 | -10.6 (68.02)
  Platelets, Year 12, Week 24, n=84 | -11.5 (60.94)
  Platelets, Year 12, Week 32, n=87 | -5.7 (70.98)
  Platelets, Year 12, Week 40, n=82 | -10.7 (67.51)
  Platelets, Year 12, Week 48, n=72 | -8.7 (80.99)
  Platelets, Year 13, Week 8, n=53 | -8.6 (70.53)
  Platelets, Year 13, Week 16, n=41 | -6.2 (61.57)
  Platelets, Year 13, Week 24, n=20 | -7.1 (47.37)
  Platelets, Year 13, Week 32, n=7 | -6.7 (51.61)
  Platelets, Year 13, Week 40, n=1 | -29.0 (NA) — No value as only one participant was analyzed.
  Platelets, Exit, n=236 | 8.4 (77.24)
  Platelets, 8-Week Follow-up, n=217 | 8.2 (71.32)
  Platelets, 24-Week Follow-up, n=194 | 4.0 (67.29)

6. Primary Outcome: Change From Baseline in Erythrocytes at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in erythrocytes is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^12 per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
10^12 per liter
  Erythrocytes, Year 1, Week 8, n=287 | 0.01 (0.313)
  Erythrocytes, Year 1, Week 16, n=288 | 0.04 (0.361)
  Erythrocytes, Year 1, Week 24, n=293 | 0.05 (0.309)
  Erythrocytes, Year 1, Week 32, n=291 | 0.07 (0.301)
  Erythrocytes, Year 1, Week 40, n=287 | 0.10 (0.321)
  Erythrocytes, Year 1, Week 48, n=287 | 0.11 (0.338)
  Erythrocytes, Year 2, Week 8, n=288 | 0.07 (0.339)
  Erythrocytes, Year 2, Week 16, n=280 | 0.09 (0.320)
  Erythrocytes, Year 2, Week 24, n=278 | 0.12 (0.331)
  Erythrocytes, Year 2, Week 32, n=281 | 0.15 (0.331)
  Erythrocytes, Year 2, Week 40, n=262 | 0.17 (0.330)
  Erythrocytes, Year 2, Week 48, n=260 | 0.19 (0.336)
  Erythrocytes, Year 3, Week 8, n=260 | 0.18 (0.331)
  Erythrocytes, Year 3, Week 16, n=258 | 0.19 (0.347)
  Erythrocytes, Year 3, Week 24, n=242 | 0.17 (0.384)
  Erythrocytes, Year 3, Week 32, n=248 | 0.16 (0.356)
  Erythrocytes, Year 3, Week 40, n=243 | 0.17 (0.369)
  Erythrocytes, Year 3, Week 48, n=240 | 0.15 (0.368)
  Erythrocytes, Year 4, Week 8, n=235 | 0.15 (0.392)
  Erythrocytes, Year 4, Week 16, n=238 | 0.15 (0.367)
  Erythrocytes, Year 4, Week 24, n=227 | 0.12 (0.363)
  Erythrocytes, Year 4, Week 32, n=229 | 0.14 (0.394)
  Erythrocytes, Year 4, Week 40, n=216 | 0.14 (0.383)
  Erythrocytes, Year 4, Week 48, n=220 | 0.14 (0.420)
  Erythrocytes, Year 5, Week 8, n=215 | 0.13 (0.435)
  Erythrocytes, Year 5, Week 16, n=214 | 0.15 (0.432)
  Erythrocytes, Year 5, Week 24, n=207 | 0.13 (0.426)
  Erythrocytes, Year 5, Week 32, n=207 | 0.12 (0.430)
  Erythrocytes, Year 5, Week 40, n=196 | 0.15 (0.417)
  Erythrocytes, Year 5, Week 48, n=209 | 0.15 (0.420)
  Erythrocytes, Year 6, Week 8, n=206 | 0.13 (0.441)
  Erythrocytes, Year 6, Week 16, n=195 | 0.10 (0.448)
  Erythrocytes, Year 6, Week 24, n=192 | 0.13 (0.380)
  Erythrocytes, Year 6, Week 32, n=197 | 0.14 (0.420)
  Erythrocytes, Year 6, Week 40, n=184 | 0.15 (0.430)
  Erythrocytes, Year 6, Week 48, n=188 | 0.13 (0.401)
  Erythrocytes, Year 7, Week 8, n=180 | 0.12 (0.397)
  Erythrocytes, Year 7, Week 16, n=181 | 0.09 (0.407)
  Erythrocytes, Year 7, Week 24, n=176 | 0.11 (0.390)
  Erythrocytes, Year 7, Week 32, n=179 | 0.14 (0.395)
  Erythrocytes, Year 7, Week 40, n=177 | 0.09 (0.391)
  Erythrocytes, Year 7, Week 48, n=173 | 0.09 (0.394)
  Erythrocytes, Year 8, Week 8, n=172 | 0.09 (0.378)
  Erythrocytes, Year 8, Week 16, n=173 | 0.08 (0.368)
  Erythrocytes, Year 8, Week 24, n=170 | 0.10 (0.388)
  Erythrocytes, Year 8, Week 32, n=169 | 0.11 (0.373)
  Erythrocytes, Year 8, Week 40, n=162 | 0.10 (0.415)
  Erythrocytes, Year 8, Week 48, n=161 | 0.12 (0.411)
  Erythrocytes, Year 9, Week 8, n=164 | 0.11 (0.402)
  Erythrocytes, Year 9, Week 16, n=161 | 0.09 (0.396)
  Erythrocytes, Year 9, Week 24, n=163 | 0.08 (0.387)
  Erythrocytes, Year 9, Week 32, n=160 | 0.11 (0.409)
  Erythrocytes, Year 9, Week 40, n=156 | 0.09 (0.407)
  Erythrocytes, Year 9, Week 48, n=151 | 0.11 (0.431)
  Erythrocytes, Year 10, Week 8, n=150 | 0.16 (0.442)
  Erythrocytes, Year 10, Week 16, n=145 | 0.17 (0.411)
  Erythrocytes, Year 10, Week 24, n=147 | 0.21 (0.427)
  Erythrocytes, Year 10, Week 32, n=142 | 0.18 (0.419)
  Erythrocytes, Year 10, Week 40, n=137 | 0.20 (0.417)
  Erythrocytes, Year 10, Week 48, n=137 | 0.19 (0.429)
  Erythrocytes, Year 11, Week 8, n=137 | 0.20 (0.430)
  Erythrocytes, Year 11, Week 16, n=130 | 0.24 (0.422)
  Erythrocytes, Year 11, Week 24, n=130 | 0.25 (0.436)
  Erythrocytes, Year 11, Week 32, n=128 | 0.27 (0.410)
  Erythrocytes, Year 11, Week 40, n=122 | 0.27 (0.426)
  Erythrocytes, Year 11, Week 48, n=106 | 0.25 (0.426)
  Erythrocytes, Year 12, Week 8, n=109 | 0.29 (0.422)
  Erythrocytes, Year 12, Week 16, n=97 | 0.28 (0.435)
  Erythrocytes, Year 12, Week 24, n=86 | 0.33 (0.483)
  Erythrocytes, Year 12, Week 32, n=88 | 0.26 (0.512)
  Erythrocytes, Year 12, Week 40, n=83 | 0.31 (0.428)
  Erythrocytes, Year 12, Week 48, n=72 | 0.32 (0.467)
  Erythrocytes, Year 13, Week 8, n=53 | 0.35 (0.400)
  Erythrocytes, Year 13, Week 16, n=42 | 0.34 (0.387)
  Erythrocytes, Year 13, Week 24, n=20 | 0.30 (0.407)
  Erythrocytes, Year 13, Week 32, n=7 | 0.20 (0.379)
  Erythrocytes, Year 13, Week 40, n=1 | 0.30 (NA) — No value as only one participant was analyzed.
  Erythrocytes, Exit, n=241 | 0.27 (0.473)
  Erythrocytes, 8-Week Follow-up, n=220 | 0.28 (0.478)
  Erythrocytes, 24-Week Follow-up , n=198 | 0.33 (0.539)

7. Primary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in hematocrit is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of blood by volume
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Percentage of blood by volume
  Hematocrit, Year 1, Week 8, n=287 | 0.11 (2.908)
  Hematocrit, Year 1, Week 16, n=288 | 0.23 (3.109)
  Hematocrit, Year 1, Week 24, n=293 | 0.28 (2.917)
  Hematocrit, Year 1, Week 32, n=291 | 0.44 (2.973)
  Hematocrit, Year 1, Week 40, n=287 | 0.60 (3.199)
  Hematocrit, Year 1, Week 48, n=287 | 0.84 (3.431)
  Hematocrit, Year 2, Week 8, n=288 | 0.67 (3.415)
  Hematocrit, Year 2, Week 16, n=280 | 0.93 (3.332)
  Hematocrit, Year 2, Week 24, n=278 | 0.96 (3.435)
  Hematocrit, Year 2, Week 32, n=281 | 1.34 (3.496)
  Hematocrit, Year 2, Week 40, n=262 | 1.43 (3.476)
  Hematocrit, Year 2, Week 48, n=260 | 1.65 (3.444)
  Hematocrit, Year 3, Week 8, n=260 | 1.54 (3.453)
  Hematocrit, Year 3, Week 16, n=258 | 1.76 (3.508)
  Hematocrit, Year 3, Week 24, n=242 | 1.68 (3.709)
  Hematocrit, Year 3, Week 32, n=248 | 1.55 (3.676)
  Hematocrit, Year 3, Week 40, n=243 | 1.55 (3.703)
  Hematocrit, Year 3, Week 48, n=240 | 1.26 (3.726)
  Hematocrit, Year 4, Week 8, n=235 | 1.33 (3.908)
  Hematocrit, Year 4, Week 16, n=238 | 1.37 (3.759)
  Hematocrit, Year 4, Week 24, n=227 | 1.27 (3.680)
  Hematocrit, Year 4, Week 32, n=229 | 1.34 (3.955)
  Hematocrit, Year 4, Week 40, n=216 | 1.39 (3.779)
  Hematocrit, Year 4, Week 48, n=220 | 1.37 (4.033)
  Hematocrit, Year 5, Week 8, n=215 | 1.27 (4.031)
  Hematocrit, Year 5, Week 16, n=214 | 1.58 (3.917)
  Hematocrit, Year 5, Week 24, n=207 | 1.45 (3.905)
  Hematocrit, Year 5, Week 32, n=207 | 1.39 (3.979)
  Hematocrit, Year 5, Week 40, n=196 | 1.59 (4.031)
  Hematocrit, Year 5, Week 48, n=209 | 1.35 (3.929)
  Hematocrit, Year 6, Week 8, n=206 | 1.24 (4.128)
  Hematocrit, Year 6, Week 16, n=195 | 1.07 (4.114)
  Hematocrit, Year 6, Week 24, n=192 | 1.43 (3.648)
  Hematocrit, Year 6, Week 32, n=197 | 1.77 (3.822)
  Hematocrit, Year 6, Week 40, n=184 | 2.07 (4.089)
  Hematocrit, Year 6, Week 48, n=188 | 2.02 (3.961)
  Hematocrit, Year 7, Week 8, n=180 | 1.80 (3.808)
  Hematocrit, Year 7, Week 16, n=181 | 1.50 (3.883)
  Hematocrit, Year 7, Week 24, n=176 | 1.88 (3.840)
  Hematocrit, Year 7, Week 32, n=179 | 2.25 (3.824)
  Hematocrit, Year 7, Week 40, n=177 | 2.07 (3.907)
  Hematocrit, Year 7, Week 48, n=173 | 1.97 (3.958)
  Hematocrit, Year 8, Week 8, n=172 | 1.89 (3.909)
  Hematocrit, Year 8, Week 16, n=173 | 1.87 (3.729)
  Hematocrit, Year 8, Week 24, n=170 | 2.12 (4.065)
  Hematocrit, Year 8, Week 32, n=169 | 2.20 (3.954)
  Hematocrit, Year 8, Week 40, n=162 | 2.10 (4.122)
  Hematocrit, Year 8, Week 48, n=161 | 2.18 (4.029)
  Hematocrit, Year 9, Week 8, n=164 | 1.99 (3.995)
  Hematocrit, Year 9, Week 16, n=161 | 1.76 (4.114)
  Hematocrit, Year 9, Week 24, n=163 | 1.70 (4.020)
  Hematocrit, Year 9, Week 32, n=160 | 1.95 (4.171)
  Hematocrit, Year 9, Week 40, n=156 | 1.88 (4.302)
  Hematocrit, Year 9, Week 48, n=151 | 2.32 (4.174)
  Hematocrit, Year 10, Week 8, n=150 | 2.87 (4.087)
  Hematocrit, Year 10, Week 16, n=145 | 2.80 (4.050)
  Hematocrit, Year 10, Week 24, n=147 | 2.94 (4.046)
  Hematocrit, Year 10, Week 32, n=142 | 2.78 (4.046)
  Hematocrit, Year 10, Week 40, n=137 | 2.95 (3.884)
  Hematocrit, Year 10, Week 48, n=137 | 3.00 (4.245)
  Hematocrit, Year 11, Week 8, n=137 | 3.04 (4.176)
  Hematocrit, Year 11, Week 16, n=130 | 3.20 (4.155)
  Hematocrit, Year 11, Week 24, n=130 | 2.93 (4.331)
  Hematocrit, Year 11, Week 32, n=128 | 3.06 (3.976)
  Hematocrit, Year 11, Week 40, n=122 | 3.15 (4.098)
  Hematocrit, Year 11, Week 48, n=106 | 2.93 (4.356)
  Hematocrit, Year 12, Week 8, n=109 | 3.12 (4.223)
  Hematocrit, Year 12, Week 16, n=97 | 3.43 (4.321)
  Hematocrit, Year 12, Week 24, n=86 | 3.74 (4.867)
  Hematocrit, Year 12, Week 32, n=88 | 2.99 (4.826)
  Hematocrit, Year 12, Week 40, n=83 | 3.57 (4.377)
  Hematocrit, Year 12, Week 48, n=72 | 3.88 (4.439)
  Hematocrit, Year 13, Week 8, n=53 | 4.20 (3.776)
  Hematocrit, Year 13, Week 16, n=42 | 4.26 (3.803)
  Hematocrit, Year 13, Week 24, n=20 | 3.81 (3.930)
  Hematocrit, Year 13, Week 32, n=7 | 3.26 (4.547)
  Hematocrit, Year 13, Week 40, n=1 | 2.20 (NA) — No value as only one participant was analyzed.
  Hematocrit, Exit, n=241 | 3.35 (4.596)
  Hematocrit, 8-Week Follow-up, n=220 | 3.46 (4.690)
  Hematocrit, 24-Week Follow-up , n=198 | 3.51 (4.627)

8. Primary Outcome: Change From Baseline in Hemoglobin at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in hemoglobin is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
grams per liter
  Hemoglobin, Year 1, Week 8, n=287 | 0.1 (9.42)
  Hemoglobin, Year 1, Week 16, n=288 | 0.6 (10.60)
  Hemoglobin, Year 1, Week 24, n=293 | 1.5 (9.86)
  Hemoglobin, Year 1, Week 32, n=291 | 2.2 (10.37)
  Hemoglobin, Year 1, Week 40, n=287 | 2.8 (10.84)
  Hemoglobin, Year 1, Week 48, n=287 | 2.9 (11.39)
  Hemoglobin, Year 2, Week 8, n=288 | 2.2 (11.62)
  Hemoglobin, Year 2, Week 16, n=280 | 2.8 (11.54)
  Hemoglobin, Year 2, Week 24, n=278 | 3.2 (12.20)
  Hemoglobin, Year 2, Week 32, n=281 | 4.5 (12.19)
  Hemoglobin, Year 2, Week 40, n=262 | 4.9 (12.15)
  Hemoglobin, Year 2, Week 48, n=260 | 5.6 (12.10)
  Hemoglobin, Year 3, Week 8, n=260 | 4.8 (12.01)
  Hemoglobin, Year 3, Week 16, n=258 | 5.2 (12.15)
  Hemoglobin, Year 3, Week 24, n=242 | 5.4 (12.47)
  Hemoglobin, Year 3, Week 32, n=248 | 5.6 (12.59)
  Hemoglobin, Year 3, Week 40, n=243 | 5.9 (12.90)
  Hemoglobin, Year 3, Week 48, n=240 | 5.1 (12.97)
  Hemoglobin, Year 4, Week 8, n=235 | 5.2 (13.49)
  Hemoglobin, Year 4, Week 16, n=238 | 5.2 (13.11)
  Hemoglobin, Year 4, Week 24, n=227 | 4.1 (13.05)
  Hemoglobin, Year 4, Week 32, n=229 | 4.9 (13.64)
  Hemoglobin, Year 4, Week 40, n=216 | 4.9 (13.25)
  Hemoglobin, Year 4, Week 48, n=220 | 5.3 (13.94)
  Hemoglobin, Year 5, Week 8, n=215 | 5.1 (14.20)
  Hemoglobin, Year 5, Week 16, n=214 | 5.5 (13.44)
  Hemoglobin, Year 5, Week 24, n=207 | 4.4 (13.73)
  Hemoglobin, Year 5, Week 32, n=207 | 4.1 (13.39)
  Hemoglobin, Year 5, Week 40, n=196 | 5.2 (14.31)
  Hemoglobin, Year 5, Week 48, n=209 | 5.4 (14.20)
  Hemoglobin, Year 6, Week 8, n=206 | 5.5 (14.72)
  Hemoglobin, Year 6, Week 16, n=195 | 4.8 (14.82)
  Hemoglobin, Year 6, Week 24, n=192 | 5.6 (12.80)
  Hemoglobin, Year 6, Week 32, n=197 | 5.9 (13.12)
  Hemoglobin, Year 6, Week 40, n=184 | 6.6 (13.96)
  Hemoglobin, Year 6, Week 48, n=188 | 6.4 (13.78)
  Hemoglobin, Year 7, Week 8, n=180 | 6.3 (13.58)
  Hemoglobin, Year 7, Week 16, n=181 | 5.5 (13.83)
  Hemoglobin, Year 7, Week 24, n=176 | 6.0 (13.51)
  Hemoglobin, Year 7, Week 32, n=179 | 7.0 (13.37)
  Hemoglobin, Year 7, Week 40, n=177 | 6.4 (13.61)
  Hemoglobin, Year 7, Week 48, n=173 | 5.6 (13.91)
  Hemoglobin, Year 8, Week 8, n=172 | 5.7 (13.69)
  Hemoglobin, Year 8, Week 16, n=173 | 5.3 (13.09)
  Hemoglobin, Year 8, Week 24, n=170 | 6.1 (14.13)
  Hemoglobin, Year 8, Week 32, n=169 | 5.8 (13.33)
  Hemoglobin, Year 8, Week 40, n=162 | 4.9 (13.93)
  Hemoglobin, Year 8, Week 48, n=161 | 5.5 (13.95)
  Hemoglobin, Year 9, Week 8, n=164 | 5.5 (13.79)
  Hemoglobin, Year 9, Week 16, n=161 | 4.9 (14.60)
  Hemoglobin, Year 9, Week 24, n=163 | 4.6 (14.32)
  Hemoglobin, Year 9, Week 32, n=160 | 5.2 (14.39)
  Hemoglobin, Year 9, Week 40, n=156 | 3.9 (15.20)
  Hemoglobin, Year 9, Week 48, n=151 | 4.8 (14.50)
  Hemoglobin, Year 10, Week 8, n=150 | 6.5 (14.46)
  Hemoglobin, Year 10, Week 16, n=145 | 6.5 (14.05)
  Hemoglobin, Year 10, Week 24, n=147 | 6.5 (14.20)
  Hemoglobin, Year 10, Week 32, n=142 | 5.9 (14.02)
  Hemoglobin, Year 10, Week 40, n=137 | 6.0 (13.29)
  Hemoglobin, Year 10, Week 48, n=137 | 5.7 (14.86)
  Hemoglobin, Year 11, Week 8, n=137 | 5.9 (14.40)
  Hemoglobin, Year 11, Week 16, n=130 | 6.4 (14.50)
  Hemoglobin, Year 11, Week 24, n=130 | 5.9 (15.02)
  Hemoglobin, Year 11, Week 32, n=128 | 6.3 (13.79)
  Hemoglobin, Year 11, Week 40, n=122 | 6.7 (14.03)
  Hemoglobin, Year 11, Week 48, n=106 | 6.2 (14.95)
  Hemoglobin, Year 12, Week 8, n=109 | 6.8 (14.55)
  Hemoglobin, Year 12, Week 16, n=97 | 8.1 (15.12)
  Hemoglobin, Year 12, Week 24, n=86 | 8.9 (16.83)
  Hemoglobin, Year 12, Week 32, n=88 | 6.6 (17.18)
  Hemoglobin, Year 12, Week 40, n=83 | 7.0 (15.41)
  Hemoglobin, Year 12, Week 48, n=72 | 8.3 (14.80)
  Hemoglobin, Year 13, Week 8, n=53 | 8.4 (12.37)
  Hemoglobin, Year 13, Week 16, n=42 | 8.0 (12.81)
  Hemoglobin, Year 13, Week 24, n=20 | 6.3 (12.01)
  Hemoglobin, Year 13, Week 32, n=7 | 5.4 (14.27)
  Hemoglobin, Year 13, Week 40, n=1 | 3.0 (NA) — No value as only one participant was analyzed.
  Hemoglobin, Exit, n=241 | 7.4 (15.11)
  Hemoglobin, 8-Week Follow-up, n=220 | 6.7 (15.46)
  Hemoglobin, 24-Week Follow-up , n=198 | 6.8 (14.91)

9. Primary Outcome: Change From Baseline in Albumin and Protein at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in albumin and protein is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
grams/liter
  Albumin, Year 1, Week 8, n=284 | 0.1 (2.36)
  Albumin, Year 1, Week 16, n=286 | -0.2 (2.68)
  Albumin, Year 1, Week 24, n=292 | 0.2 (2.74)
  Albumin, Year 1, Week 32, n=287 | 0.1 (2.91)
  Albumin, Year 1, Week 40, n=284 | 0.2 (3.06)
  Albumin, Year 1, Week 48, n=287 | 0.3 (3.21)
  Albumin, Year 2, Week 8, n=288 | 0.4 (2.84)
  Albumin, Year 2, Week 16, n=278 | 0.4 (2.95)
  Albumin, Year 2, Week 24, n=273 | 0.1 (3.17)
  Albumin, Year 2, Week 32, n=284 | 0.7 (3.08)
  Albumin, Year 2, Week 40, n=264 | 0.8 (2.92)
  Albumin, Year 2, Week 48, n=269 | 1.1 (3.25)
  Albumin, Year 3, Week 8, n=265 | 0.7 (3.39)
  Albumin, Year 3, Week 16, n=260 | 1.0 (3.05)
  Albumin, Year 3, Week 24, n=244 | 1.2 (3.23)
  Albumin, Year 3, Week 32, n=249 | 1.3 (3.13)
  Albumin, Year 3, Week 40, n=245 | 1.4 (3.11)
  Albumin, Year 3, Week 48, n=244 | 1.5 (3.12)
  Albumin, Year 4, Week 8, n=239 | 1.4 (3.36)
  Albumin, Year 4, Week 16, n=238 | 1.3 (3.21)
  Albumin, Year 4, Week 24, n=227 | 1.2 (3.15)
  Albumin, Year 4, Week 32, n=233 | 1.3 (3.31)
  Albumin, Year 4, Week 40, n=220 | 1.2 (3.29)
  Albumin, Year 4, Week 48, n=218 | 1.6 (3.57)
  Albumin, Year 5, Week 8, n=218 | 1.6 (3.37)
  Albumin, Year 5, Week 16, n=214 | 1.5 (3.07)
  Albumin, Year 5, Week 24, n=211 | 1.5 (3.36)
  Albumin, Year 5, Week 32, n=211 | 1.9 (3.34)
  Albumin, Year 5, Week 40, n=198 | 1.8 (3.40)
  Albumin, Year 5, Week 48, n=207 | 1.7 (3.41)
  Albumin, Year 6, Week 8, n=206 | 1.8 (3.27)
  Albumin, Year 6, Week 16, n=198 | 1.5 (3.72)
  Albumin, Year 6, Week 24, n=190 | 1.6 (3.32)
  Albumin, Year 6, Week 32, n=193 | 2.0 (3.71)
  Albumin, Year 6, Week 40, n=185 | 1.9 (3.52)
  Albumin, Year 6, Week 48, n=186 | 1.9 (3.64)
  Albumin, Year 7, Week 8, n=179 | 1.9 (3.36)
  Albumin, Year 7, Week 16, n=179 | 1.7 (3.57)
  Albumin, Year 7, Week 24, n=173 | 1.7 (3.88)
  Albumin, Year 7, Week 32, n=180 | 1.9 (3.53)
  Albumin, Year 7, Week 40, n=175 | 1.6 (3.41)
  Albumin, Year 7, Week 48, n=175 | 1.6 (3.60)
  Albumin, Year 8, Week 8, n=171 | 1.7 (3.61)
  Albumin, Year 8, Week 16, n=170 | 1.5 (3.31)
  Albumin, Year 8, Week 24, n=168 | 1.6 (3.47)
  Albumin, Year 8, Week 32, n=168 | 1.7 (3.25)
  Albumin, Year 8, Week 40, n=162 | 1.3 (3.46)
  Albumin, Year 8, Week 48, n=159 | 1.7 (3.56)
  Albumin, Year 9, Week 8, n=164 | 2.0 (3.97)
  Albumin, Year 9, Week 16, n=162 | 1.9 (3.58)
  Albumin, Year 9, Week 24, n=161 | 1.6 (3.38)
  Albumin, Year 9, Week 32, n=163 | 1.9 (3.27)
  Albumin, Year 9, Week 40, n=156 | 1.6 (3.54)
  Albumin, Year 9, Week 48, n=151 | 1.9 (3.55)
  Albumin, Year 10, Week 8, n=152 | 1.9 (3.64)
  Albumin, Year 10, Week 16, n=143 | 2.1 (3.55)
  Albumin, Year 10, Week 24, n=145 | 2.0 (3.85)
  Albumin, Year 10, Week 32, n=142 | 2.1 (4.05)
  Albumin, Year 10, Week 40, n=138 | 1.8 (3.78)
  Albumin, Year 10, Week 48, n=135 | 2.0 (3.52)
  Albumin, Year 11, Week 8, n=138 | 2.0 (3.74)
  Albumin, Year 11, Week 16, n=128 | 2.2 (3.58)
  Albumin, Year 11, Week 24, n=130 | 2.1 (3.87)
  Albumin, Year 11, Week 32, n=125 | 1.8 (3.89)
  Albumin, Year 11, Week 40, n=124 | 1.7 (3.69)
  Albumin, Year 11, Week 48, n=108 | 1.8 (3.91)
  Albumin, Year 12, Week 8, n=110 | 1.8 (3.43)
  Albumin, Year 12, Week 16, n=97 | 1.9 (3.68)
  Albumin, Year 12, Week 24, n=87 | 2.5 (4.01)
  Albumin, Year 12, Week 32, n=84 | 1.9 (4.01)
  Albumin, Year 12, Week 40, n=82 | 1.7 (3.76)
  Albumin, Year 12, Week 48, n=72 | 2.1 (3.67)
  Albumin, Year 13, Week 8, n=53 | 2.8 (3.68)
  Albumin, Year 13, Week 16, n=42 | 2.3 (3.61)
  Albumin, Year 13, Week 24, n=20 | 2.5 (3.30)
  Albumin, Year 13, Week 32, n=7 | 1.1 (2.67)
  Albumin, Year 13, Week 40, n=1 | 5.0 (NA) — No value as only one participant was analyzed.
  Albumin, Exit, n=248 | 2.0 (4.02)
  Albumin, 8-Week Follow-up, n=220 | 1.6 (3.92)
  Albumin, 24-Week Follow-up , n=200 | 2.2 (4.24)
  Protein, Year 1, Week 8, n=284 | -1.3 (4.31)
  Protein, Year 1, Week 16, n=286 | -1.8 (4.63)
  Protein, Year 1, Week 24, n=292 | -1.5 (4.76)
  Protein, Year 1, Week 32, n=287 | -1.7 (4.69)
  Protein, Year 1, Week 40, n=284 | -1.6 (5.0)
  Protein, Year 1, Week 48, n=287 | -2.0 (5.01)
  Protein, Year 2, Week 8, n=288 | -2.1 (4.74)
  Protein, Year 2, Week 16, n=278 | -2.5 (4.66)
  Protein, Year 2, Week 24, n=273 | -2.9 (5.07)
  Protein, Year 2, Week 32, n=284 | -2.4 (5.13)
  Protein, Year 2, Week 40, n=264 | -2.4 (4.87)
  Protein, Year 2, Week 48, n=269 | -1.5 (5.18)
  Protein, Year 3, Week 8, n=265 | -2.2 (5.49)
  Protein, Year 3, Week 16, n=260 | -2.0 (5.19)
  Protein, Year 3, Week 24, n=244 | -1.9 (5.63)
  Protein, Year 3, Week 32, n=249 | -1.8 (5.19)
  Protein, Year 3, Week 40, n=245 | -1.6 (5.34)
  Protein, Year 3, Week 48, n=244 | -1.8 (5.16)
  Protein, Year 4, Week 8, n=239 | -2.1 (5.27)
  Protein, Year 4, Week 16, n=238 | -1.8 (4.93)
  Protein, Year 4, Week 24, n=227 | -2.5 (5.06)
  Protein, Year 4, Week 32, n=233 | -2.3 (5.02)
  Protein, Year 4, Week 40, n=220 | -2.8 (4.97)
  Protein, Year 4, Week 48, n=218 | -2.2 (5.44)
  Protein, Year 5, Week 8, n=218 | -2.5 (5.34)
  Protein, Year 5, Week 16, n=214 | -2.6 (5.09)
  Protein, Year 5, Week 24, n=211 | -3.2 (5.22)
  Protein, Year 5, Week 32, n=211 | -2.5 (5.05)
  Protein, Year 5, Week 40, n=198 | -2.9 (5.47)
  Protein, Year 5, Week 48, n=207 | -2.8 (5.67)
  Protein, Year 6, Week 8, n=206 | -3.1 (5.39)
  Protein, Year 6, Week 16, n=198 | -3.4 (5.75)
  Protein, Year 6, Week 24, n=190 | -3.5 (5.6)
  Protein, Year 6, Week 32, n=193 | -3.0 (5.77)
  Protein, Year 6, Week 40, n=185 | -3.4 (5.84)
  Protein, Year 6, Week 48, n=186 | -3.5 (6.0)
  Protein, Year 7, Week 8, n=179 | -3.6 (5.52)
  Protein, Year 7, Week 16, n=179 | -4.1 (5.87)
  Protein, Year 7, Week 24, n=173 | -3.9 (5.96)
  Protein, Year 7, Week 32, n=180 | -3.7 (5.68)
  Protein, Year 7, Week 40, n=175 | -4.2 (5.39)
  Protein, Year 7, Week 48, n=175 | -4.5 (5.6)
  Protein, Year 8, Week 8, n=171 | -4.6 (5.75)
  Protein, Year 8, Week 16, n=170 | -4.7 (5.37)
  Protein, Year 8, Week 24, n=168 | -4.7 (5.54)
  Protein, Year 8, Week 32, n=168 | -4.5 (5.46)
  Protein, Year 8, Week 40, n=162 | -5.2 (5.36)
  Protein, Year 8, Week 48, n=159 | -4.5 (5.3)
  Protein, Year 9, Week 8, n=164 | -4.5 (5.75)
  Protein, Year 9, Week 16, n=162 | -4.8 (5.34)
  Protein, Year 9, Week 24, n=161 | -5.0 (5.32)
  Protein, Year 9, Week 32, n=163 | -4.8 (5.18)
  Protein, Year 9, Week 40, n=156 | -5.4 (5.51)
  Protein, Year 9, Week 48, n=151 | -5.1 (5.6)
  Protein, Year 10, Week 8, n=152 | -5.2 (5.86)
  Protein, Year 10, Week 16, n=143 | -5.0 (5.79)
  Protein, Year 10, Week 24, n=145 | -5.2 (5.88)
  Protein, Year 10, Week 32, n=142 | -5.1 (5.98)
  Protein, Year 10, Week 40, n=138 | -5.4 (5.98)
  Protein, Year 10, Week 48, n=135 | -5.4 (5.62)
  Protein, Year 11, Week 8, n=138 | -5.4 (6.15)
  Protein, Year 11, Week 16, n=128 | -5.1 (5.51)
  Protein, Year 11, Week 24, n=130 | -5.1 (6.15)
  Protein, Year 11, Week 32, n=125 | -5.6 (6.12)
  Protein, Year 11, Week 40, n=124 | -5.6 (5.81)
  Protein, Year 11, Week 48, n=108 | -5.4 (6.42)
  Protein, Year 12, Week 8, n=110 | -5.0 (5.65)
  Protein, Year 12, Week 16, n=97 | -5.1 (5.86)
  Protein, Year 12, Week 24, n=87 | -4.6 (6.26)
  Protein, Year 12, Week 32, n=84 | -5.1 (5.82)
  Protein, Year 12, Week 40, n=82 | -5.7 (5.35)
  Protein, Year 12, Week 48, n=72 | -5.0 (5.86)
  Protein, Year 13, Week 8, n=53 | -4.8 (6.0)
  Protein, Year 13, Week 16, n=42 | -5.6 (6.04)
  Protein, Year 13, Week 24, n=20 | -4.4 (6.3)
  Protein, Year 13, Week 32, n=7 | -8.9 (5.08)
  Protein, Year 13, Week 40, n=1 | 1.0 (NA) — No value as only one participant was analyzed.
  Protein, Exit, n=248 | -3.2 (6.12)
  Protein, 8-Week Follow-up, n=220 | -3.7 (6.39)
  Protein, 24-Week Follow-up , n=200 | -2.6 (6.72)

10. Primary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN), Glucose, Calcium, Carbon Dioxide, Chloride, Magnesium, Phosphate, Potassium and Sodium at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in BUN, glucose, calcium, carbon dioxide, chloride, magnesium, phosphate, potassium and sodium is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
millimoles per liter
  BUN, Year 1, Week 8, n=284 | 0.0189 (1.4412)
  BUN, Year 1, Week 16, n=286 | -0.0836 (1.4928)
  BUN, Year 1, Week 24, n=292 | -0.0281 (1.5612)
  BUN, Year 1, Week 32, n=287 | -0.0199 (1.4020)
  BUN, Year 1, Week 40, n=284 | -0.1823 (1.3626)
  BUN, Year 1, Week 48, n=287 | 0.0224 (1.6607)
  BUN, Year 2, Week 8, n=288 | -0.0607 (1.5714)
  BUN, Year 2, Week 16, n=278 | -0.0796 (1.6220)
  BUN, Year 2, Week 24, n=273 | -0.0850 (1.6900)
  BUN, Year 2, Week 32, n=284 | -0.0779 (1.8263)
  BUN, Year 2, Week 40, n=264 | -0.1136 (1.7293)
  BUN, Year 2, Week 48, n=269 | -0.0571 (1.7035)
  BUN, Year 3, Week 8, n=265 | -0.0620 (1.6580)
  BUN, Year 3, Week 16, n=260 | -0.0357 (1.7963)
  BUN, Year 3, Week 24, n=244 | 0.0775 (1.9949)
  BUN, Year 3, Week 32, n=249 | 0.0129 (1.8758)
  BUN, Year 3, Week 40, n=245 | 0.0903 (1.9922)
  BUN, Year 3, Week 48, n=244 | 0.1346 (2.1131)
  BUN, Year 4, Week 8, n=239 | 0.1658 (1.9076)
  BUN, Year 4, Week 16, n=238 | 0.0900 (1.7799)
  BUN, Year 4, Week 24, n=227 | 0.1258 (2.0386)
  BUN, Year 4, Week 32, n=233 | 0.0812 (1.8611)
  BUN, Year 4, Week 40, n=220 | 0.0325 (2.0164)
  BUN, Year 4, Week 48, n=218 | 0.2948 (2.3008)
  BUN, Year 5, Week 8, n=218 | 0.2047 (2.0007)
  BUN, Year 5, Week 16, n=214 | 0.2669 (1.8316)
  BUN, Year 5, Week 24, n=211 | 0.2064 (2.0558)
  BUN, Year 5, Week 32, n=211 | 0.0558 (1.7962)
  BUN, Year 5, Week 40, n=198 | 0.2632 (2.0944)
  BUN, Year 5, Week 48, n=207 | 0.1794 (2.0505)
  BUN, Year 6, Week 8, n=206 | 0.2773 (1.8758)
  BUN, Year 6, Week 16, n=198 | 0.2632 (1.8983)
  BUN, Year 6, Week 24, n=190 | 0.1447 (2.0291)
  BUN, Year 6, Week 32, n=193 | 0.2960 (2.1213)
  BUN, Year 6, Week 40, n=185 | 0.3184 (2.1795)
  BUN, Year 6, Week 48, n=186 | 0.3647 (1.9359)
  BUN, Year 7, Week 8, n=179 | 0.2852 (2.1528)
  BUN, Year 7, Week 16, n=179 | 0.3191 (2.0398)
  BUN, Year 7, Week 24, n=173 | 0.2683 (2.5539)
  BUN, Year 7, Week 32, n=180 | 0.1686 (2.1547)
  BUN, Year 7, Week 40, n=175 | 0.2285 (1.9007)
  BUN, Year 7, Week 48, n=175 | 0.2326 (2.3098)
  BUN, Year 8, Week 8, n=171 | 0.2234 (2.3330)
  BUN, Year 8, Week 16, n=170 | 0.1932 (2.1219)
  BUN, Year 8, Week 24, n=168 | 0.2189 (2.0413)
  BUN, Year 8, Week 32, n=168 | 0.0680 (2.0995)
  BUN, Year 8, Week 40, n=162 | 0.1234 (2.0504)
  BUN, Year 8, Week 48, n=159 | 0.2560 (1.8494)
  BUN, Year 9, Week 8, n=164 | 0.1197 (1.6667)
  BUN, Year 9, Week 16, n=162 | 0.1719 (1.8226)
  BUN, Year 9, Week 24, n=161 | 0.1397 (1.9255)
  BUN, Year 9, Week 32, n=163 | 0.2979 (1.9020)
  BUN, Year 9, Week 40, n=156 | 0.1304 (1.8027)
  BUN, Year 9, Week 48, n=151 | 0.0804 (1.9432)
  BUN, Year 10, Week 8, n=152 | 0.1973 (2.1517)
  BUN, Year 10, Week 16, n=143 | 0.1098 (1.8916)
  BUN, Year 10, Week 24, n=145 | 0.1847 (1.8330)
  BUN, Year 10, Week 32, n=142 | 0.1911 (1.8808)
  BUN, Year 10, Week 40, n=138 | -0.0440 (1.8103)
  BUN, Year 10, Week 48, n=135 | 0.0926 (1.8219)
  BUN, Year 11, Week 8, n=138 | 0.1837 (2.0925)
  BUN, Year 11, Week 16, n=128 | 0.1060 (1.9866)
  BUN, Year 11, Week 24, n=130 | 0.1291 (1.8654)
  BUN, Year 11, Week 32, n=125 | 0.0029 (1.7563)
  BUN, Year 11, Week 40, n=124 | 0.0576 (1.9364)
  BUN, Year 11, Week 48, n=108 | -0.0926 (1.8134)
  BUN, Year 12, Week 8, n=110 | 0.1266 (2.0325)
  BUN, Year 12, Week 16, n=97 | 0.2687 (1.9561)
  BUN, Year 12, Week 24, n=87 | 0.0780 (1.8996)
  BUN, Year 12, Week 32, n=84 | -0.2167 (1.6336)
  BUN, Year 12, Week 40, n=82 | -0.1741 (1.8725)
  BUN, Year 12, Week 48, n=72 | -0.0992 (1.8146)
  BUN, Year 13, Week 8, n=53 | 0.0808 (1.7244)
  BUN, Year 13, Week 16, n=42 | 0.5695 (1.6690)
  BUN, Year 13, Week 24, n=20 | 0.1964 (1.0708)
  BUN, Year 13, Week 32, n=7 | -0.4590 (1.6961)
  BUN, Year 13, Week 40, n=1 | -1.7850 (NA) — No value as only one participant was analyzed.
  BUN, Exit, n=248 | 0.2519 (2.3492)
  BUN, 8-Week Follow-up, n=220 | 0.0471 (2.3709)
  BUN, 24-Week Follow-up , n=200 | -0.0268 (2.1652)
  Glucose, Year 1, Week 8, n=284 | -0.0264 (1.4683)
  Glucose, Year 1, Week 16, n=286 | 0.0314 (1.5221)
  Glucose, Year 1, Week 24, n=292 | -0.0375 (1.6213)
  Glucose, Year 1, Week 32, n=287 | -0.0265 (1.6241)
  Glucose, Year 1, Week 40, n=284 | 0.0031 (1.4590)
  Glucose, Year 1, Week 48, n=287 | 0.0232 (1.8176)
  Glucose, Year 2, Week 8, n=288 | 0.0168 (1.6196)
  Glucose, Year 2, Week 16, n=278 | 0.0327 (1.6027)
  Glucose, Year 2, Week 24, n=273 | 0.1194 (1.6450)
  Glucose, Year 2, Week 32, n=284 | 0.0510 (1.4905)
  Glucose, Year 2, Week 40, n=264 | 0.0639 (1.5995)
  Glucose, Year 2, Week 48, n=269 | 0.0017 (1.6178)
  Glucose, Year 3, Week 8, n=265 | -0.0161 (1.3878)
  Glucose, Year 3, Week 16, n=260 | -0.1223 (1.5965)
  Glucose, Year 3, Week 24, n=244 | 0.0348 (1.9713)
  Glucose, Year 3, Week 32, n=249 | -0.0887 (1.7057)
  Glucose, Year 3, Week 40, n=245 | -0.0242 (1.3532)
  Glucose, Year 3, Week 48, n=244 | -0.0271 (2.1535)
  Glucose, Year 4, Week 8, n=239 | -0.0451 (1.6912)
  Glucose, Year 4, Week 16, n=238 | -0.1199 (1.7495)
  Glucose, Year 4, Week 24, n=227 | -0.1142 (1.8087)
  Glucose, Year 4, Week 32, n=233 | 0.0741 (1.7592)
  Glucose, Year 4, Week 40, n=220 | 0.1204 (2.0200)
  Glucose, Year 4, Week 48, n=218 | -0.0410 (1.9212)
  Glucose, Year 5, Week 8, n=218 | 0.1350 (1.8331)
  Glucose, Year 5, Week 16, n=214 | 0.0999 (1.9373)
  Glucose, Year 5, Week 24, n=211 | 0.2402 (1.7548)
  Glucose, Year 5, Week 32, n=211 | -0.0873 (1.5258)
  Glucose, Year 5, Week 40, n=198 | 0.0535 (1.7957)
  Glucose, Year 5, Week 48, n=207 | -0.0107 (1.3758)
  Glucose, Year 6, Week 8, n=206 | 0.0385 (2.0336)
  Glucose, Year 6, Week 16, n=198 | 0.0112 (1.6676)
  Glucose, Year 6, Week 24, n=190 | 0.0894 (2.1875)
  Glucose, Year 6, Week 32, n=193 | 0.0380 (1.9025)
  Glucose, Year 6, Week 40, n=185 | 0.0939 (1.9242)
  Glucose, Year 6, Week 48, n=186 | -0.0176 (1.7507)
  Glucose, Year 7, Week 8, n=179 | 0.1098 (1.9999)
  Glucose, Year 7, Week 16, n=179 | 0.0558 (2.0164)
  Glucose, Year 7, Week 24, n=173 | 0.2118 (2.3731)
  Glucose, Year 7, Week 32, n=180 | 0.1588 (1.6939)
  Glucose, Year 7, Week 40, n=175 | 0.1380 (2.1777)
  Glucose, Year 7, Week 48, n=175 | 0.0698 (1.9178)
  Glucose, Year 8, Week 8, n=171 | 0.0217 (2.0227)
  Glucose, Year 8, Week 16, n=170 | 0.0307 (1.9951)
  Glucose, Year 8, Week 24, n=168 | 0.0430 (1.5670)
  Glucose, Year 8, Week 32, n=168 | 0.2029 (2.1886)
  Glucose, Year 8, Week 40, n=162 | 0.3481 (1.8895)
  Glucose, Year 8, Week 48, n=159 | 0.2821 (2.3294)
  Glucose, Year 9, Week 8, n=164 | 0.2065 (2.3063)
  Glucose, Year 9, Week 16, n=162 | 0.2457 (2.2362)
  Glucose, Year 9, Week 24, n=161 | 0.2065 (2.3096)
  Glucose, Year 9, Week 32, n=163 | 0.1437 (1.7266)
  Glucose, Year 9, Week 40, n=156 | 0.2619 (2.4664)
  Glucose, Year 9, Week 48, n=151 | 0.3110 (1.7497)
  Glucose, Year 10, Week 8, n=152 | 0.2184 (2.5367)
  Glucose, Year 10, Week 16, n=143 | 0.2713 (2.2189)
  Glucose, Year 10, Week 24, n=145 | 0.2695 (1.9119)
  Glucose, Year 10, Week 32, n=142 | 0.0192 (2.0309)
  Glucose, Year 10, Week 40, n=138 | 0.2277 (1.8718)
  Glucose, Year 10, Week 48, n=135 | 0.2919 (2.2420)
  Glucose, Year 11, Week 8, n=138 | 0.3524 (2.4257)
  Glucose, Year 11, Week 16, n=128 | 0.1778 (2.4430)
  Glucose, Year 11, Week 24, n=130 | 0.2818 (1.9155)
  Glucose, Year 11, Week 32, n=125 | 0.2203 (2.2945)
  Glucose, Year 11, Week 40, n=124 | 0.0877 (2.0564)
  Glucose, Year 11, Week 48, n=108 | 0.1778 (2.2984)
  Glucose, Year 12, Week 8, n=110 | 0.2861 (2.5700)
  Glucose, Year 12, Week 16, n=97 | 0.0830 (2.1347)
  Glucose, Year 12, Week 24, n=87 | 0.1448 (1.8433)
  Glucose, Year 12, Week 32, n=84 | -0.0886 (2.2813)
  Glucose, Year 12, Week 40, n=82 | 0.3209 (1.4176)
  Glucose, Year 12, Week 48, n=72 | 0.3870 (1.4519)
  Glucose, Year 13, Week 8, n=53 | 0.3561 (1.1963)
  Glucose, Year 13, Week 16, n=42 | 0.2498 (1.2196)
  Glucose, Year 13, Week 24, n=20 | 0.4663 (1.6396)
  Glucose, Year 13, Week 32, n=7 | 0.3727 (0.8144)
  Glucose, Year 13, Week 40, n=1 | -0.8326 (NA) — No value as only one participant was analyzed.
  Glucose, Exit, n=248 | 0.1744 (1.9656)
  Glucose, 8-Week Follow-up, n=220 | 0.2707 (1.5879)
  Glucose, 24-Week Follow-up , n=200 | 0.3295 (2.1561)
  Calcium, Year 1, Week 8, n=281 | -0.0033 (0.1012)
  Calcium, Year 1, Week 16, n=283 | -0.0025 (0.1175)
  Calcium, Year 1, Week 24, n=287 | 0.0156 (0.1036)
  Calcium, Year 1, Week 32, n=283 | 0.0159 (0.1067)
  Calcium, Year 1, Week 40, n=282 | 0.0203 (0.1102)
  Calcium, Year 1, Week 48, n=284 | 0.0011 (0.1193)
  Calcium, Year 2, Week 8, n=288 | 0.0010 (0.1093)
  Calcium, Year 2, Week 16, n=276 | -0.0080 (0.1104)
  Calcium, Year 2, Week 24, n=269 | -0.0180 (0.1171)
  Calcium, Year 2, Week 32, n=284 | -0.0131 (0.1120)
  Calcium, Year 2, Week 40, n=261 | -0.0071 (0.1091)
  Calcium, Year 2, Week 48, n=267 | -0.0081 (0.1158)
  Calcium, Year 3, Week 8, n=262 | -0.0273 (0.1291)
  Calcium, Year 3, Week 16, n=258 | -0.0189 (0.1102)
  Calcium, Year 3, Week 24, n=241 | -0.0205 (0.1165)
  Calcium, Year 3, Week 32, n=245 | -0.0205 (0.1044)
  Calcium, Year 3, Week 40, n=242 | -0.0121 (0.1122)
  Calcium, Year 3, Week 48, n=239 | -0.0156 (0.1112)
  Calcium, Year 4, Week 8, n=237 | -0.0183 (0.1147)
  Calcium, Year 4, Week 16, n=235 | -0.0264 (0.1118)
  Calcium, Year 4, Week 24, n=225 | -0.0250 (0.1140)
  Calcium, Year 4, Week 32, n=230 | -0.0221 (0.1074)
  Calcium, Year 4, Week 40, n=218 | -0.0220 (0.1105)
  Calcium, Year 4, Week 48, n=214 | -0.0192 (0.1162)
  Calcium, Year 5, Week 8, n=217 | -0.0297 (0.1112)
  Calcium, Year 5, Week 16, n=213 | -0.0274 (0.1149)
  Calcium, Year 5, Week 24, n=206 | -0.0292 (0.1179)
  Calcium, Year 5, Week 32, n=211 | -0.0104 (0.1132)
  Calcium, Year 5, Week 40, n=196 | -0.0140 (0.1166)
  Calcium, Year 5, Week 48, n=207 | -0.0036 (0.1133)
  Calcium, Year 6, Week 8, n=205 | -0.0127 (0.1086)
  Calcium, Year 6, Week 16, n=198 | -0.0263 (0.1269)
  Calcium, Year 6, Week 24, n=189 | -0.0037 (0.1155)
  Calcium, Year 6, Week 32, n=192 | -0.0044 (0.1150)
  Calcium, Year 6, Week 40, n=181 | -0.0123 (0.1068)
  Calcium, Year 6, Week 48, n=186 | -0.0025 (0.1107)
  Calcium, Year 7, Week 8, n=177 | -0.0162 (0.1076)
  Calcium, Year 7, Week 16, n=178 | -0.0175 (0.1217)
  Calcium, Year 7, Week 24, n=171 | -0.0163 (0.1169)
  Calcium, Year 7, Week 32, n=179 | -0.0114 (0.1097)
  Calcium, Year 7, Week 40, n=172 | -0.0144 (0.1111)
  Calcium, Year 7, Week 48, n=175 | -0.0234 (0.1058)
  Calcium, Year 8, Week 8, n=170 | -0.0203 (0.1144)
  Calcium, Year 8, Week 16, n=169 | -0.0176 (0.1099)
  Calcium, Year 8, Week 24, n=167 | -0.0121 (0.1047)
  Calcium, Year 8, Week 32, n=166 | -0.0153 (0.1015)
  Calcium, Year 8, Week 40, n=161 | -0.0254 (0.1111)
  Calcium, Year 8, Week 48, n=159 | -0.0210 (0.1138)
  Calcium, Year 9, Week 8, n=163 | -0.0167 (0.1283)
  Calcium, Year 9, Week 16, n=160 | -0.0198 (0.1181)
  Calcium, Year 9, Week 24, n=160 | -0.0253 (0.1231)
  Calcium, Year 9, Week 32, n=162 | -0.0205 (0.1150)
  Calcium, Year 9, Week 40, n=156 | -0.0157 (0.1246)
  Calcium, Year 9, Week 48, n=150 | -0.0075 (0.1116)
  Calcium, Year 10, Week 8, n=151 | -0.0114 (0.1050)
  Calcium, Year 10, Week 16, n=143 | 0.0026 (0.1015)
  Calcium, Year 10, Week 24, n=145 | -0.0067 (0.1115)
  Calcium, Year 10, Week 32, n=140 | -0.0066 (0.1109)
  Calcium, Year 10, Week 40, n=137 | -0.0067 (0.1157)
  Calcium, Year 10, Week 48, n=135 | -0.0033 (0.1268)
  Calcium, Year 11, Week 8, n=138 | -0.0043 (0.1185)
  Calcium, Year 11, Week 16, n=128 | -0.0033 (0.1078)
  Calcium, Year 11, Week 24, n=129 | -0.0116 (0.1304)
  Calcium, Year 11, Week 32, n=124 | -0.0131 (0.1131)
  Calcium, Year 11, Week 40, n=124 | -0.0093 (0.1157)
  Calcium, Year 11, Week 48, n=107 | -0.0061 (0.1238)
  Calcium, Year 12, Week 8, n=109 | -0.0153 (0.1214)
  Calcium, Year 12, Week 16, n=97 | -0.0005 (0.1189)
  Calcium, Year 12, Week 24, n=85 | 0.0220 (0.1251)
  Calcium, Year 12, Week 32, n=84 | 0.0009 (0.1265)
  Calcium, Year 12, Week 40, n=82 | -0.0103 (0.1247)
  Calcium, Year 12, Week 48, n=72 | -0.0028 (0.1206)
  Calcium, Year 13, Week 8, n=53 | -0.0151 (0.1402)
  Calcium, Year 13, Week 16, n=42 | -0.0154 (0.1595)
  Calcium, Year 13, Week 24, n=20 | 0.0037 (0.1435)
  Calcium, Year 13, Week 32, n=7 | -0.0784 (0.1234)
  Calcium, Year 13, Week 40, n=1 | 0.0000 (NA) — No value as only one participant was analyzed.
  Calcium, Exit, n=248 | 0.0141 (0.1239)
  Calcium, 8-Week Follow-up, n=220 | 0.0082 (0.1152)
  Calcium, 24-Week Follow-up , n=200 | 0.0181 (0.1211)
  Carbon dioxide, Year 1, Week 8, n=281 | 0.2 (2.54)
  Carbon dioxide, Year 1, Week 16, n=283 | 0.7 (2.73)
  Carbon dioxide, Year 1, Week 24, n=287 | 0.9 (2.78)
  Carbon dioxide, Year 1, Week 32, n=283 | 1.0 (2.51)
  Carbon dioxide, Year 1, Week 40, n=282 | 1.0 (2.75)
  Carbon dioxide, Year 1, Week 48, n=284 | 1.3 (2.71)
  Carbon dioxide, Year 2, Week 8, n=288 | 1.0 (2.74)
  Carbon dioxide, Year 2, Week 16, n=275 | 1.2 (2.74)
  Carbon dioxide, Year 2, Week 24, n=269 | 1.2 (2.96)
  Carbon dioxide, Year 2, Week 32, n=284 | 1.3 (2.77)
  Carbon dioxide, Year 2, Week 40, n=261 | 1.1 (2.72)
  Carbon dioxide, Year 2, Week 48, n=267 | 1.7 (3.02)
  Carbon dioxide, Year 3, Week 8, n=262 | 1.3 (2.83)
  Carbon dioxide, Year 3, Week 16, n=258 | 1.5 (2.95)
  Carbon dioxide, Year 3, Week 24, n=241 | 1.0 (2.81)
  Carbon dioxide, Year 3, Week 32, n=245 | 1.1 (2.96)
  Carbon dioxide, Year 3, Week 40, n=242 | 1.0 (2.94)
  Carbon dioxide, Year 3, Week 48, n=239 | 1.3 (3.29)
  Carbon dioxide, Year 4, Week 8, n=237 | 1.1 (2.81)
  Carbon dioxide, Year 4, Week 16, n=235 | 1.3 (3.04)
  Carbon dioxide, Year 4, Week 24, n=225 | 1.0 (2.84)
  Carbon dioxide, Year 4, Week 32, n=230 | 1.1 (2.90)
  Carbon dioxide, Year 4, Week 40, n=218 | 1.2 (3.11)
  Carbon dioxide, Year 4, Week 48, n=214 | 1.6 (3.17)
  Carbon dioxide, Year 5, Week 8, n=217 | 1.4 (2.93)
  Carbon dioxide, Year 5, Week 16, n=213 | 1.7 (2.93)
  Carbon dioxide, Year 5, Week 24, n=206 | 1.4 (2.82)
  Carbon dioxide, Year 5, Week 32, n=211 | 1.5 (2.98)
  Carbon dioxide, Year 5, Week 40, n=196 | 1.5 (2.91)
  Carbon dioxide, Year 5, Week 48, n=207 | 1.7 (2.82)
  Carbon dioxide, Year 6, Week 8, n=205 | 1.8 (3.10)
  Carbon dioxide, Year 6, Week 16, n=198 | 1.8 (2.94)
  Carbon dioxide, Year 6, Week 24, n=189 | 1.7 (2.77)
  Carbon dioxide, Year 6, Week 32, n=192 | 1.7 (2.82)
  Carbon dioxide, Year 6, Week 40, n=181 | 1.8 (3.07)
  Carbon dioxide, Year 6, Week 48, n=186 | 1.9 (2.97)
  Carbon dioxide, Year 7, Week 8, n=177 | 1.8 (3.12)
  Carbon dioxide, Year 7, Week 16, n=178 | 1.6 (3.11)
  Carbon dioxide, Year 7, Week 24, n=171 | 1.6 (3.08)
  Carbon dioxide, Year 7, Week 32, n=179 | 1.6 (3.10)
  Carbon dioxide, Year 7, Week 40, n=172 | 1.6 (2.83)
  Carbon dioxide, Year 7, Week 48, n=175 | 1.6 (2.97)
  Carbon dioxide, Year 8, Week 8, n=170 | 1.5 (3.00)
  Carbon dioxide, Year 8, Week 16, n=169 | 1.5 (3.17)
  Carbon dioxide, Year 8, Week 24, n=167 | 1.5 (3.08)
  Carbon dioxide, Year 8, Week 32, n=166 | 1.5 (3.27)
  Carbon dioxide, Year 8, Week 40, n=161 | 1.6 (3.32)
  Carbon dioxide, Year 8, Week 48, n=159 | 1.5 (3.25)
  Carbon dioxide, Year 9, Week 8, n=163 | 1.1 (3.26)
  Carbon dioxide, Year 9, Week 16, n=160 | 1.4 (3.08)
  Carbon dioxide, Year 9, Week 24, n=160 | 1.1 (2.93)
  Carbon dioxide, Year 9, Week 32, n=162 | 1.4 (3.13)
  Carbon dioxide, Year 9, Week 40, n=156 | 1.0 (3.30)
  Carbon dioxide, Year 9, Week 48, n=150 | 1.0 (3.16)
  Carbon dioxide, Year 10, Week 8, n=151 | 1.1 (2.95)
  Carbon dioxide, Year 10, Week 16, n=143 | 1.2 (3.14)
  Carbon dioxide, Year 10, Week 24, n=145 | 1.0 (3.14)
  Carbon dioxide, Year 10, Week 32, n=140 | 1.5 (3.12)
  Carbon dioxide, Year 10, Week 40, n=137 | 1.5 (3.21)
  Carbon dioxide, Year 10, Week 48, n=135 | 1.3 (3.03)
  Carbon dioxide, Year 11, Week 8, n=138 | 1.0 (3.13)
  Carbon dioxide, Year 11, Week 16, n=128 | 1.5 (3.04)
  Carbon dioxide, Year 11, Week 24, n=129 | 1.5 (3.13)
  Carbon dioxide, Year 11, Week 32, n=124 | 1.6 (2.99)
  Carbon dioxide, Year 11, Week 40, n=124 | 1.7 (3.03)
  Carbon dioxide, Year 11, Week 48, n=107 | 1.7 (3.10)
  Carbon dioxide, Year 12, Week 8, n=109 | 1.1 (3.12)
  Carbon dioxide, Year 12, Week 16, n=97 | 2.1 (3.05)
  Carbon dioxide, Year 12, Week 24, n=85 | 2.0 (3.12)
  Carbon dioxide, Year 12, Week 32, n=84 | 2.3 (3.58)
  Carbon dioxide, Year 12, Week 40, n=82 | 2.0 (3.26)
  Carbon dioxide, Year 12, Week 48, n=72 | 1.7 (3.39)
  Carbon dioxide, Year 13, Week 8, n=53 | 1.6 (2.90)
  Carbon dioxide, Year 13, Week 16, n=42 | 2.0 (2.76)
  Carbon dioxide, Year 13, Week 24, n=20 | 2.5 (3.19)
  Carbon dioxide, Year 13, Week 32, n=7 | 1.3 (3.59)
  Carbon dioxide, Year 13, Week 40, n=1 | 4.0 (NA) — No value as only one participant was analyzed.
  Carbon dioxide, Exit, n=248 | 1.8 (2.93)
  Carbon dioxide, 8-Week Follow-up, n=220 | 1.8 (3.26)
  Carbon dioxide, 24-Week Follow-up , n=200 | 1.8 (3.25)
  Chloride, Year 1, Week 8, n=284 | 0.1 (2.52)
  Chloride, Year 1, Week 16, n=286 | 0.4 (2.76)
  Chloride, Year 1, Week 24, n=292 | 0.0 (2.64)
  Chloride, Year 1, Week 32, n=287 | 0.0 (2.66)
  Chloride, Year 1, Week 40, n=284 | 0.0 (2.74)
  Chloride, Year 1, Week 48, n=287 | 0.4 (2.90)
  Chloride, Year 2, Week 8, n=288 | 0.2 (2.77)
  Chloride, Year 2, Week 16, n=278 | 0.4 (2.95)
  Chloride, Year 2, Week 24, n=273 | 0.6 (2.82)
  Chloride, Year 2, Week 32, n=284 | 0.4 (2.80)
  Chloride, Year 2, Week 40, n=264 | 0.3 (3.05)
  Chloride, Year 2, Week 48, n=269 | 0.2 (2.94)
  Chloride, Year 3, Week 8, n=265 | 0.3 (3.07)
  Chloride, Year 3, Week 16, n=260 | 0.0 (2.91)
  Chloride, Year 3, Week 24, n=244 | 0.1 (2.93)
  Chloride, Year 3, Week 32, n=249 | -0.1 (2.99)
  Chloride, Year 3, Week 40, n=245 | -0.2 (2.87)
  Chloride, Year 3, Week 48, n=244 | -0.3 (3.29)
  Chloride, Year 4, Week 8, n=239 | -0.2 (2.93)
  Chloride, Year 4, Week 16, n=238 | -0.2 (3.16)
  Chloride, Year 4, Week 24, n=227 | 0.1 (2.85)
  Chloride, Year 4, Week 32, n=233 | -0.3 (3.12)
  Chloride, Year 4, Week 40, n=220 | -0.4 (2.94)
  Chloride, Year 4, Week 48, n=218 | -0.3 (3.15)
  Chloride, Year 5, Week 8, n=218 | -0.1 (3.20)
  Chloride, Year 5, Week 16, n=214 | 0.1 (2.80)
  Chloride, Year 5, Week 24, n=211 | 0.2 (3.05)
  Chloride, Year 5, Week 32, n=211 | -0.2 (3.08)
  Chloride, Year 5, Week 40, n=198 | 0.1 (2.97)
  Chloride, Year 5, Week 48, n=207 | -0.3 (3.00)
  Chloride, Year 6, Week 8, n=206 | -0.2 (3.11)
  Chloride, Year 6, Week 16, n=198 | -0.2 (3.23)
  Chloride, Year 6, Week 24, n=190 | -0.2 (3.11)
  Chloride, Year 6, Week 32, n=193 | -0.4 (3.31)
  Chloride, Year 6, Week 40, n=185 | -0.3 (3.25)
  Chloride, Year 6, Week 48, n=186 | -0.4 (3.07)
  Chloride, Year 7, Week 8, n=179 | -0.3 (2.95)
  Chloride, Year 7, Week 16, n=179 | -0.3 (3.10)
  Chloride, Year 7, Week 24, n=173 | -0.2 (3.18)
  Chloride, Year 7, Week 32, n=180 | -0.3 (4.06)
  Chloride, Year 7, Week 40, n=175 | -0.4 (3.32)
  Chloride, Year 7, Week 48, n=175 | -0.4 (3.24)
  Chloride, Year 8, Week 8, n=171 | -0.3 (3.46)
  Chloride, Year 8, Week 16, n=170 | -0.5 (3.75)
  Chloride, Year 8, Week 24, n=168 | -0.5 (3.37)
  Chloride, Year 8, Week 32, n=168 | -0.6 (3.30)
  Chloride, Year 8, Week 40, n=162 | -0.4 (3.26)
  Chloride, Year 8, Week 48, n=159 | -0.4 (3.49)
  Chloride, Year 9, Week 8, n=164 | -0.7 (3.36)
  Chloride, Year 9, Week 16, n=162 | -0.7 (3.26)
  Chloride, Year 9, Week 24, n=161 | -0.3 (3.21)
  Chloride, Year 9, Week 32, n=163 | -0.6 (3.43)
  Chloride, Year 9, Week 40, n=156 | -0.3 (3.72)
  Chloride, Year 9, Week 48, n=151 | -0.6 (3.76)
  Chloride, Year 10, Week 8, n=152 | -0.6 (3.61)
  Chloride, Year 10, Week 16, n=143 | -0.7 (3.59)
  Chloride, Year 10, Week 24, n=145 | -0.3 (3.87)
  Chloride, Year 10, Week 32, n=142 | -0.3 (3.72)
  Chloride, Year 10, Week 40, n=138 | -0.2 (3.18)
  Chloride, Year 10, Week 48, n=135 | -0.2 (3.48)
  Chloride, Year 11, Week 8, n=138 | -0.1 (3.28)
  Chloride, Year 11, Week 16, n=128 | -0.4 (3.41)
  Chloride, Year 11, Week 24, n=130 | -0.5 (3.39)
  Chloride, Year 11, Week 32, n=125 | -0.7 (3.69)
  Chloride, Year 11, Week 40, n=124 | -0.4 (3.22)
  Chloride, Year 11, Week 48, n=108 | -0.4 (3.33)
  Chloride, Year 12, Week 8, n=110 | -0.3 (3.51)
  Chloride, Year 12, Week 16, n=97 | -0.6 (3.23)
  Chloride, Year 12, Week 24, n=87 | -0.3 (3.18)
  Chloride, Year 12, Week 32, n=84 | -0.4 (3.01)
  Chloride, Year 12, Week 40, n=82 | -0.4 (3.32)
  Chloride, Year 12, Week 48, n=72 | -1.3 (3.09)
  Chloride, Year 13, Week 8, n=53 | -0.8 (3.31)
  Chloride, Year 13, Week 16, n=42 | -0.8 (3.00)
  Chloride, Year 13, Week 24, n=20 | 0.0 (3.03)
  Chloride, Year 13, Week 32, n=7 | 1.1 (3.13)
  Chloride, Year 13, Week 40, n=1 | 0.0 (NA) — No value as only one participant was analyzed.
  Chloride, Exit, n=248 | -0.8 (3.38)
  Chloride, 8-Week Follow-up, n=220 | -0.8 (3.33)
  Chloride, 24-Week Follow-up, n=200 | -0.8 (3.52)
  Magnesium, Year 1, Week 8, n=284 | -0.003 (0.0646)
  Magnesium, Year 1, Week 16, n=286 | -0.006 (0.0707)
  Magnesium, Year 1, Week 24, n=292 | -0.002 (0.0660)
  Magnesium, Year 1, Week 32, n=287 | -0.007 (0.0680)
  Magnesium, Year 1, Week 40, n=284 | -0.007 (0.0657)
  Magnesium, Year 1, Week 48, n=287 | -0.017 (0.0724)
  Magnesium, Year 2, Week 8, n=288 | -0.016 (0.0694)
  Magnesium, Year 2, Week 16, n=278 | -0.015 (0.0723)
  Magnesium, Year 2, Week 24, n=273 | -0.020 (0.0704)
  Magnesium, Year 2, Week 32, n=284 | -0.018 (0.0642)
  Magnesium, Year 2, Week 40, n=264 | -0.018 (0.0699)
  Magnesium, Year 2, Week 48, n=269 | -0.021 (0.0720)
  Magnesium, Year 3, Week 8, n=265 | -0.029 (0.0709)
  Magnesium, Year 3, Week 16, n=260 | -0.027 (0.0672)
  Magnesium, Year 3, Week 24, n=244 | -0.040 (0.0646)
  Magnesium, Year 3, Week 32, n=249 | -0.042 (0.0742)
  Magnesium, Year 3, Week 40, n=245 | -0.054 (0.0712)
  Magnesium, Year 3, Week 48, n=244 | -0.051 (0.0724)
  Magnesium, Year 4, Week 8, n=239 | -0.052 (0.0692)
  Magnesium, Year 4, Week 16, n=238 | -0.049 (0.0764)
  Magnesium, Year 4, Week 24, n=227 | -0.046 (0.0720)
  Magnesium, Year 4, Week 32, n=233 | -0.049 (0.0709)
  Magnesium, Year 4, Week 40, n=220 | -0.053 (0.0702)
  Magnesium, Year 4, Week 48, n=218 | -0.050 (0.0757)
  Magnesium, Year 5, Week 8, n=218 | -0.052 (0.0676)
  Magnesium, Year 5, Week 16, n=214 | -0.054 (0.0633)
  Magnesium, Year 5, Week 24, n=211 | -0.062 (0.0648)
  Magnesium, Year 5, Week 32, n=211 | -0.068 (0.0700)
  Magnesium, Year 5, Week 40, n=198 | -0.063 (0.0709)
  Magnesium, Year 5, Week 48, n=207 | -0.067 (0.0754)
  Magnesium, Year 6, Week 8, n=206 | -0.059 (0.0724)
  Magnesium, Year 6, Week 16, n=198 | -0.067 (0.0786)
  Magnesium, Year 6, Week 24, n=190 | -0.065 (0.0724)
  Magnesium, Year 6, Week 32, n=193 | -0.063 (0.0712)
  Magnesium, Year 6, Week 40, n=185 | -0.060 (0.0750)
  Magnesium, Year 6, Week 48, n=186 | -0.068 (0.0721)
  Magnesium, Year 7, Week 8, n=179 | -0.052 (0.0746)
  Magnesium, Year 7, Week 16, n=179 | -0.058 (0.0711)
  Magnesium, Year 7, Week 24, n=173 | -0.056 (0.0712)
  Magnesium, Year 7, Week 32, n=180 | -0.054 (0.0747)
  Magnesium, Year 7, Week 40, n=175 | -0.050 (0.0826)
  Magnesium, Year 7, Week 48, n=175 | -0.057 (0.0772)
  Magnesium, Year 8, Week 8, n=171 | -0.052 (0.0761)
  Magnesium, Year 8, Week 16, n=170 | -0.060 (0.0748)
  Magnesium, Year 8, Week 24, n=168 | -0.051 (0.0739)
  Magnesium, Year 8, Week 32, n=168 | -0.055 (0.0777)
  Magnesium, Year 8, Week 40, n=162 | -0.050 (0.0737)
  Magnesium, Year 8, Week 48, n=159 | -0.047 (0.0788)
  Magnesium, Year 9, Week 8, n=164 | -0.049 (0.0793)
  Magnesium, Year 9, Week 16, n=162 | -0.047 (0.0776)
  Magnesium, Year 9, Week 24, n=161 | -0.052 (0.0825)
  Magnesium, Year 9, Week 32, n=163 | -0.052 (0.0771)
  Magnesium, Year 9, Week 40, n=156 | -0.048 (0.0840)
  Magnesium, Year 9, Week 48, n=151 | -0.056 (0.0771)
  Magnesium, Year 10, Week 8, n=152 | -0.050 (0.0795)
  Magnesium, Year 10, Week 16, n=143 | -0.054 (0.0772)
  Magnesium, Year 10, Week 24, n=145 | -0.055 (0.0770)
  Magnesium, Year 10, Week 32, n=142 | -0.050 (0.0750)
  Magnesium, Year 10, Week 40, n=138 | -0.055 (0.0798)
  Magnesium, Year 10, Week 48, n=135 | -0.055 (0.0825)
  Magnesium, Year 11, Week 8, n=138 | -0.057 (0.0823)
  Magnesium, Year 11, Week 16, n=128 | -0.055 (0.0809)
  Magnesium, Year 11, Week 24, n=130 | -0.055 (0.0810)
  Magnesium, Year 11, Week 32, n=125 | -0.055 (0.0889)
  Magnesium, Year 11, Week 40, n=124 | -0.044 (0.0842)
  Magnesium, Year 11, Week 48, n=108 | -0.057 (0.0800)
  Magnesium, Year 12, Week 8, n=110 | -0.041 (0.0855)
  Magnesium, Year 12, Week 16, n=97 | -0.047 (0.0797)
  Magnesium, Year 12, Week 24, n=87 | -0.040 (0.0846)
  Magnesium, Year 12, Week 32, n=84 | -0.056 (0.0808)
  Magnesium, Year 12, Week 40, n=82 | -0.049 (0.0909)
  Magnesium, Year 12, Week 48, n=72 | -0.047 (0.0809)
  Magnesium, Year 13, Week 8, n=53 | -0.045 (0.0834)
  Magnesium, Year 13, Week 16, n=42 | -0.046 (0.0752)
  Magnesium, Year 13, Week 24, n=20 | -0.055 (0.0776)
  Magnesium, Year 13, Week 32, n=7 | -0.050 (0.0500)
  Magnesium, Year 13, Week 40, n=1 | 0.050 (NA) — No value as only one participant was analyzed.
  Magnesium, Exit, n=248 | -0.037 (0.0793)
  Magnesium, 8-Week Follow-up, n=220 | -0.037 (0.0794)
  Magnesium, 24-Week Follow-up , n=200 | -0.040 (0.0790)
  Phosphate, Year 1, Week 8, n=284 | -0.0259 (0.1980)
  Phosphate, Year 1, Week 16, n=286 | -0.0215 (0.1849)
  Phosphate, Year 1, Week 24, n=292 | -0.0001 (0.2023)
  Phosphate, Year 1, Week 32, n=287 | -0.0154 (0.1983)
  Phosphate, Year 1, Week 40, n=284 | -0.0024 (0.1913)
  Phosphate, Year 1, Week 48, n=287 | -0.0234 (0.1926)
  Phosphate, Year 2, Week 8, n=288 | -0.0185 (0.1959)
  Phosphate, Year 2, Week 16, n=278 | -0.0194 (0.2003)
  Phosphate, Year 2, Week 24, n=273 | -0.0209 (0.1991)
  Phosphate, Year 2, Week 32, n=284 | -0.0318 (0.2122)
  Phosphate, Year 2, Week 40, n=264 | -0.0297 (0.2103)
  Phosphate, Year 2, Week 48, n=269 | -0.0116 (0.2050)
  Phosphate, Year 3, Week 8, n=265 | -0.04112 (0.2073)
  Phosphate, Year 3, Week 16, n=260 | -0.0451 (0.2059)
  Phosphate, Year 3, Week 24, n=244 | -0.0639 (0.2068)
  Phosphate, Year 3, Week 32, n=249 | -0.0484 (0.2139)
  Phosphate, Year 3, Week 40, n=245 | -0.0583 (0.2190)
  Phosphate, Year 3, Week 48, n=244 | -0.0658 (0.2179)
  Phosphate, Year 4, Week 8, n=239 | -0.0621 (0.2103)
  Phosphate, Year 4, Week 16, n=238 | -0.0532 (0.2217)
  Phosphate, Year 4, Week 24, n=227 | -0.0700 (0.2106)
  Phosphate, Year 4, Week 32, n=233 | -0.0601 (0.2034)
  Phosphate, Year 4, Week 40, n=220 | -0.0710 (0.2098)
  Phosphate, Year 4, Week 48, n=218 | -0.0400 (0.2213)
  Phosphate, Year 5, Week 8, n=218 | -0.0529 (0.2222)
  Phosphate, Year 5, Week 16, n=214 | -0.0429 (0.2240)
  Phosphate, Year 5, Week 24, n=211 | -0.0502 (0.1996)
  Phosphate, Year 5, Week 32, n=211 | -0.0435 (0.2313)
  Phosphate, Year 5, Week 40, n=198 | -0.0452 (0.2147)
  Phosphate, Year 5, Week 48, n=207 | -0.0323 (0.2167)
  Phosphate, Year 6, Week 8, n=206 | -0.0417 (0.2246)
  Phosphate, Year 6, Week 16, n=198 | -0.0354 (0.2253)
  Phosphate, Year 6, Week 24, n=190 | -0.0262 (0.2326)
  Phosphate, Year 6, Week 32, n=193 | -0.0341 (0.2154)
  Phosphate, Year 6, Week 40, n=185 | -0.0086 (0.2179)
  Phosphate, Year 6, Week 48, n=186 | -0.0085 (0.2256)
  Phosphate, Year 7, Week 8, n=179 | -0.0316 (0.2254)
  Phosphate, Year 7, Week 16, n=179 | -0.0372 (0.1999)
  Phosphate, Year 7, Week 24, n=173 | -0.0390 (0.2099)
  Phosphate, Year 7, Week 32, n=180 | -0.0321 (0.2099)
  Phosphate, Year 7, Week 40, n=175 | -0.0138 (0.2146)
  Phosphate, Year 7, Week 48, n=175 | -0.0400 (0.2031)
  Phosphate, Year 8, Week 8, n=171 | -0.0453 (0.2135)
  Phosphate, Year 8, Week 16, n=170 | -0.0319 (0.2088)
  Phosphate, Year 8, Week 24, n=168 | -0.0450 (0.2136)
  Phosphate, Year 8, Week 32, n=168 | -0.0530 (0.2073)
  Phosphate, Year 8, Week 40, n=162 | -0.0429 (0.2341)
  Phosphate, Year 8, Week 48, n=159 | -0.0266 (0.2158)
  Phosphate, Year 9, Week 8, n=164 | -0.0329 (0.2133)
  Phosphate, Year 9, Week 16, n=162 | -0.0255 (0.2140)
  Phosphate, Year 9, Week 24, n=161 | -0.0327 (0.2372)
  Phosphate, Year 9, Week 32, n=163 | -0.0487 (0.2039)
  Phosphate, Year 9, Week 40, n=156 | -0.0230 (0.2123)
  Phosphate, Year 9, Week 48, n=151 | -0.0385 (0.2170)
  Phosphate, Year 10, Week 8, n=152 | -0.0310 (0.2136)
  Phosphate, Year 10, Week 16, n=143 | -0.0458 (0.2087)
  Phosphate, Year 10, Week 24, n=145 | -0.0307 (0.2130)
  Phosphate, Year 10, Week 32, n=142 | -0.0241 (0.2227)
  Phosphate, Year 10, Week 40, n=138 | -0.0459 (0.2184)
  Phosphate, Year 10, Week 48, n=135 | -0.0335 (0.2158)
  Phosphate, Year 11, Week 8, n=138 | -0.0314 (0.2311)
  Phosphate, Year 11, Week 16, n=128 | -0.0560 (0.2327)
  Phosphate, Year 11, Week 24, n=130 | -0.0365 (0.2371)
  Phosphate, Year 11, Week 32, n=125 | -0.0302 (0.2140)
  Phosphate, Year 11, Week 40, n=124 | -0.0370 (0.2215)
  Phosphate, Year 11, Week 48, n=108 | -0.0287 (0.2361)
  Phosphate, Year 12, Week 8, n=110 | -0.0470 (0.2230)
  Phosphate, Year 12, Week 16, n=97 | -0.0333 (0.2264)
  Phosphate, Year 12, Week 24, n=87 | -0.0238 (0.2169)
  Phosphate, Year 12, Week 32, n=84 | -0.0488 (0.2235)
  Phosphate, Year 12, Week 40, n=82 | -0.0555 (0.2188)
  Phosphate, Year 12, Week 48, n=72 | -0.0341 (0.2213)
  Phosphate, Year 13, Week 8, n=53 | -0.0804 (0.2002)
  Phosphate, Year 13, Week 16, n=42 | -0.0461 (0.2669)
  Phosphate, Year 13, Week 24, n=20 | 0.0533 (0.1881)
  Phosphate, Year 13, Week 32, n=7 | 0.0784 (0.2075)
  Phosphate, Year 13, Week 40, n=1 | -0.1615 (NA) — No value as only one participant was analyzed.
  Phosphate, Exit, n=248 | -0.0328 (0.2385)
  Phosphate, 8-Week Follow-up, n=220 | -0.0631 (0.2221)
  Phosphate, 24-Week Follow-up , n=200 | -0.0375 (0.2183)
  Potassium, Year 1, Week 8, n=281 | -0.01 (0.354)
  Potassium, Year 1, Week 16, n=283 | 0.04 (0.394)
  Potassium, Year 1, Week 24, n=287 | 0.04 (0.406)
  Potassium, Year 1, Week 32, n=283 | 0.01 (0.381)
  Potassium, Year 1, Week 40, n=282 | 0.03 (0.378)
  Potassium, Year 1, Week 48, n=284 | 0.00 (0.406)
  Potassium, Year 2, Week 8, n=288 | 0.00 (0.370)
  Potassium, Year 2, Week 16, n=275 | 0.03 (0.385)
  Potassium, Year 2, Week 24, n=269 | 0.02 (0.398)
  Potassium, Year 2, Week 32, n=284 | 0.00 (0.397)
  Potassium, Year 2, Week 40, n=261 | 0.04 (0.378)
  Potassium, Year 2, Week 48, n=267 | 0.01 (0.386)
  Potassium, Year 3, Week 8, n=262 | 0.00 (0.415)
  Potassium, Year 3, Week 16, n=258 | 0.02 (0.413)
  Potassium, Year 3, Week 24, n=241 | 0.02 (0.407)
  Potassium, Year 3, Week 32, n=245 | -0.02 (0.406)
  Potassium, Year 3, Week 40, n=242 | 0.02 (0.428)
  Potassium, Year 3, Week 48, n=239 | 0.00 (0.400)
  Potassium, Year 4, Week 8, n=237 | 0.03 (0.414)
  Potassium, Year 4, Week 16, n=236 | 0.00 (0.423)
  Potassium, Year 4, Week 24, n=225 | 0.03 (0.400)
  Potassium, Year 4, Week 32, n=230 | 0.02 (0.383)
  Potassium, Year 4, Week 40, n=218 | -0.02 (0.396)
  Potassium, Year 4, Week 48, n=214 | 0.02 (0.391)
  Potassium, Year 5, Week 8, n=217 | 0.01 (0.413)
  Potassium, Year 5, Week 16, n=213 | 0.00 (0.390)
  Potassium, Year 5, Week 24, n=206 | 0.03 (0.420)
  Potassium, Year 5, Week 32, n=211 | -0.01 (0.393)
  Potassium, Year 5, Week 40, n=196 | 0.03 (0.416)
  Potassium, Year 5, Week 48, n=207 | -0.01 (0.375)
  Potassium, Year 6, Week 8, n=205 | -0.02 (0.424)
  Potassium, Year 6, Week 16, n=198 | -0.04 (0.429)
  Potassium, Year 6, Week 24, n=189 | 0.00 (0.411)
  Potassium, Year 6, Week 32, n=192 | -0.02 (0.395)
  Potassium, Year 6, Week 40, n=181 | 0.03 (0.435)
  Potassium, Year 6, Week 48, n=186 | -0.01 (0.388)
  Potassium,Year 7, Week 8, n=177 | 0.00 (0.424)
  Potassium, Year 7, Week 16, n=178 | -0.02 (0.412)
  Potassium, Year 7, Week 24, n=171 | 0.03 (0.388)
  Potassium, Year 7, Week 32, n=179 | 0.02 (0.406)
  Potassium, Year 7, Week 40, n=172 | 0.03 (0.453)
  Potassium, Year 7, Week 48, n=175 | -0.03 (0.403)
  Potassium, Year 8, Week 8, n=170 | -0.05 (0.426)
  Potassium, Year 8, Week 16, n=169 | -0.05 (0.455)
  Potassium, Year 8, Week 24, n=167 | 0.00 (0.386)
  Potassium, Year 8, Week 32, n=166 | -0.06 (0.382)
  Potassium, Year 8, Week 40, n=161 | 0.00 (0.401)
  Potassium, Year 8, Week 48, n=159 | -0.07 (0.377)
  Potassium, Year 9, Week 8, n=163 | -0.02 (0.448)
  Potassium, Year 9, Week 16, n=160 | -0.02 (0.385)
  Potassium, Year 9, Week 24, n=160 | -0.03 (0.391)
  Potassium, Year 9, Week 32, n=162 | -0.05 (0.391)
  Potassium, Year 9, Week 40, n=156 | -0.04 (0.447)
  Potassium, Year 9, Week 48, n=150 | -0.04 (0.432)
  Potassium, Year 10, Week 8, n=151 | -0.03 (0.417)
  Potassium, Year 10, Week 16, n=143 | -0.05 (0.415)
  Potassium, Year 10, Week 24, n=145 | 0.00 (0.428)
  Potassium, Year 10, Week 32, n=140 | -0.03 (0.452)
  Potassium, Year 10, Week 40, n=137 | -0.02 (0.433)
  Potassium, Year 10, Week 48, n=135 | -0.02 (0.442)
  Potassium, Year 11, Week 8, n=138 | -0.03 (0.438)
  Potassium, Year 11, Week 16, n=128 | -0.04 (0.395)
  Potassium, Year 11, Week 24, n=129 | 0.02 (0.433)
  Potassium, Year 11, Week 32, n=124 | -0.08 (0.399)
  Potassium, Year 11, Week 40, n=124 | -0.01 (0.383)
  Potassium, Year 11, Week 48, n=107 | 0.01 (0.413)
  Potassium, Year 12, Week 8, n=109 | 0.01 (0.422)
  Potassium, Year 12, Week 16, n=97 | -0.02 (0.433)
  Potassium, Year 12, Week 24, n=85 | 0.00 (0.447)
  Potassium, Year 12, Week 32, n=84 | -0.06 (0.443)
  Potassium, Year 12, Week 40, n=82 | -0.02 (0.411)
  Potassium, Year 12, Week 48, n=72 | -0.06 (0.527)
  Potassium, Year 13, Week 8, n=53 | -0.14 (0.401)
  Potassium, Year 13, Week 16, n=42 | -0.09 (0.416)
  Potassium, Year 13, Week 24, n=20 | 0.01 (0.525)
  Potassium, Year 13, Week 32, n=7 | -0.19 (0.389)
  Potassium, Year 13, Week 40, n=1 | 0.60 (NA) — No value as only one participant was analyzed.
  Potassium, Exit, n=248 | 0.03 (0.409)
  Potassium, 8-Week Follow-up, n=220 | 0.01 (0.415)
  Potassium, 24-Week Follow-up , n=200 | 0.02 (0.411)
  Sodium, Year 1, Week 8, n=284 | 0.1 (2.76)
  Sodium, Year 1, Week 16, n=286 | 0.2 (2.91)
  Sodium, ,Year 1, Week 24, n=292 | 0.0 (2.78)
  Sodium, Year 1, Week 32, n=287 | 0.0 (2.83)
  Sodium, Year 1, Week 40, n=284 | -0.2 (2.64)
  Sodium, Year 1, Week 48, n=287 | -0.1 (2.75)
  Sodium, Year 2, Week 8, n=288 | 0.0 (2.64)
  Sodium, Year 2, Week 16, n=278 | 0.1 (2.74)
  Sodium, Year 2, Week 24, n=273 | 0.1 (2.72)
  Sodium, Year 2, Week 32, n=284 | -0.3 (2.79)
  Sodium, Year 2, Week 40, n=264 | -0.2 (2.67)
  Sodium, Year 2, Week 48, n=269 | -0.1 (2.86)
  Sodium, Year 3, Week 8, n=265 | -0.3 (2.81)
  Sodium, Year 3, Week 16, n=260 | -0.3 (2.90)
  Sodium, Year 3, Week 24, n=244 | -0.2 (2.76)
  Sodium, Year 3, Week 32, n=249 | -0.2 (2.74)
  Sodium, Year 3, Week 40, n=245 | -0.2 (2.77)
  Sodium, Year 3, Week 48, n=244 | -0.3 (2.91)
  Sodium, Year 4, Week 8, n=239 | -0.2 (2.72)
  Sodium, Year 4, Week 16, n=238 | -0.2 (2.71)
  Sodium, Year 4, Week 24, n=227 | -0.1 (2.64)
  Sodium, Year 4, Week 32, n=233 | -0.2 (2.57)
  Sodium, Year 4, Week 40, n=220 | -0.1 (2.55)
  Sodium, Year 4, Week 48, n=218 | -0.1 (2.64)
  Sodium, Year 5, Week 8, n=218 | -0.1 (2.85)
  Sodium, Year 5, Week 16, n=214 | -0.1 (2.60)
  Sodium, Year 5, Week 24, n=211 | 0.0 (2.92)
  Sodium, Year 5, Week 32, n=211 | -0.1 (2.74)
  Sodium, Year 5, Week 40, n=198 | 0.1 (3.04)
  Sodium, Year 5, Week 48, n=207 | -0.3 (2.90)
  Sodium, Year 6, Week 8, n=206 | -0.1 (2.96)
  Sodium, Year 6, Week 16, n=198 | -0.3 (2.85)
  Sodium, Year 6, Week 24, n=190 | -0.3 (2.90)
  Sodium, Year 6, Week 32, n=193 | -0.3 (2.90)
  Sodium, Year 6, Week 40, n=185 | -0.3 (2.91)
  Sodium, Year 6, Week 48, n=186 | -0.4 (2.77)
  Sodium,Year 7, Week 8, n=179 | -0.4 (2.90)
  Sodium, Year 7, Week 16, n=179 | -0.5 (2.86)
  Sodium, Year 7, Week 24, n=173 | -0.5 (2.86)
  Sodium, Year 7, Week 32, n=180 | -0.4 (4.24)
  Sodium, Year 7, Week 40, n=175 | -0.2 (2.98)
  Sodium, Year 7, Week 48, n=175 | -0.5 (3.01)
  Sodium, Year 8, Week 8, n=171 | -0.2 (2.96)
  Sodium, Year 8, Week 16, n=170 | -0.3 (3.22)
  Sodium, Year 8, Week 24, n=168 | -0.3 (2.79)
  Sodium, Year 8, Week 32, n=168 | -0.5 (3.01)
  Sodium, Year 8, Week 40, n=162 | -0.3 (2.94)
  Sodium, Year 8, Week 48, n=159 | -0.3 (2.88)
  Sodium, Year 9, Week 8, n=164 | -0.4 (2.94)
  Sodium, Year 9, Week 16, n=162 | -0.4 (3.14)
  Sodium, Year 9, Week 24, n=161 | -0.3 (3.05)
  Sodium, Year 9, Week 32, n=163 | -0.7 (2.94)
  Sodium, Year 9, Week 40, n=156 | -0.4 (3.13)
  Sodium, Year 9, Week 48, n=151 | -0.6 (3.22)
  Sodium, Year 10, Week 8, n=152 | -0.5 (3.25)
  Sodium, Year 10, Week 16, n=143 | -0.3 (3.31)
  Sodium, Year 10, Week 24, n=145 | -0.4 (3.56)
  Sodium, Year 10, Week 32, n=142 | -0.2 (3.15)
  Sodium, Year 10, Week 40, n=138 | -0.1 (2.80)
  Sodium, Year 10, Week 48, n=135 | -0.4 (3.26)
  Sodium, Year 11, Week 8, n=138 | -0.2 (3.21)
  Sodium, Year 11, Week 16, n=128 | -0.5 (3.30)
  Sodium, Year 11, Week 24, n=130 | -0.4 (3.27)
  Sodium, Year 11, Week 32, n=125 | -0.6 (3.19)
  Sodium, Year 11, Week 40, n=124 | -0.5 (3.25)
  Sodium, Year 11, Week 48, n=108 | -0.7 (3.16)
  Sodium, Year 12, Week 8, n=110 | -0.9 (3.07)
  Sodium, Year 12, Week 16, n=97 | -0.7 (3.12)
  Sodium, Year 12, Week 24, n=87 | -0.1 (3.26)
  Sodium, Year 12, Week 32, n=84 | -0.3 (2.91)
  Sodium, Year 12, Week 40, n=82 | -0.5 (3.18)
  Sodium, Year 12, Week 48, n=72 | -1.1 (2.98)
  Sodium, Year 13, Week 8, n=53 | -0.3 (3.04)
  Sodium, Year 13, Week 16, n=42 | -0.3 (2.68)
  Sodium, Year 13, Week 24, n=20 | 0.2 (3.47)
  Sodium, Year 13, Week 32, n=7 | 0.0 (3.21)
  Sodium, Year 13, Week 40, n=1 | 2.0 (NA) — No value as only one participant was analyzed.
  Sodium, Exit, n=248 | -0.7 (2.96)
  Sodium, 8-Week Follow-up, n=220 | -0.5 (3.06)
  Sodium, 24-Week Follow-up , n=200 | -0.3 (3.16)

11. Primary Outcome: Change From Baseline in Creatinine, Urate and Bilirubin at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in creatinine, urate, and bilirubin is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post- Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
micromoles per liter
  Creatinine, Year 1, Week 8, n=284 | 0.436 (11.3838)
  Creatinine, Year 1, Week 16, n=286 | 0.464 (12.4820)
  Creatinine, Year 1, Week 24, n=292 | 1.211 (12.9503)
  Creatinine, Year 1, Week 32, n=287 | 1.047 (12.5885)
  Creatinine, Year 1, Week 40, n=284 | 0.965 (12.0245)
  Creatinine, Year 1, Week 48, n=287 | 0.955 (12.4760)
  Creatinine, Year 2, Week 8, n=288 | 0.583 (11.9874)
  Creatinine, Year 2, Week 16, n=278 | 1.558 (11.7857)
  Creatinine, Year 2, Week 24, n=273 | 1.036 (13.7310)
  Creatinine, Year 2, Week 32, n=284 | 0.716 (14.1894)
  Creatinine, Year 2, Week 40, n=264 | 1.976 (15.7590)
  Creatinine, Year 2, Week 48, n=269 | 1.413 (13.7896)
  Creatinine, Year 3, Week 8, n=265 | -1.268 (14.8256)
  Creatinine, Year 3, Week 16, n=260 | -2.006 (14.6735)
  Creatinine, Year 3, Week 24, n=244 | -2.464 (15.3328)
  Creatinine, Year 3, Week 32, n=249 | -3.089 (14.8793)
  Creatinine, Year 3, Week 40, n=245 | -3.320 (18.5589)
  Creatinine, Year 3, Week 48, n=244 | -3.297 (17.3222)
  Creatinine, Year 4, Week 8, n=239 | -3.440 (14.6181)
  Creatinine, Year 4, Week 16, n=238 | -3.417 (17.3832)
  Creatinine, Year 4, Week 24, n=227 | -3.271 (15.7446)
  Creatinine, Year 4, Week 32, n=233 | -2.238 (15.9372)
  Creatinine, Year 4, Week 40, n=220 | -2.331 (15.0967)
  Creatinine, Year 4, Week 48, n=218 | -1.987 (18.0028)
  Creatinine, Year 5, Week 8, n=218 | -2.514 (16.1511)
  Creatinine, Year 5, Week 16, n=214 | -2.602 (16.0764)
  Creatinine, Year 5, Week 24, n=211 | -1.843 (16.8703)
  Creatinine, Year 5, Week 32, n=211 | -1.634 (17.1000)
  Creatinine, Year 5, Week 40, n=198 | -2.456 (17.8333)
  Creatinine, Year 5, Week 48, n=207 | -3.203 (17.3533)
  Creatinine, Year 6, Week 8, n=206 | -3.562 (16.8131)
  Creatinine, Year 6, Week 16, n=198 | -2.634 (26.0097)
  Creatinine, Year 6, Week 24, n=190 | -4.373 (15.1824)
  Creatinine, Year 6, Week 32, n=193 | -3.527 (18.6685)
  Creatinine, Year 6, Week 40, n=185 | -3.488 (19.8547)
  Creatinine, Year 6, Week 48, n=186 | -3.565 (18.7328)
  Creatinine, Year 7, Week 8, n=179 | -4.198 (19.0041)
  Creatinine, Year 7, Week 16, n=179 | -5.185 (20.4159)
  Creatinine, Year 7, Week 24, n=173 | -6.438 (20.9087)
  Creatinine, Year 7, Week 32, n=180 | -7.907 (19.4999)
  Creatinine, Year 7, Week 40, n=175 | -8.486 (15.0558)
  Creatinine, Year 7, Week 48, n=175 | -8.789 (17.9447)
  Creatinine, Year 8, Week 8, n=171 | -9.202 (17.7671)
  Creatinine, Year 8, Week 16, n=170 | -8.008 (19.5492)
  Creatinine, Year 8, Week 24, n=168 | -8.630 (19.0791)
  Creatinine, Year 8, Week 32, n=168 | -8.682 (19.2383)
  Creatinine, Year 8, Week 40, n=162 | -8.349 (21.3658)
  Creatinine, Year 8, Week 48, n=159 | -8.228 (18.9524)
  Creatinine, Year 9, Week 8, n=164 | -8.517 (14.5862)
  Creatinine, Year 9, Week 16, n=162 | -7.585 (20.0682)
  Creatinine, Year 9, Week 24, n=161 | -8.291 (21.4197)
  Creatinine, Year 9, Week 32, n=163 | -7.593 (18.2143)
  Creatinine, Year 9, Week 40, n=156 | -7.763 (18.4432)
  Creatinine, Year 9, Week 48, n=151 | -8.430 (15.7255)
  Creatinine, Year 10, Week 8, n=152 | -8.258 (19.3747)
  Creatinine, Year 10, Week 16, n=143 | -9.273 (14.3973)
  Creatinine, Year 10, Week 24, n=145 | -7.986 (17.3492)
  Creatinine, Year 10, Week 32, n=142 | -8.217 (17.1597)
  Creatinine, Year 10, Week 40, n=138 | -9.417 (16.4848)
  Creatinine, Year 10, Week 48, n=135 | -8.120 (15.7637)
  Creatinine, Year 11, Week 8, n=138 | -8.584 (16.5792)
  Creatinine, Year 11, Week 16, n=128 | -9.254 (16.0322)
  Creatinine, Year 11, Week 24, n=130 | -8.500 (16.4151)
  Creatinine, Year 11, Week 32, n=125 | -8.699 (15.1035)
  Creatinine, Year 11, Week 40, n=124 | -7.058 (19.1292)
  Creatinine, Year 11, Week 48, n=108 | -7.858 (15.6339)
  Creatinine, Year 12, Week 8, n=110 | -7.715 (14.5236)
  Creatinine, Year 12, Week 16, n=97 | -6.744 (13.1845)
  Creatinine, Year 12, Week 24, n=87 | -7.316 (13.4273)
  Creatinine, Year 12, Week 32, n=84 | -7.998 (14.5624)
  Creatinine, Year 12, Week 40, n=82 | -7.331 (14.9482)
  Creatinine, Year 12, Week 48, n=72 | -8.103 (14.0558)
  Creatinine, Year 13, Week 8, n=53 | -7.672 (12.1403)
  Creatinine, Year 13, Week 16, n=42 | -6.104 (9.8570)
  Creatinine, Year 13, Week 24, n=20 | -9.282 (9.7155)
  Creatinine, Year 13, Week 32, n=7 | -3.789 (15.1893)
  Creatinine, Year 13, Week 40, n=1 | -8.840 (NA) — No value as only one participant was analyzed.
  Creatinine, Exit, n=248 | -3.707 (21.7147)
  Creatinine, 8-Week Follow-up, n=220 | -4.058 (21.6587)
  Creatinine, 24-Week Follow-up , n=200 | -5.216 (19.0936)
  Urate, Year 1, Week 8, n=284 | 1.8849 (44.3384)
  Urate, Year 1, Week 16, n=286 | -2.8076 (47.4812)
  Urate, Year 1, Week 24, n=292 | -2.6888 (47.8723)
  Urate, Year 1, Week 32, n=287 | -4.9739 (51.9503)
  Urate, Year 1, Week 40, n=284 | -10.2415 (52.6846)
  Urate, Year 1, Week 48, n=287 | -9.6785 (52.9454)
  Urate, Year 2, Week 8, n=288 | -5.8034 (54.3409)
  Urate, Year 2, Week 16, n=278 | -2.2679 (55.1544)
  Urate, Year 2, Week 24, n=273 | -2.5709 (59.5925)
  Urate, Year 2, Week 32, n=284 | -2.1153 (62.2559)
  Urate, Year 2, Week 40, n=264 | 0.8111 (59.7227)
  Urate, Year 2, Week 48, n=269 | 2.1448 (60.1246)
  Urate, Year 3, Week 8, n=265 | 2.1772 (66.2923)
  Urate, Year 3, Week 16, n=260 | 8.6246 (60.1972)
  Urate, Year 3, Week 24, n=244 | 17.1614 (64.9072)
  Urate, Year 3, Week 32, n=249 | 20.6627 (69.7507)
  Urate, Year 3, Week 40, n=245 | 15.5862 (64.9204)
  Urate, Year 3, Week 48, n=244 | 17.2346 (69.9632)
  Urate, Year 4, Week 8, n=239 | 18.8644 (69.2770)
  Urate, Year 4, Week 16, n=238 | 17.0443 (65.9764)
  Urate, Year 4, Week 24, n=227 | 22.1150 (73.0409)
  Urate, Year 4, Week 32, n=233 | 27.1872 (67.0773)
  Urate, Year 4, Week 40, n=220 | 20.6017 (77.3509)
  Urate, Year 4, Week 48, n=218 | 27.3663 (74.9898)
  Urate, Year 5, Week 8, n=218 | 26.3294 (73.0884)
  Urate, Year 5, Week 16, n=214 | 26.4325 (75.1583)
  Urate, Year 5, Week 24, n=211 | 25.6525 (73.5651)
  Urate, Year 5, Week 32, n=211 | 32.0515 (75.9635)
  Urate, Year 5, Week 40, n=198 | 26.8862 (77.2803)
  Urate, Year 5, Week 48, n=207 | 24.9126 (79.1890)
  Urate, Year 6, Week 8, n=206 | 26.3329 (80.0258)
  Urate, Year 6, Week 16, n=198 | 27.2166 (79.2525)
  Urate, Year 6, Week 24, n=190 | 32.5888 (81.4485)
  Urate, Year 6, Week 32, n=193 | 32.3904 (81.4550)
  Urate, Year 6, Week 40, n=185 | 34.4019 (75.0211)
  Urate, Year 6, Week 48, n=186 | 39.1737 (75.6743)
  Urate, Year 7, Week 8, n=179 | 34.0930 (75.0241)
  Urate, Year 7, Week 16, n=179 | 35.0566 (77.2918)
  Urate, Year 7, Week 24, n=173 | 34.7941 (80.7184)
  Urate, Year 7, Week 32, n=180 | 32.8792 (75.6337)
  Urate, Year 7, Week 40, n=175 | 31.7453 (81.9889)
  Urate, Year 7, Week 48, n=175 | 31.9832 (78.3131)
  Urate, Year 8, Week 8, n=171 | 26.6790 (79.7678)
  Urate, Year 8, Week 16, n=170 | 30.7197 (83.1681)
  Urate, Year 8, Week 24, n=168 | 25.4560 (83.0349)
  Urate, Year 8, Week 32, n=168 | 30.0940 (81.9997)
  Urate, Year 8, Week 40, n=162 | 29.4096 (76.1203)
  Urate, Year 8, Week 48, n=159 | 29.9270 (82.9390)
  Urate, Year 9, Week 8, n=164 | 37.6828 (78.7998)
  Urate, Year 9, Week 16, n=162 | 27.2066 (79.3972)
  Urate, Year 9, Week 24, n=161 | 25.9717 (78.7793)
  Urate, Year 9, Week 32, n=163 | 26.1639 (78.0704)
  Urate, Year 9, Week 40, n=156 | 24.7833 (81.4956)
  Urate, Year 9, Week 48, n=151 | 21.9012 (82.0174)
  Urate, Year 10, Week 8, n=152 | 24.8486 (75.5325)
  Urate, Year 10, Week 16, n=143 | 17.5528 (82.4129)
  Urate, Year 10, Week 24, n=145 | 17.6389 (88.8154)
  Urate, Year 10, Week 32, n=142 | 16.9644 (84.0128)
  Urate, Year 10, Week 40, n=138 | 16.0768 (88.6943)
  Urate, Year 10, Week 48, n=135 | 20.9722 (92.2400)
  Urate, Year 11, Week 8, n=138 | 16.3354 (88.7370)
  Urate, Year 11, Week 16, n=128 | 19.0057 (80.9138)
  Urate, Year 11, Week 24, n=129 | 13.8326 (91.9844)
  Urate, Year 11, Week 32, n=125 | 14.4180 (81.6362)
  Urate, Year 11, Week 40, n=124 | 17.8920 (97.1467)
  Urate, Year 11, Week 48, n=108 | 15.9164 (86.7371)
  Urate, Year 12, Week 8, n=110 | 18.3307 (92.3013)
  Urate, Year 12, Week 16, n=97 | 15.3912 (85.1873)
  Urate, Year 12, Week 24, n=87 | 15.3828 (87.1985)
  Urate, Year 12, Week 32, n=84 | 16.7817 (89.8376)
  Urate, Year 12, Week 40, n=82 | 12.2587 (83.5304)
  Urate, Year 12, Week 48, n=72 | 9.9133 (85.1185)
  Urate, Year 13, Week 8, n=53 | 32.4334 (79.1035)
  Urate, Year 13, Week 16, n=42 | 42.6273 (74.2314)
  Urate, Year 13, Week 24, n=20 | 25.5764 (56.8583)
  Urate, Year 13, Week 32, n=7 | 64.5783 (59.0251)
  Urate, Year 13, Week 40, n=1 | 53.5320 (NA) — No value as only one participant was analyzed.
  Urate, Exit, n=248 | 18.5635 (89.4280)
  Urate, 8-Week Follow-up, n=220 | 19.6014 (89.9097)
  Urate, 24-Week Follow-up , n=200 | 17.5763 (82.1420)
  Bilirubin, Year 1, Week 8, n=283 | 0.145 (2.2995)
  Bilirubin, Year 1, Week 16, n=285 | 0.168 (2.3476)
  Bilirubin, Year 1, Week 24, n=292 | 0.287 (2.4529)
  Bilirubin, Year 1, Week 32, n=287 | 0.346 (2.6100)
  Bilirubin, Year 1, Week 40, n=283 | 0.236 (2.3829)
  Bilirubin, Year 1, Week 48, n=286 | 0.293 (2.5315)
  Bilirubin, Year 2, Week 8, n=288 | 0.243 (2.6498)
  Bilirubin, Year 2, Week 16, n=277 | 0.019 (2.5896)
  Bilirubin, Year 2, Week 24, n=272 | 0.176 (2.5041)
  Bilirubin, Year 2, Week 32, n=284 | 0.331 (2.6475)
  Bilirubin, Year 2, Week 40, n=262 | 0.398 (2.9233)
  Bilirubin, Year 2, Week 48, n=269 | 0.464 (2.5138)
  Bilirubin, Year 3, Week 8, n=264 | 0.343 (2.6599)
  Bilirubin, Year 3, Week 16, n=258 | 0.252 (2.8788)
  Bilirubin, Year 3, Week 24, n=243 | 0.274 (3.0754)
  Bilirubin, Year 3, Week 32, n=249 | 0.494 (2.5860)
  Bilirubin, Year 3, Week 40, n=244 | 0.182 (2.8589)
  Bilirubin, Year 3, Week 48, n=243 | 0.267 (3.0780)
  Bilirubin, Year 4, Week 8, n=239 | 0.336 (2.7639)
  Bilirubin, Year 4, Week 16, n=238 | 0.481 (2.8625)
  Bilirubin, Year 4, Week 24, n=227 | 0.309 (2.8038)
  Bilirubin, Year 4, Week 32, n=231 | 0.326 (2.9524)
  Bilirubin, Year 4, Week 40, n=220 | -0.023 (2.5236)
  Bilirubin, Year 4, Week 48, n=218 | 0.157 (2.8815)
  Bilirubin, Year 5, Week 8, n=218 | 0.329 (2.4013)
  Bilirubin, Year 5, Week 16, n=214 | 0.304 (2.6180)
  Bilirubin, Year 5, Week 24, n=211 | 0.259 (2.5450)
  Bilirubin, Year 5, Week 32, n=211 | 0.575 (2.6520)
  Bilirubin, Year 5, Week 40, n=198 | 0.544 (2.6496)
  Bilirubin, Year 5, Week 48, n=207 | 0.322 (2.5320)
  Bilirubin, Year 6, Week 8, n=206 | 0.282 (2.5233)
  Bilirubin, Year 6, Week 16, n=198 | 0.138 (2.6093)
  Bilirubin, Year 6, Week 24, n=190 | 0.099 (2.7600)
  Bilirubin, Year 6, Week 32, n=193 | 0.284 (2.6431)
  Bilirubin, Year 6, Week 40, n=185 | 0.296 (2.8314)
  Bilirubin, Year 6, Week 48, n=186 | 0.248 (3.0097)
  Bilirubin, Year 7, Week 8, n=179 | 0.258 (2.6974)
  Bilirubin, Year 7, Week 16, n=179 | 0.143 (2.6134)
  Bilirubin, Year 7, Week 24, n=173 | 0.287 (2.6082)
  Bilirubin, Year 7, Week 32, n=180 | 0.313 (2.9727)
  Bilirubin, Year 7, Week 40, n=175 | 0.137 (2.7527)
  Bilirubin, Year 7, Week 48, n=175 | 0.156 (2.9747)
  Bilirubin, Year 8, Week 8, n=171 | 0.020 (2.9559)
  Bilirubin, Year 8, Week 16, n=170 | -0.050 (2.6856)
  Bilirubin, Year 8, Week 24, n=168 | 0.010 (2.4720)
  Bilirubin, Year 8, Week 32, n=168 | -0.336 (2.5471)
  Bilirubin, Year 8, Week 40, n=162 | -0.032 (2.8934)
  Bilirubin, Year 8, Week 48, n=159 | -0.097 (3.2550)
  Bilirubin, Year 9, Week 8, n=164 | -0.125 (2.7616)
  Bilirubin, Year 9, Week 16, n=162 | -0.095 (2.9603)
  Bilirubin, Year 9, Week 24, n=161 | -0.234 (3.1385)
  Bilirubin, Year 9, Week 32, n=163 | -0.126 (2.7175)
  Bilirubin, Year 9, Week 40, n=156 | -0.296 (3.3709)
  Bilirubin, Year 9, Week 48, n=151 | 0.057 (2.8231)
  Bilirubin, Year 10, Week 8, n=152 | -0.158 (3.0763)
  Bilirubin, Year 10, Week 16, n=143 | -0.179 (3.1616)
  Bilirubin, Year 10, Week 24, n=145 | -0.024 (2.8853)
  Bilirubin, Year 10, Week 32, n=142 | 0.120 (3.3068)
  Bilirubin, Year 10, Week 40, n=138 | -0.248 (3.0684)
  Bilirubin, Year 10, Week 48, n=135 | 0.190 (3.0751)
  Bilirubin, Year 11, Week 8, n=138 | 0.050 (2.9936)
  Bilirubin, Year 11, Week 16, n=128 | 0.281 (2.9640)
  Bilirubin, Year 11, Week 24, n=130 | 0.026 (2.8004)
  Bilirubin, Year 11, Week 32, n=125 | 0.192 (2.5160)
  Bilirubin, Year 11, Week 40, n=124 | 0.193 (3.2650)
  Bilirubin, Year 11, Week 48, n=108 | 0.538 (2.9261)
  Bilirubin, Year 12, Week 8, n=110 | 0.311 (2.8762)
  Bilirubin, Year 12, Week 16, n=97 | 0.776 (3.0231)
  Bilirubin, Year 12, Week 24, n=87 | 0.511 (3.4508)
  Bilirubin, Year 12, Week 32, n=84 | 1.282 (3.3563)
  Bilirubin, Year 12, Week 40, n=82 | 0.542 (3.2454)
  Bilirubin, Year 12, Week 48, n=72 | 0.570 (3.8398)
  Bilirubin, Year 13, Week 8, n=53 | 0.129 (2.8623)
  Bilirubin, Year 13, Week 16, n=42 | -0.244 (3.1046)
  Bilirubin, Year 13, Week 24, n=20 | -0.513 (2.0080)
  Bilirubin, Year 13, Week 32, n=7 | -0.244 (2.5032)
  Bilirubin, Year 13, Week 40, n=1 | 0.000 (NA) — No value as only one participant was analyzed.
  Bilirubin, Exit, n=248 | 0.510 (3.0619)
  Bilirubin, 8-Week Follow-up, n=220 | 0.389 (2.7311)
  Bilirubin, 24-Week Follow-up , n=200 | 0.650 (3.3222)

12. Primary Outcome: Change From Baseline in BUN/Creatinine at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in BUN/creatinine is summarized. The Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Ratio
  BUN/Creatinine, Year 1, Week 8, n=284 | -0.1 (4.13)
  BUN/Creatinine, Year 1, Week 16, n=286 | -0.4 (4.31)
  BUN/Creatinine, Year 1, Week 24, n=292 | -0.4 (4.67)
  BUN/Creatinine, Year 1, Week 32, n=287 | -0.4 (4.07)
  BUN/Creatinine, Year 1, Week 40, n=284 | -0.8 (4.26)
  BUN/Creatinine, Year 1, Week 48, n=287 | -0.3 (4.80)
  BUN/Creatinine, Year 2, Week 8, n=288 | -0.4 (4.91)
  BUN/Creatinine, Year 2, Week 16, n=278 | -0.6 (4.95)
  BUN/Creatinine, Year 2, Week 24, n=273 | -0.6 (5.00)
  BUN/Creatinine, Year 2, Week 32, n=284 | -0.4 (4.82)
  BUN/Creatinine, Year 2, Week 40, n=264 | -0.8 (4.80)
  BUN/Creatinine, Year 2, Week 48, n=269 | -0.5 (4.90)
  BUN/Creatinine, Year 3, Week 8, n=265 | 0.2 (4.81)
  BUN/Creatinine, Year 3, Week 16, n=260 | 0.2 (4.95)
  BUN/Creatinine, Year 3, Week 24, n=244 | 0.6 (4.93)
  BUN/Creatinine, Year 3, Week 32, n=249 | 0.5 (5.16)
  BUN/Creatinine, Year 3, Week 40, n=245 | 0.9 (4.83)
  BUN/Creatinine, Year 3, Week 48, n=244 | 0.8 (4.99)
  BUN/Creatinine, Year 4, Week 8, n=239 | 1.1 (4.99)
  BUN/Creatinine, Year 4, Week 16, n=238 | 0.8 (4.86)
  BUN/Creatinine, Year 4, Week 24, n=227 | 0.9 (5.15)
  BUN/Creatinine, Year 4, Week 32, n=233 | 0.5 (4.93)
  BUN/Creatinine, Year 4, Week 40, n=220 | 0.3 (4.81)
  BUN/Creatinine, Year 4, Week 48, n=218 | 1.1 (5.35)
  BUN/Creatinine, Year 5, Week 8, n=218 | 0.8 (5.34)
  BUN/Creatinine, Year 5, Week 16, n=214 | 1.2 (5.03)
  BUN/Creatinine, Year 5, Week 24, n=211 | 0.8 (5.01)
  BUN/Creatinine, Year 5, Week 32, n=211 | 0.3 (4.93)
  BUN/Creatinine, Year 5, Week 40, n=198 | 1.2 (5.04)
  BUN/Creatinine, Year 5, Week 48, n=207 | 0.9 (5.11)
  BUN/Creatinine, Year 6, Week 8, n=206 | 1.4 (5.04)
  BUN/Creatinine, Year 6, Week 16, n=198 | 1.3 (5.03)
  BUN/Creatinine, Year 6, Week 24, n=190 | 1.2 (5.37)
  BUN/Creatinine, Year 6, Week 32, n=193 | 1.6 (5.76)
  BUN/Creatinine, Year 6, Week 40, n=185 | 1.5 (4.73)
  BUN/Creatinine, Year 6, Week 48, n=186 | 1.8 (5.08)
  BUN/Creatinine, Year 7, Week 8, n=179 | 1.6 (5.07)
  BUN/Creatinine, Year 7, Week 16, n=179 | 2.1 (5.04)
  BUN/Creatinine, Year 7, Week 24, n=173 | 2.1 (5.55)
  BUN/Creatinine, Year 7, Week 32, n=180 | 2.3 (5.39)
  BUN/Creatinine, Year 7, Week 40, n=175 | 2.6 (5.19)
  BUN/Creatinine, Year 7, Week 48, n=175 | 2.6 (5.31)
  BUN/Creatinine, Year 8, Week 8, n=171 | 2.7 (5.65)
  BUN/Creatinine, Year 8, Week 16, n=170 | 2.5 (5.54)
  BUN/Creatinine, Year 8, Week 24, n=168 | 2.6 (5.37)
  BUN/Creatinine, Year 8, Week 32, n=168 | 2.2 (5.11)
  BUN/Creatinine, Year 8, Week 40, n=162 | 2.3 (5.36)
  BUN/Creatinine, Year 8, Week 48, n=159 | 2.9 (5.20)
  BUN/Creatinine, Year 9, Week 8, n=164 | 2.4 (5.26)
  BUN/Creatinine, Year 9, Week 16, n=162 | 2.5 (6.15)
  BUN/Creatinine, Year 9, Week 24, n=161 | 2.4 (5.89)
  BUN/Creatinine, Year 9, Week 32, n=163 | 2.7 (5.54)
  BUN/Creatinine, Year 9, Week 40, n=156 | 2.4 (5.90)
  BUN/Creatinine, Year 9, Week 48, n=151 | 2.2 (6.01)
  BUN/Creatinine, Year 10, Week 8, n=152 | 2.6 (5.98)
  BUN/Creatinine, Year 10, Week 16, n=143 | 2.6 (6.13)
  BUN/Creatinine, Year 10, Week 24, n=145 | 2.5 (5.72)
  BUN/Creatinine, Year 10, Week 32, n=142 | 2.8 (6.03)
  BUN/Creatinine, Year 10, Week 40, n=138 | 2.0 (5.87)
  BUN/Creatinine, Year 10, Week 48, n=135 | 2.4 (6.07)
  BUN/Creatinine, Year 11, Week 8, n=138 | 2.7 (6.13)
  BUN/Creatinine, Year 11, Week 16, n=128 | 2.6 (6.28)
  BUN/Creatinine, Year 11, Week 24, n=130 | 2.8 (6.12)
  BUN/Creatinine, Year 11, Week 32, n=125 | 2.2 (6.10)
  BUN/Creatinine, Year 11, Week 40, n=124 | 2.3 (6.68)
  BUN/Creatinine, Year 11, Week 48, n=108 | 1.7 (5.65)
  BUN/Creatinine, Year 12, Week 8, n=110 | 2.4 (6.36)
  BUN/Creatinine, Year 12, Week 16, n=97 | 2.4 (6.38)
  BUN/Creatinine, Year 12, Week 24, n=87 | 2.2 (6.62)
  BUN/Creatinine, Year 12, Week 32, n=84 | 1.5 (5.75)
  BUN/Creatinine, Year 12, Week 40, n=82 | 1.4 (6.50)
  BUN/Creatinine, Year 12, Week 48, n=72 | 1.6 (6.42)
  BUN/Creatinine, Year 13, Week 8, n=53 | 2.1 (5.44)
  BUN/Creatinine, Year 13, Week 16, n=42 | 3.5 (6.22)
  BUN/Creatinine, Year 13, Week 24, n=20 | 3.6 (4.36)
  BUN/Creatinine, Year 13, Week 32, n=7 | 0.3 (2.93)
  BUN/Creatinine, Year 13, Week 40, n=1 | -6.0 (NA) — No value as only one participant was analyzed.
  BUN/Creatinine, Exit, n=248 | 1.6 (5.66)
  BUN/Creatinine, 8-Week Follow-up, n=220 | 1.1 (5.88)
  BUN/Creatinine, 24-Week Follow-up , n=200 | 1.3 (5.53)

13. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase (LD) at the Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline, Week 8, 16, 24, 32, 40 and 48 during Year 1 to 12; Week 8, 16, 24, 32, and 40 during Year 13; Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Change from Baseline in ALT, AP, AST, GGT and LD are summarized. Baseline is defined as the Extension Year 1 Day 0 values for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
International units per liter
  ALT, Year 1, Week 8, n=284 | -0.7 (12.05)
  ALT, Year 1, Week 16, n=286 | 0.2 (17.32)
  ALT, Year 1, Week 24, n=292 | 0.9 (17.04)
  ALT, Year 1, Week 32, n=287 | -0.6 (12.36)
  ALT, Year 1, Week 40, n=284 | -0.6 (14.15)
  ALT, Year 1, Week 48, n=287 | -1.3 (11.56)
  ALT, Year 2, Week 8, n=288 | -0.7 (13.36)
  ALT, Year 2, Week 16, n=278 | -1.2 (11.44)
  ALT, Year 2, Week 24, n=273 | 0.3 (13.35)
  ALT, Year 2, Week 32, n=284 | 0.1 (15.85)
  ALT, Year 2, Week 40, n=264 | 0.0 (14.02)
  ALT, Year 2, Week 48, n=269 | 0.9 (15.65)
  ALT, Year 3, Week 8, n=265 | 0.5 (14.46)
  ALT, Year 3, Week 16, n=260 | 1.3 (21.94)
  ALT, Year 3, Week 24, n=244 | -0.1 (13.95)
  ALT, Year 3, Week 32, n=249 | 0.0 (12.55)
  ALT, Year 3, Week 40, n=245 | -0.3 (13.08)
  ALT, Year 3, Week 48, n=244 | -0.4 (13.62)
  ALT, Year 4, Week 8, n=239 | -0.5 (10.97)
  ALT, Year 4, Week 16, n=238 | -1.3 (14.28)
  ALT, Year 4, Week 24, n=227 | -1.3 (13.29)
  ALT, Year 4, Week 32, n=233 | -0.4 (13.60)
  ALT, Year 4, Week 40, n=220 | -1.6 (12.83)
  ALT, Year 4, Week 48, n=218 | -1.3 (12.45)
  ALT, Year 5, Week 8, n=218 | 0.1 (12.76)
  ALT, Year 5, Week 16, n=214 | -0.5 (12.67)
  ALT, Year 5, Week 24, n=211 | -0.9 (14.68)
  ALT, Year 5, Week 32, n=211 | -1.5 (13.23)
  ALT, Year 5, Week 40, n=198 | -1.3 (13.90)
  ALT, Year 5, Week 48, n=207 | -0.1 (17.16)
  ALT, Year 6, Week 8, n=206 | -1.4 (12.09)
  ALT, Year 6, Week 16, n=198 | -1.4 (13.55)
  ALT, Year 6, Week 24, n=190 | -1.6 (13.87)
  ALT, Year 6, Week 32, n=193 | -1.4 (13.58)
  ALT, Year 6, Week 40, n=185 | -1.4 (14.78)
  ALT, Year 6, Week 48, n=186 | -0.9 (14.98)
  ALT, Year 7, Week 8, n=179 | -0.4 (14.50)
  ALT, Year 7, Week 16, n=179 | 0.5 (15.78)
  ALT, Year 7, Week 24, n=173 | 0.1 (16.09)
  ALT, Year 7, Week 32, n=180 | -0.2 (14.71)
  ALT, Year 7, Week 40, n=175 | -0.1 (16.43)
  ALT, Year 7, Week 48, n=175 | -0.4 (16.15)
  ALT, Year 8, Week 8, n=171 | 0.9 (16.58)
  ALT, Year 8, Week 16, n=170 | -0.2 (17.74)
  ALT, Year 8, Week 24, n=168 | -0.2 (15.62)
  ALT, Year 8, Week 32, n=168 | -0.4 (14.82)
  ALT, Year 8, Week 40, n=162 | -0.7 (14.79)
  ALT, Year 8, Week 48, n=159 | -0.7 (15.14)
  ALT, Year 9, Week 8, n=164 | 1.5 (21.38)
  ALT, Year 9, Week 16, n=162 | -0.8 (14.31)
  ALT, Year 9, Week 24, n=161 | -1.5 (14.35)
  ALT, Year 9, Week 32, n=163 | 0.0 (15.62)
  ALT, Year 9, Week 40, n=156 | -0.5 (14.61)
  ALT, Year 9, Week 48, n=151 | -0.2 (15.69)
  ALT, Year 10, Week 8, n=152 | -0.6 (14.25)
  ALT, Year 10, Week 16, n=143 | -0.3 (13.88)
  ALT, Year 10, Week 24, n=145 | -1.1 (15.71)
  ALT, Year 10, Week 32, n=142 | -0.8 (15.97)
  ALT, Year 10, Week 40, n=138 | -1.9 (15.56)
  ALT, Year 10, Week 48, n=135 | -0.7 (19.61)
  ALT, Year 11, Week 8, n=138 | -1.9 (15.75)
  ALT, Year 11, Week 16, n=128 | -1.3 (16.74)
  ALT, Year 11, Week 24, n=130 | -2.5 (15.11)
  ALT, Year 11, Week 32, n=125 | -3.2 (14.71)
  ALT, Year 11, Week 40, n=124 | -2.8 (15.31)
  ALT, Year 11, Week 48, n=108 | -1.7 (18.29)
  ALT, Year 12, Week 8, n=110 | -1.9 (16.30)
  ALT, Year 12, Week 16, n=97 | -2.9 (12.74)
  ALT, Year 12, Week 24, n=87 | -2.0 (13.47)
  ALT, Year 12, Week 32, n=84 | -2.4 (13.39)
  ALT, Year 12, Week 40, n=82 | -2.3 (14.74)
  ALT, Year 12, Week 48, n=72 | -3.6 (14.92)
  ALT, Year 13, Week 8, n=53 | -5.3 (16.58)
  LT, Year 13, Week 16, n=42 | -5.7 (20.42)
  ALT, Year 13, Week 24, n=20 | -1.0 (6.55)
  ALT, Year 13, Week 32, n=7 | -0.6 (9.14)
  ALT, Year 13, Week 40, n=1 | 3.0 (NA) — No value as only one participant was analyzed.
  ALT, Exit, n=248 | -1.2 (13.39)
  ALT, 8-Week Follow-up, n=220 | -0.6 (15.74)
  ALT, 24-Week Follow-up , n=200 | 1.5 (36.52)
  AP, Year 1, Week 8, n=284 | -0.1 (11.43)
  AP, Year 1, Week 16, n=286 | 0.9 (14.08)
  AP, Year 1, Week 24, n=292 | 0.7 (13.87)
  AP, Year 1, Week 32, n=287 | 0.6 (14.03)
  AP, Year 1, Week 40, n=284 | 1.1 (14.61)
  AP, Year 1, Week 48, n=287 | 0.5 (16.94)
  AP, Year 2, Week 8, n=288 | 1.2 (17.67)
  AP, Year 2, Week 16, n=278 | 0.2 (15.87)
  AP, Year 2, Week 24, n=273 | 1.3 (16.91)
  AP, Year 2, Week 32, n=284 | 2.5 (17.17)
  AP, Year 2, Week 40, n=264 | 3.5 (19.55)
  AP, Year 2, Week 48, n=269 | 5.6 (23.81)
  AP, Year 3, Week 8, n=265 | 4.0 (18.04)
  AP, Year 3, Week 16, n=260 | 3.2 (19.53)
  AP, Year 3, Week 24, n=244 | 2.0 (19.26)
  AP, Year 3, Week 32, n=249 | 3.7 (21.48)
  AP, Year 3, Week 40, n=245 | 3.4 (18.62)
  AP, Year 3, Week 48, n=244 | 3.4 (19.32)
  AP, Year 4, Week 8, n=239 | 2.5 (19.33)
  AP, Year 4, Week 16, n=238 | 2.8 (17.37)
  AP, Year 4, Week 24, n=227 | 2.5 (21.94)
  AP, Year 4, Week 32, n=233 | 3.7 (21.17)
  AP, Year 4, Week 40, n=220 | 2.9 (20.93)
  AP, Year 4, Week 48, n=218 | 3.7 (22.97)
  AP, Year 5, Week 8, n=218 | 4.9 (24.65)
  AP, Year 5, Week 16, n=214 | 4.1 (23.87)
  AP, Year 5, Week 24, n=211 | 4.0 (20.17)
  AP, Year 5, Week 32, n=211 | 5.7 (20.68)
  AP, Year 5, Week 40, n=198 | 5.5 (21.34)
  AP, Year 5, Week 48, n=207 | 6.6 (21.74)
  AP, Year 6, Week 8, n=206 | 7.1 (23.65)
  AP, Year 6, Week 16, n=198 | 7.5 (21.41)
  AP, Year 6, Week 24, n=190 | 7.5 (22.41)
  AP, Year 6, Week 32, n=193 | 14.0 (67.61)
  AP, Year 6, Week 40, n=185 | 10.2 (24.43)
  AP, Year 6, Week 48, n=186 | 9.1 (22.93)
  AP, Year 7, Week 8, n=179 | 9.0 (24.52)
  AP, Year 7, Week 16, n=179 | 9.6 (25.70)
  AP, Year 7, Week 24, n=173 | 9.9 (25.38)
  AP, Year 7, Week 32, n=180 | 11.5 (27.02)
  AP, Year 7, Week 40, n=175 | 9.6 (25.13)
  AP, Year 7, Week 48, n=175 | 11.1 (24.96)
  AP, Year 8, Week 8, n=171 | 10.0 (23.29)
  AP, Year 8, Week 16, n=170 | 10.1 (27.16)
  AP, Year 8, Week 24, n=168 | 10.4 (26.44)
  AP, Year 8, Week 32, n=168 | 12.9 (27.45)
  AP, Year 8, Week 40, n=162 | 11.1 (25.66)
  AP, Year 8, Week 48, n=159 | 11.5 (30.97)
  AP, Year 9, Week 8, n=164 | 12.0 (25.38)
  AP, Year 9, Week 16, n=162 | 10.9 (25.48)
  AP, Year 9, Week 24, n=161 | 10.5 (22.81)
  AP, Year 9, Week 32, n=163 | 10.4 (24.05)
  AP, Year 9, Week 40, n=156 | 9.5 (24.43)
  AP, Year 9, Week 48, n=151 | 10.2 (22.77)
  AP, Year 10, Week 8, n=152 | 10.6 (24.51)
  AP, Year 10, Week 16, n=143 | 11.9 (29.31)
  AP, Year 10, Week 24, n=145 | 13.0 (22.92)
  AP, Year 10, Week 32, n=142 | 14.4 (24.55)
  AP, Year 10, Week 40, n=138 | 13.7 (23.20)
  AP, Year 10, Week 48, n=135 | 12.5 (23.89)
  AP, Year 11, Week 8, n=138 | 13.3 (26.11)
  AP, Year 11, Week 16, n=128 | 14.2 (26.05)
  AP, Year 11, Week 24, n=130 | 12.9 (23.22)
  AP, Year 11, Week 32, n=125 | 13.3 (23.74)
  AP, Year 11, Week 40, n=124 | 13.3 (23.05)
  AP, Year 11, Week 48, n=108 | 11.9 (25.59)
  AP, Year 12, Week 8, n=110 | 12.3 (25.69)
  AP, Year 12, Week 16, n=97 | 10.2 (22.48)
  AP, Year 12, Week 24, n=87 | 11.5 (20.69)
  AP, Year 12, Week 32, n=84 | 10.7 (19.91)
  AP, Year 12, Week 40, n=82 | 10.8 (21.35)
  AP, Year 12, Week 48, n=72 | 11.6 (21.77)
  AP, Year 13, Week 8, n=53 | 12.2 (19.25)
  AP, Year 13, Week 16, n=42 | 16.9 (37.69)
  AP, Year 13, Week 24, n=20 | 20.7 (23.57)
  AP, Year 13, Week 32, n=7 | 18.1 (21.47)
  AP, Year 13, Week 40, n=1 | 15.0 (NA) — No value as only one participant was analyzed.
  AP, Exit, n=248 | 8.3 (26.49)
  AP, 8-Week Follow-up, n=220 | 10.3 (42.15)
  AP, 24-Week Follow-up , n=200 | 10.7 (32.86)
  AST, Year 1, Week 8, n=281 | -0.3 (8.68)
  AST, Year 1, Week 16, n=283 | 2.0 (22.78)
  AST, Year 1, Week 24, n=287 | 2.3 (26.94)
  AST, Year 1, Week 32, n=283 | 0.5 (12.19)
  AST, Year 1, Week 40, n=282 | -0.1 (9.63)
  AST, Year 1, Week 48, n=284 | -1.2 (6.98)
  AST, Year 2, Week 8, n=288 | -0.8 (9.15)
  AST, Year 2, Week 16, n=275 | -1.2 (8.51)
  AST, Year 2, Week 24, n=269 | -0.3 (9.04)
  AST, Year 2, Week 32, n=284 | 0.2 (13.80)
  AST, Year 2, Week 40, n=261 | -0.2 (10.44)
  AST, Year 2, Week 48, n=267 | 0.7 (10.95)
  AST, Year 3, Week 8, n=262 | 0.3 (10.81)
  AST, Year 3, Week 16, n=258 | 1.0 (11.84)
  AST, Year 3, Week 24, n=241 | 0.4 (10.36)
  AST, Year 3, Week 32, n=245 | 1.3 (11.19)
  AST, Year 3, Week 40, n=242 | 0.2 (10.99)
  AST, Year 3, Week 48, n=239 | 0.6 (10.60)
  AST, Year 4, Week 8, n=237 | 0.5 (7.73)
  AST, Year 4, Week 16, n=235 | -0.2 (12.78)
  AST, Year 4, Week 24, n=226 | 0.4 (11.45)
  AST, Year 4, Week 32, n=230 | 0.8 (9.26)
  AST, Year 4, Week 40, n=218 | -0.3 (9.44)
  AST, Year 4, Week 48, n=214 | -0.2 (9.48)
  AST, Year 5, Week 8, n=217 | 0.3 (12.79)
  AST, Year 5, Week 16, n=213 | 0.8 (15.76)
  AST, Year 5, Week 24, n=206 | -0.5 (11.36)
  AST, Year 5, Week 32, n=211 | -0.8 (10.64)
  AST, Year 5, Week 40, n=197 | 0.3 (14.39)
  AST, Year 5, Week 48, n=207 | 0.0 (11.58)
  AST, Year 6, Week 8, n=205 | -0.4 (9.04)
  AST, Year 6, Week 16, n=198 | -0.7 (9.83)
  AST, Year 6, Week 24, n=189 | -0.9 (11.35)
  AST, Year 6, Week 32, n=192 | -0.6 (11.04)
  AST, Year 6, Week 40, n=181 | -0.7 (10.56)
  AST, Year 6, Week 48, n=186 | 0.1 (12.21)
  AST, Year 7, Week 8, n=177 | -0.2 (10.76)
  AST, Year 7, Week 16, n=178 | 1.0 (12.91)
  AST, Year 7, Week 24, n=171 | 1.5 (14.44)
  AST, Year 7, Week 32, n=179 | 0.5 (10.56)
  AST, Year 7, Week 40, n=172 | 0.4 (14.51)
  AST, Year 7, Week 48, n=175 | 0.2 (11.15)
  AST, Year 8, Week 8, n=170 | 1.0 (16.78)
  AST, Year 8, Week 16, n=169 | 1.0 (21.12)
  AST, Year 8, Week 24, n=167 | 0.5 (13.61)
  AST, Year 8, Week 32, n=166 | 0.7 (14.74)
  AST, Year 8, Week 40, n=161 | 1.4 (16.28)
  AST, Year 8, Week 48, n=159 | 0.2 (11.00)
  AST, Year 9, Week 8, n=163 | 1.6 (16.09)
  AST, Year 9, Week 16, n=160 | 0.8 (13.55)
  AST, Year 9, Week 24, n=160 | 0.3 (12.60)
  AST, Year 9, Week 32, n=162 | 1.3 (17.39)
  AST, Year 9, Week 40, n=156 | 1.0 (14.17)
  AST, Year 9, Week 48, n=150 | 1.5 (15.79)
  AST, Year 10, Week 8, n=151 | 0.0 (11.05)
  AST, Year 10, Week 16, n=143 | 0.1 (13.75)
  AST, Year 10, Week 24, n=145 | 0.1 (13.80)
  AST, Year 10, Week 32, n=140 | 0.5 (13.90)
  AST, Year 10, Week 40, n=137 | -0.4 (13.30)
  AST, Year 10, Week 48, n=135 | 0.9 (14.71)
  AST, Year 11, Week 8, n=138 | -0.2 (12.04)
  AST, Year 11, Week 16, n=128 | -0.1 (12.72)
  AST, Year 11, Week 24, n=129 | -0.3 (12.69)
  AST, Year 11, Week 32, n=124 | -1.0 (10.03)
  AST, Year 11, Week 40, n=124 | 0.1 (14.28)
  AST, Year 11, Week 48, n=107 | 1.3 (17.70)
  AST, Year 12, Week 8, n=109 | 0.1 (16.11)
  AST, Year 12, Week 16, n=97 | -0.5 (7.74)
  AST, Year 12, Week 24, n=85 | 1.0 (13.58)
  AST, Year 12, Week 32, n=84 | 0.5 (11.11)
  AST, Year 12, Week 40, n=82 | 0.2 (11.60)
  AST, Year 12, Week 48, n=72 | -1.0 (12.48)
  AST, Year 13, Week 8, n=53 | -2.5 (10.00)
  AST, Year 13, Week 16, n=42 | -3.4 (14.32)
  AST, Year 13, Week 24, n=20 | 0.1 (7.94)
  AST, Year 13, Week 32, n=7 | 0.3 (4.96)
  AST, Year 13, Week 40, n=1 | 1.0 (NA) — No value as only one participant was analyzed.
  AST, Exit, n=248 | -0.9 (10.19)
  AST, 8-Week Follow-up, n=220 | -0.3 (11.02)
  AST, 24-Week Follow-up , n=200 | 3.3 (52.99)
  GGT, Year 1, Week 8, n=284 | 0.6 (23.57)
  GGT, Year 1, Week 16, n=286 | 5.0 (32.94)
  GGT, Year 1, Week 24, n=292 | 6.3 (48.10)
  GGT, Year 1, Week 32, n=287 | 4.9 (46.96)
  GGT, Year 1, Week 40, n=284 | 6.7 (55.51)
  GGT, Year 1, Week 48, n=287 | 5.2 (58.66)
  GGT, Year 2, Week 8, n=288 | 4.6 (50.82)
  GGT, Year 2, Week 16, n=278 | 2.9 (37.57)
  GGT, Year 2, Week 24, n=273 | 4.5 (42.01)
  GGT, Year 2, Week 32, n=284 | 3.8 (38.55)
  GGT, Year 2, Week 40, n=264 | 4.2 (41.34)
  GGT, Year 2, Week 48, n=269 | 5.7 (48.48)
  GGT, Year 3, Week 8, n=265 | 3.9 (33.83)
  GGT, Year 3, Week 16, n=260 | 5.3 (44.46)
  GGT, Year 3, Week 24, n=244 | 4.0 (51.58)
  GGT, Year 3, Week 32, n=249 | 6.7 (57.32)
  GGT, Year 3, Week 40, n=245 | 3.7 (29.97)
  GGT, Year 3, Week 48, n=244 | 1.7 (39.47)
  GGT, Year 4, Week 8, n=239 | 3.1 (53.57)
  GGT, Year 4, Week 16, n=238 | 1.2 (36.22)
  GGT, Year 4, Week 24, n=226 | 3.0 (55.72)
  GGT, Year 4, Week 32, n=233 | 3.4 (47.24)
  GGT, Year 4, Week 40, n=220 | 2.0 (40.20)
  GGT, Year 4, Week 48, n=218 | 2.6 (39.26)
  GGT, Year 5, Week 8, n=218 | 4.8 (40.08)
  GGT, Year 5, Week 16, n=214 | 1.6 (41.04)
  GGT, Year 5, Week 24, n=211 | 3.0 (39.90)
  GGT, Year 5, Week 32, n=211 | 1.7 (36.58)
  GGT, Year 5, Week 40, n=198 | 1.4 (41.74)
  GGT, Year 5, Week 48, n=207 | 3.6 (46.10)
  GGT, Year 6, Week 8, n=206 | 1.9 (48.45)
  GGT, Year 6, Week 16, n=198 | 1.8 (37.61)
  GGT, Year 6, Week 24, n=190 | 1.6 (43.58)
  GGT, Year 6, Week 32, n=193 | 5.9 (55.25)
  GGT, Year 6, Week 40, n=185 | 2.0 (34.66)
  GGT, Year 6, Week 48, n=186 | 2.2 (38.05)
  GGT, Year 7, Week 8, n=179 | 2.3 (36.39)
  GGT, Year 7, Week 16, n=179 | 3.8 (43.49)
  GGT, Year 7, Week 24, n=173 | 4.5 (33.15)
  GGT, Year 7, Week 32, n=180 | 4.6 (41.12)
  GGT, Year 7, Week 40, n=175 | 4.9 (36.94)
  GGT, Year 7, Week 48, n=175 | 4.9 (40.27)
  GGT, Year 8, Week 8, n=171 | 7.0 (41.53)
  GGT, Year 8, Week 16, n=170 | 6.8 (41.70)
  GGT, Year 8, Week 24, n=168 | 8.5 (48.16)
  GGT, Year 8, Week 32, n=168 | 8.5 (44.76)
  GGT, Year 8, Week 40, n=162 | 3.5 (38.79)
  GGT, Year 8, Week 48, n=159 | 7.3 (37.89)
  GGT, Year 9, Week 8, n=164 | 7.1 (39.19)
  GGT, Year 9, Week 16, n=162 | 5.0 (37.32)
  GGT, Year 9, Week 24, n=161 | 2.6 (33.54)
  GGT, Year 9, Week 32, n=163 | 2.4 (29.43)
  GGT, Year 9, Week 40, n=156 | 2.9 (32.70)
  GGT, Year 9, Week 48, n=151 | 4.5 (33.25)
  GGT, Year 10, Week 8, n=152 | 2.7 (28.57)
  GGT, Year 10, Week 16, n=143 | 4.5 (33.50)
  GGT, Year 10, Week 24, n=145 | 3.0 (31.51)
  GGT, Year 10, Week 32, n=142 | 4.2 (31.74)
  GGT, Year 10, Week 40, n=138 | 2.9 (31.64)
  GGT, Year 10, Week 48, n=135 | 5.9 (29.18)
  GGT, Year 11, Week 8, n=138 | 3.8 (33.68)
  GGT, Year 11, Week 16, n=128 | 4.8 (32.72)
  GGT, Year 11, Week 24, n=130 | 3.4 (26.42)
  GGT, Year 11, Week 32, n=125 | 2.8 (29.33)
  GGT, Year 11, Week 40, n=124 | 2.5 (28.02)
  GGT, Year 11, Week 48, n=108 | 7.0 (37.14)
  GGT, Year 12, Week 8, n=110 | 7.9 (37.22)
  GGT, Year 12, Week 16, n=97 | 2.3 (19.42)
  GGT, Year 12, Week 24, n=87 | 5.2 (32.26)
  GGT, Year 12, Week 32, n=84 | 4.4 (26.44)
  GGT, Year 12, Week 40, n=82 | 2.0 (27.54)
  GGT, Year 12, Week 48, n=72 | 1.6 (18.01)
  GGT, Year 13, Week 8, n=53 | 2.4 (18.65)
  GGT, Year 13, Week 16, n=42 | 8.8 (57.73)
  GGT, Year 13, Week 24, n=20 | 10.5 (40.97)
  GGT, Year 13, Week 32, n=7 | 6.1 (19.07)
  GGT, Year 13, Week 40, n=1 | 3.0 (NA) — No value as only one participant was analyzed.
  GGT, Exit, n=248 | 1.8 (53.15)
  GGT, 8-Week Follow-up, n=220 | 3.3 (24.91)
  GGT, 24-Week Follow-up , n=200 | 3.1 (55.20)
  LD, Year 1, Week 8, n=281 | -0.4 (23.41)
  LD, Year 1, Week 16, n=283 | -0.4 (29.97)
  LD, Year 1, Week 24, n=287 | -0.8 (31.43)
  LD, Year 1, Week 32, n=283 | -5.1 (26.19)
  LD, Year 1, Week 40, n=282 | -3.6 (27.97)
  LD, Year 1, Week 48, n=284 | -4.5 (28.66)
  LD, Year 2, Week 8, n=288 | -1.7 (28.26)
  LD, Year 2, Week 16, n=275 | -0.3 (30.16)
  LD, Year 2, Week 24, n=269 | -0.4 (29.91)
  LD, Year 2, Week 32, n=284 | -2.1 (34.05)
  LD, Year 2, Week 40, n=261 | -4.7 (29.69)
  LD, Year 2, Week 48, n=267 | -1.9 (29.81)
  LD, Year 3, Week 8, n=262 | -5.1 (29.71)
  LD, Year 3, Week 16, n=258 | -2.9 (31.27)
  LD, Year 3, Week 24, n=241 | 1.0 (32.12)
  LD, Year 3, Week 32, n=245 | 0.9 (36.26)
  LD, Year 3, Week 40, n=242 | 1.3 (34.00)
  LD, Year 3, Week 48, n=239 | 4.5 (35.46)
  LD, Year 4, Week 8, n=237 | 3.9 (36.59)
  LD, Year 4, Week 16, n=235 | 4.2 (38.16)
  LD, Year 4, Week 24, n=225 | 3.8 (38.59)
  LD, Year 4, Week 32, n=230 | 6.3 (37.05)
  LD, Year 4, Week 40, n=218 | 2.0 (37.75)
  LD, Year 4, Week 48, n=214 | 8.5 (39.80)
  LD, Year 5, Week 8, n=217 | 6.7 (39.42)
  LD, Year 5, Week 16, n=213 | 7.9 (42.94)
  LD, Year 5, Week 24, n=206 | 7.6 (40.54)
  LD, Year 5, Week 32, n=211 | 7.0 (36.84)
  LD, Year 5, Week 40, n=196 | 5.0 (40.29)
  LD, Year 5, Week 48, n=207 | 6.1 (37.15)
  LD, Year 6, Week 8, n=205 | 8.4 (36.82)
  LD, Year 6, Week 16, n=198 | 6.4 (36.98)
  LD, Year 6, Week 24, n=189 | 5.2 (38.41)
  LD, Year 6, Week 32, n=192 | 6.1 (34.07)
  LD, Year 6, Week 40, n=181 | 6.0 (39.60)
  LD, Year 6, Week 48, n=186 | 2.9 (39.20)
  LD, Year 7, Week 8, n=177 | 4.8 (37.46)
  LD, Year 7, Week 16, n=178 | 3.3 (37.02)
  LD, Year 7, Week 24, n=171 | 8.9 (39.81)
  LD, Year 7, Week 32, n=179 | 4.7 (40.87)
  LD, Year 7, Week 40, n=172 | 6.8 (39.49)
  LD, Year 7, Week 48, n=175 | 3.5 (37.36)
  LD, Year 8, Week 8, n=170 | 3.0 (36.88)
  LD, Year 8, Week 16, n=169 | 2.4 (36.06)
  LD, Year 8, Week 24, n=167 | 2.4 (37.06)
  LD, Year 8, Week 32, n=166 | 7.4 (36.86)
  LD, Year 8, Week 40, n=161 | 2.1 (35.04)
  LD, Year 8, Week 48, n=159 | 6.6 (39.01)
  LD, Year 9, Week 8, n=163 | 4.5 (36.82)
  LD, Year 9, Week 16, n=160 | 1.8 (36.46)
  LD, Year 9, Week 24, n=160 | 3.9 (35.65)
  LD, Year 9, Week 32, n=162 | 3.8 (37.69)
  LD, Year 9, Week 40, n=156 | 7.5 (39.97)
  LD, Year 9, Week 48, n=150 | 5.8 (39.05)
  LD, Year 10, Week 8, n=151 | 4.5 (42.02)
  LD, Year 10, Week 16, n=143 | 2.5 (34.44)
  LD, Year 10, Week 24, n=145 | 2.1 (38.80)
  LD, Year 10, Week 32, n=140 | 5.4 (41.37)
  LD, Year 10, Week 40, n=137 | 7.6 (37.07)
  LD, Year 10, Week 48, n=135 | 5.4 (37.12)
  LD, Year 11, Week 8, n=138 | 6.1 (45.90)
  LD, Year 11, Week 16, n=128 | 2.4 (38.69)
  LD, Year 11, Week 24, n=129 | 5.5 (42.10)
  LD, Year 11, Week 32, n=124 | 0.8 (44.21)
  LD, Year 11, Week 40, n=124 | 2.1 (41.89)
  LD, Year 11, Week 48, n=107 | 8.8 (40.94)
  LD, Year 12, Week 8, n=109 | 5.9 (51.46)
  LD, Year 12, Week 16, n=97 | 5.2 (45.81)
  LD, Year 12, Week 24, n=85 | 6.6 (47.18)
  LD, Year 12, Week 32, n=84 | 2.0 (47.59)
  LD, Year 12, Week 40, n=82 | 2.2 (47.71)
  LD, Year 12, Week 48, n=72 | 1.9 (61.71)
  LD, Year 13, Week 8, n=53 | -0.3 (31.81)
  LD, Year 13, Week 16, n=42 | -6.3 (38.99)
  LD, Year 13, Week 24, n=20 | 0.3 (51.57)
  LD, Year 13, Week 32, n=7 | -27.3 (63.45)
  LD, Year 13, Week 40, n=1 | 26.0 (NA) — No value as only one participant was analyzed.
  LD, Exit, n=248 | 6.4 (44.59)
  LD, 8-Week Follow-up, n=220 | 7.7 (51.21)
  LD, 24-Week Follow-up , n=200 | 6.5 (49.90)

14. Secondary Outcome: Percentage of Participants Achieving SLE Responder Index (SRI) Response at Indicated Time Points
Description: SRI response was assessed at Week 16, 32, and 48 during Year 1 to 12 and Week 16 and 32 during Year 13. Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. SRI response is defined as:>=4 point reduction from the Baseline in safety of estrogen in lupus national assessment (SELENA) SLE disease activity index (SLEDAI) score and no worsening (increase of <0.30 points from the Baseline) in Physician's Global Assessment (PGA), and no new British Isles Lupus Assessment Group (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with the Baseline at the time of assessment.
Time Frame: Approximately up to 13 years
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Percentage of participants
  Year 1 , Week 16, n=268: number analyzed (Participants) | 268
  Year 1 , Week 16, n=268 | 32.8
  Year 1 , Week 32, n=269: number analyzed (Participants) | 269
  Year 1 , Week 32, n=269 | 41.6
  Year 1 , Week 48, n=266: number analyzed (Participants) | 266
  Year 1 , Week 48, n=266 | 47.0
  Year 2 , Week 16, n=266: number analyzed (Participants) | 266
  Year 2 , Week 16, n=266 | 50.8
  Year 2, Week 32, n=262: number analyzed (Participants) | 262
  Year 2, Week 32, n=262 | 56.5
  Year 2, Week 48, n=251: number analyzed (Participants) | 251
  Year 2, Week 48, n=251 | 57.0
  Year 3, Week 16, n=245: number analyzed (Participants) | 245
  Year 3, Week 16, n=245 | 59.2
  Year 3, Week 32, n=235: number analyzed (Participants) | 235
  Year 3, Week 32, n=235 | 54.5
  Year 3, Week 48, n=225: number analyzed (Participants) | 225
  Year 3, Week 48, n=225 | 57.8
  Year 4, Week 16, n=225: number analyzed (Participants) | 225
  Year 4, Week 16, n=225 | 56.9
  Year 4, Week 32, n=212: number analyzed (Participants) | 212
  Year 4, Week 32, n=212 | 56.6
  Year 4, Week 48, n=206: number analyzed (Participants) | 206
  Year 4, Week 48, n=206 | 59.7
  Year 5, Week 16, n=198: number analyzed (Participants) | 198
  Year 5, Week 16, n=198 | 65.7
  Year 5, Week 32, n=194: number analyzed (Participants) | 194
  Year 5, Week 32, n=194 | 64.4
  Year 5, Week 48, n=192: number analyzed (Participants) | 192
  Year 5, Week 48, n=192 | 62.5
  Year 6, Week 16, n=182: number analyzed (Participants) | 182
  Year 6, Week 16, n=182 | 64.8
  Year 6, Week 32, n=181: number analyzed (Participants) | 181
  Year 6, Week 32, n=181 | 65.7
  Year 6, Week 48, n=176: number analyzed (Participants) | 176
  Year 6, Week 48, n=176 | 63.6
  Year 7, Week 16, n=169: number analyzed (Participants) | 169
  Year 7, Week 16, n=169 | 63.9
  Year 7, Week 32, n=173: number analyzed (Participants) | 173
  Year 7, Week 32, n=173 | 69.4
  Year 7, Week 48, n=162: number analyzed (Participants) | 162
  Year 7, Week 48, n=162 | 69.1
  Year 8, Week 16, n=161: number analyzed (Participants) | 161
  Year 8, Week 16, n=161 | 68.3
  Year 8, Week 32, n=158: number analyzed (Participants) | 158
  Year 8, Week 32, n=158 | 67.7
  Year 8, Week 48, n=149: number analyzed (Participants) | 149
  Year 8, Week 48, n=149 | 62.4
  Year 9, Week 16, n=151: number analyzed (Participants) | 151
  Year 9, Week 16, n=151 | 64.2
  Year 9, Week 32, n=148: number analyzed (Participants) | 148
  Year 9, Week 32, n=148 | 66.2
  Year 9, Week 48, n=142: number analyzed (Participants) | 142
  Year 9, Week 48, n=142 | 66.2
  Year 10, Week 16, n=141: number analyzed (Participants) | 141
  Year 10, Week 16, n=141 | 66.0
  Year 10, Week 32, n=135: number analyzed (Participants) | 135
  Year 10, Week 32, n=135 | 66.7
  Year 10, Week 48, n=126: number analyzed (Participants) | 126
  Year 10, Week 48, n=126 | 65.1
  Year 11, Week 16, n=125: number analyzed (Participants) | 125
  Year 11, Week 16, n=125 | 73.6
  Year 11, Week 32, n=120: number analyzed (Participants) | 120
  Year 11, Week 32, n=120 | 64.2
  Year 11, Week 48, n=109: number analyzed (Participants) | 109
  Year 11, Week 48, n=109 | 65.1
  Year 12, Week 16, n=100: number analyzed (Participants) | 100
  Year 12, Week 16, n=100 | 69.0
  Year 12, Week 32, n=90: number analyzed (Participants) | 90
  Year 12, Week 32, n=90 | 75.6
  Year 12, Week 48, n=71: number analyzed (Participants) | 71
  Year 12, Week 48, n=71 | 71.8
  Year 13, Week 16, n=42: number analyzed (Participants) | 42
  Year 13, Week 16, n=42 | 73.8
  Year 13, Week 32, n=7: number analyzed (Participants) | 7
  Year 13, Week 32, n=7 | 57.1

15. Secondary Outcome: Observed Anti-double Stranded DNA Levels in Participants Positive at Baseline at Indicated Time Points
Description: Anti-double stranded DNA levels in participants positive at Baseline were assessed at Baseline, Week 16, 32, and 48 during Year 1 to 11, Week 16 and 32 during Year 13, Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). The Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. For Year 1, Baseline included Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with belimumab in the parent study.
Time Frame: Approximately up to 13 years
Population: MITT Population. Only those participants positive at Baseline and available at the specified time points (represented by n=X in the category titles) were analyzed.
Measure: Median (Full Range); unit: International units (IU)/milliliter (mL)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 149
International units (IU)/milliliter (mL)
  Baseline, n=149 | 147.00 [31.0 to 418.0]
  Year 1 , Week 16, n=147 | 114.00 [6.0 to 418.0]
  Year 1 , Week 32, n=147 | 113.00 [5.0 to 349.0]
  Year 1 , Week 48, n=144 | 106.50 [5.0 to 464.0]
  Year 2 , Week 16, n=144 | 93.50 [3.0 to 328.0]
  Year 2, Week 32, n=143 | 85.00 [5.0 to 271.0]
  Year 2, Week 48, n=128 | 83.50 [5.0 to 271.0]
  Year 3, Week 16, n=134 | 83.50 [5.0 to 271.0]
  Year 3, Week 32, n=127 | 76.00 [5.0 to 271.0]
  Year 3, Week 48, n=125 | 73.00 [5.0 to 271.0]
  Year 4, Week 16, n=124 | 80.00 [5.0 to 271.0]
  Year 4, Week 32, n=120 | 72.00 [5.0 to 271.0]
  Year 4, Week 48, n=116 | 66.50 [5.0 to 271.0]
  Year 5, Week 16, n=112 | 54.00 [5.0 to 271.0]
  Year 5, Week 32, n=111 | 61.00 [5.0 to 271.0]
  Year 5, Week 48, n=108 | 49.50 [5.0 to 271.0]
  Year 6, Week 16, n=105 | 41.00 [5.0 to 271.0]
  Year 6, Week 32, n=101 | 44.00 [5.0 to 271.0]
  Year 6, Week 48, n=99 | 36.00 [5.0 to 271.0]
  Year 7, Week 16, n=89 | 41.00 [5.0 to 271.0]
  Year 7, Week 32, n=94 | 36.50 [5.0 to 271.0]
  Year 7, Week 48, n=89 | 38.00 [5.0 to 586.0]
  Year 8, Week 16, n=87 | 30.00 [5.0 to 468.0]
  Year 8, Week 32, n=89 | 43.00 [5.0 to 890.0]
  Year 8, Week 48, n=80 | 27.50 [5.0 to 1826.0]
  Year 9, Week 16, n=85 | 32.00 [5.0 to 745.0]
  Year 9, Week 32, n=83 | 20.00 [5.0 to 2120.0]
  Year 9, Week 48, n=77 | 16.00 [5.0 to 423.0]
  Year 10, Week 16, n=77 | 18.00 [5.0 to 593.0]
  Year 10, Week 32, n=75 | 22.00 [5.0 to 607.0]
  Year 10, Week 48, n=71 | 18.00 [5.0 to 500.0]
  Year 11, Week 16, n=67 | 17.00 [5.0 to 445.0]
  Year 11, Week 32, n=66 | 15.00 [5.0 to 611.0]
  Year 11, Week 48, n=63 | 11.00 [5.0 to 546.0]
  Year 12, Week 16, n=54 | 11.00 [5.0 to 330.0]
  Year 12, Week 32, n=47 | 8.00 [5.0 to 219.0]
  Year 12, Week 48, n=39 | 14.00 [5.0 to 402.0]
  Year 13, Week 16, n=20 | 13.50 [5.0 to 549.0]
  Year 13, Week 32, n=3 | 7.00 [5.0 to 8.0]
  Exit, n=124 | 31.00 [5.0 to 1073.0]

16. Secondary Outcome: Median Percent Change From Baseline in Anti-double Stranded DNA in Participants Positive at Baseline at Indicated Time Points
Description: Anti-double stranded DNA levels for participants positive at Baseline were assessed at Baseline, Week 16, 32, and 48 during Year 1 to 11, Week 16 and 32 during Year 13, Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). The Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. For Year 1, Baseline included Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with belimumab in the parent study. Percent change from Baseline is defined as the percentage of the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 15
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 149
Percent change
  Year 1 , Week 16, n=147 | -16.26 [-87.5 to 252.1]
  Year 1 , Week 32, n=147 | -25.57 [-93.8 to 168.8]
  Year 1 , Week 48, n=144 | -30.17 [-93.4 to 177.1]
  Year 2 , Week 16, n=144 | -30.26 [-96.3 to 344.3]
  Year 2, Week 32, n=143 | -31.25 [-90.0 to 224.6]
  Year 2, Week 48, n=128 | -41.63 [-93.8 to 133.6]
  Year 3, Week 16, n=134 | -41.10 [-94.1 to 232.4]
  Year 3, Week 32, n=127 | -44.44 [-94.8 to 208.3]
  Year 3, Week 48, n=125 | -45.29 [-95.4 to 133.6]
  Year 4, Week 16, n=124 | -47.33 [-95.2 to 243.0]
  Year 4, Week 32, n=120 | -48.53 [-95.4 to 243.0]
  Year 4, Week 48, n=116 | -48.45 [-96.7 to 243.0]
  Year 5, Week 16, n=112 | -53.97 [-96.1 to 243.0]
  Year 5, Week 32, n=111 | -47.27 [-96.7 to 411.3]
  Year 5, Week 48, n=108 | -57.76 [-96.7 to 453.1]
  Year 6, Week 16, n=105 | -60.00 [-97.4 to 361.2]
  Year 6, Week 32, n=101 | -65.38 [-96.8 to 411.3]
  Year 6, Week 48, n=99 | -66.42 [-97.7 to 243.0]
  Year 7, Week 16, n=89 | -64.14 [-97.2 to 243.0]
  Year 7, Week 32, n=94 | -68.93 [-96.7 to 243.0]
  Year 7, Week 48, n=89 | -68.63 [-98.1 to 182.3]
  Year 8, Week 16, n=87 | -73.77 [-98.1 to 111.7]
  Year 8, Week 32, n=89 | -71.02 [-98.3 to 249.0]
  Year 8, Week 48, n=80 | -76.62 [-98.1 to 1326.6]
  Year 9, Week 16, n=85 | -75.00 [-97.4 to 1452.1]
  Year 9, Week 32, n=83 | -80.13 [-98.1 to 4316.7]
  Year 9, Week 48, n=77 | -81.38 [-97.7 to 152.1]
  Year 10, Week 16, n=77 | -81.25 [-97.4 to 363.3]
  Year 10, Week 32, n=75 | -78.11 [-98.1 to 175.0]
  Year 10, Week 48, n=71 | -81.13 [-98.4 to 124.2]
  Year 11, Week 16, n=67 | -82.86 [-98.4 to 99.6]
  Year 11, Week 32, n=66 | -85.39 [-97.7 to 377.3]
  Year 11, Week 48, n=63 | -85.29 [-98.4 to 326.6]
  Year 12, Week 16, n=54 | -85.39 [-97.8 to 132.8]
  Year 12, Week 32, n=47 | -88.52 [-98.4 to 71.1]
  Year 12, Week 48, n=39 | -87.76 [-98.4 to 135.2]
  Year 13, Week 16, n=20 | -86.87 [-98.4 to 192.0]
  Year 13, Week 32, n=3 | -91.49 [-98.4 to -86.8]
  Exit, n=124 | -75.68 [-98.4 to 257.7]

17. Secondary Outcome: Observed Complement C3 and C4 Levels in Participants Low at Baseline at Indicated Time Points
Description: Complement C3 and C4 levels were assessed in participants low at Baseline at Baseline, Week 16, 32, and 48 during Year 1 to 12, Week 16 and 32 during Year 13, and Exit visit. The Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. For Year 1, Baseline included Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with belimumab in the parent study.
Time Frame: Approximately up to 13 years
Population: as for outcome 15
Measure: Median (Full Range); unit: grams per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 88
grams per liter
  C3, Baseline, n=88 | 0.77 [0.4 to 0.9]
  C3, Year 1, Week 16, n=86 | 0.81 [0.5 to 1.3]
  C3, Year 1, Week 32, n=88 | 0.81 [0.2 to 1.5]
  C3, Year 1, Week 48, n=86 | 0.82 [0.5 to 1.3]
  C3, Year 2, Week 16, n=83 | 0.82 [0.6 to 1.4]
  C3, Year 2, Week 32, n=83 | 0.84 [0.5 to 1.4]
  C3, Year 2, Week 48, n=76 | 0.88 [0.5 to 1.3]
  C3, Year 3, Week 16, n=75 | 0.88 [0.3 to 1.3]
  C3, Year 3, Week 32, n=75 | 0.90 [0.5 to 1.4]
  C3, Year 3, Week 48, n=73 | 0.90 [0.3 to 1.5]
  C3, Year 4, Week 16, n=74 | 0.93 [0.5 to 1.4]
  C3, Year 4, Week 32, n=72 | 0.96 [0.4 to 1.3]
  C3, Year 4, Week 48, n=67 | 0.93 [0.5 to 1.4]
  C3, Year 5, Week 16, n=65 | 0.94 [0.4 to 1.5]
  C3, Year 5, Week 32, n=65 | 0.97 [0.4 to 1.5]
  C3, Year 5, Week 48, n=65 | 1.01 [0.4 to 1.5]
  C3, Year 6, Week 16, n=61 | 1.02 [0.4 to 1.4]
  C3, Year 6, Week 32, n=59 | 1.03 [0.5 to 1.5]
  C3, Year 6, Week 48, n=57 | 1.00 [0.4 to 1.5]
  C3, Year 7, Week 16, n=50 | 0.94 [0.5 to 1.6]
  C3, Year 7, Week 32, n=54 | 0.99 [0.2 to 1.5]
  C3, Year 7, Week 48, n=52 | 0.98 [0.3 to 1.7]
  C3, Year 8, Week 16, n=46 | 0.98 [0.3 to 1.6]
  C3, Year 8, Week 32, n=48 | 1.01 [0.5 to 1.6]
  C3, Year 8, Week 48, n=45 | 1.01 [0.6 to 2.0]
  C3, Year 9, Week 16, n=49 | 1.02 [0.5 to 2.1]
  C3, Year 9, Week 32, n=46 | 0.95 [0.5 to 2.0]
  C3, Year 9, Week 48, n=47 | 0.98 [0.5 to 1.9]
  C3, Year 10, Week 16, n=43 | 0.91 [0.4 to 1.6]
  C3, Year 10, Week 32, n=45 | 0.99 [0.3 to 2.0]
  C3, Year 10, Week 48, n=44 | 0.90 [0.5 to 1.9]
  C3, Year 11, Week 16, n=43 | 0.97 [0.4 to 1.7]
  C3, Year 11, Week 32, n=42 | 0.99 [0.6 to 1.9]
  C3, Year 11, Week 48, n=37 | 0.88 [0.5 to 1.7]
  C3, Year 12, Week 16, n=31 | 0.92 [0.5 to 1.9]
  C3, Year 12, Week 32, n=28 | 0.94 [0.5 to 1.7]
  C3, Year 12, Week 48, n=28 | 0.84 [0.4 to 1.6]
  C3, Year 13, Week 16, n=12 | 0.95 [0.6 to 1.6]
  C3, Year 13, Week 32, n=2 | 0.99 [0.8 to 1.2]
  C3, Exit, n=74 | 0.98 [0.4 to 1.6]
  C4, Baseline, n=116 | 0.10 [0.0 to 0.2]
  C4, Year 1, Week 16, n=112 | 0.12 [0.0 to 0.4]
  C4, Year 1, Week 32, n=113 | 0.13 [0.0 to 0.3]
  C4, Year 1, Week 48, n=112 | 0.14 [0.0 to 0.3]
  C4, Year 2, Week 16, n=110 | 0.15 [0.0 to 0.3]
  C4, Year 2, Week 32, n=110 | 0.15 [0.0 to 0.3]
  C4, Year 2, Week 48, n=103 | 0.17 [0.0 to 0.5]
  C4, Year 3, Week 16, n=101 | 0.16 [0.0 to 0.4]
  C4, Year 3, Week 32, n=100 | 0.17 [0.0 to 0.5]
  C4, Year 3, Week 48, n=97 | 0.17 [0.0 to 0.5]
  C4, Year 4, Week 16, n=97 | 0.17 [0.0 to 0.4]
  C4, Year 4, Week 32, n=93 | 0.17 [0.0 to 0.4]
  C4, Year 4, Week 48, n=90 | 0.18 [0.0 to 0.4]
  C4, Year 5, Week 16, n=83 | 0.18 [0.0 to 0.4]
  C4, Year 5, Week 32, n=81 | 0.19 [0.0 to 0.4]
  C4, Year 5, Week 48, n=81 | 0.19 [0.0 to 0.4]
  C4, Year 6, Week 16, n=78 | 0.20 [0.0 to 0.4]
  C4, Year 6, Week 32, n=74 | 0.19 [0.0 to 0.4]
  C4, Year 6, Week 48, n=71 | 0.19 [0.0 to 0.4]
  C4, Year 7, Week 16, n=66 | 0.19 [0.0 to 0.4]
  C4, Year 7, Week 32, n=67 | 0.20 [0.0 to 0.4]
  C4, Year 7, Week 48, n=65 | 0.20 [0.0 to 0.5]
  C4, Year 8, Week 16, n=61 | 0.20 [0.0 to 0.4]
  C4, Year 8, Week 32, n=62 | 0.20 [0.0 to 0.4]
  C4, Year 8, Week 48, n=56 | 0.20 [0.1 to 0.6]
  C4, Year 9, Week 16, n=62 | 0.20 [0.0 to 0.5]
  C4, Year 9, Week 32, n=59 | 0.19 [0.0 to 0.4]
  C4, Year 9, Week 48, n=55 | 0.19 [0.0 to 0.4]
  C4, Year 10, Week 16, n=54 | 0.2 [0.1 to 0.4]
  C4, Year 10, Week 32, n=52 | 0.19 [0.0 to 0.5]
  C4, Year 10, Week 48, n=51 | 0.18 [0.0 to 0.4]
  C4, Year 11, Week 16, n=50 | 0.2 [0.1 to 0.4]
  C4, Year 11, Week 32, n=48 | 0.20 [0.1 to 0.4]
  C4, Year 11, Week 48, n=44 | 0.21 [0.1 to 0.4]
  C4, Year 12, Week 16, n=41 | 0.18 [0.1 to 0.4]
  C4, Year 12, Week 32, n=37 | 0.21 [0.1 to 0.4]
  C4, Year 12, Week 48, n=31 | 0.18 [0.1 to 0.3]
  C4, Year 13, Week 16, n=16 | 0.21 [0.1 to 0.4]
  C4, Year 13, Week 32, n=3 | 0.29 [0.2 to 0.4]
  C4, Exit, n=93 | 0.18 [0.0 to 0.4]

18. Secondary Outcome: Median Percent Change From Baseline in Complement C3 and C4 Levels in Participants Low at Baseline at Indicated Time Points
Description: Complement C3 and C4 levels were assessed in participants low at Baseline at Baseline, Week 16, 32, and 48 during Year 1 to 12, Week 16 and 32 during Year 13, and Exit visit. The Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. For Year 1, Baseline included Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with belimumab in the parent study. Percent change from Baseline is defined as the percentage of the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 15
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 88
Percent change
  C3, Year 1, Week 16, n=86 | 8.87 [-32.1 to 72.1]
  C3, Year 1, Week 32, n=88 | 8.43 [-68.0 to 68.5]
  C3, Year 1, Week 48, n=86 | 11.71 [-33.3 to 56.5]
  C3, Year 2, Week 16, n=83 | 13.10 [-29.5 to 83.8]
  C3, Year 2, Week 32, n=83 | 13.21 [-19.5 to 135.3]
  C3, Year 2, Week 48, n=76 | 17.16 [-25.0 to 74.6]
  C3, Year 3, Week 16, n=75 | 15.48 [-50.8 to 129.4]
  C3, Year 3, Week 32, n=75 | 19.05 [-42.4 to 176.0]
  C3, Year 3, Week 48, n=73 | 16.46 [-61.7 to 182.0]
  C3, Year 4, Week 16, n=74 | 22.51 [-34.2 to 178.0]
  C3, Year 4, Week 32, n=72 | 30.41 [-56.8 to 158.0]
  C3, Year 4, Week 48, n=67 | 26.58 [-34.1 to 148.0]
  C3, Year 5, Week 16, n=65 | 27.38 [-47.7 to 156.0]
  C3, Year 5, Week 32, n=65 | 23.17 [-39.5 to 148.0]
  C3, Year 5, Week 48, n=65 | 35.96 [-26.2 to 129.4]
  C3, Year 6, Week 16, n=61 | 29.41 [-20.8 to 158.0]
  C3, Year 6, Week 32, n=59 | 31.03 [-21.7 to 138.0]
  C3, Year 6, Week 48, n=57 | 28.24 [-36.7 to 151.0]
  C3, Year 7, Week 16, n=50 | 20.95 [-32.5 to 149.0]
  C3, Year 7, Week 32, n=54 | 29.25 [-63.8 to 168.0]
  C3, Year 7, Week 48, n=52 | 39.88 [-51.7 to 186.0]
  C3, Year 8, Week 16, n=46 | 28.35 [-62.5 to 167.3]
  C3, Year 8, Week 32, n=48 | 30.88 [-34.2 to 138.8]
  C3, Year 8, Week 48, n=45 | 32.88 [-34.5 to 200.0]
  C3, Year 9, Week 16, n=49 | 36.99 [-45.9 to 208.8]
  C3, Year 9, Week 32, n=46 | 21.76 [-26.1 to 186.8]
  C3, Year 9, Week 48, n=47 | 23.29 [-34.1 to 180.0]
  C3, Year 10, Week 16, n=43 | 22.35 [-35.6 to 206.0]
  C3, Year 10, Week 32, n=45 | 23.81 [-60.7 to 186.8]
  C3, Year 10, Week 48, n=44 | 26.90 [-38.6 to 172.1]
  C3, Year 11, Week 16, n=43 | 26.97 [-48.5 to 146.0]
  C3, Year 11, Week 32, n=42 | 30.36 [-36.4 to 148.7]
  C3, Year 11, Week 48, n=37 | 20.78 [-39.0 to 149.3]
  C3, Year 12, Week 16, n=31 | 15.58 [-43.2 to 181.2]
  C3, Year 12, Week 32, n=28 | 26.39 [-39.5 to 123.7]
  C3, Year 12, Week 48, n=28 | 14.1 [-58.0 to 114.5]
  C3, Year 13, Week 16, n=12 | 35.33 [-8.3 to 97.2]
  C3, Year 13, Week 32, n=2 | 22.04 [9.6 to 34.5]
  C3, Exit, n=74 | 29.19 [-48.8 to 152.6]
  C4, Year 1, Week 16, n=112 | 25.00 [-57.1 to 200.0]
  C4, Year 1, Week 32, n=113 | 33.33 [-70.0 to 180.0]
  C4, Year 1, Week 48, n=112 | 34.52 [-60.0 to 183.3]
  C4, Year 2, Week 16, n=110 | 50.00 [-70.0 to 300.0]
  C4, Year 2, Week 32, n=110 | 53.33 [-25.0 to 400.0]
  C4, Year 2, Week 48, n=103 | 53.85 [-12.5 to 308.3]
  C4, Year 3, Week 16, n=101 | 53.33 [-33.3 to 275.0]
  C4, Year 3, Week 32, n=100 | 63.39 [-58.3 to 400.0]
  C4, Year 3, Week 48, n=97 | 53.33 [-66.7 to 422.2]
  C4, Year 4, Week 16, n=97 | 70.00 [-70.0 to 400.0]
  C4, Year 4, Week 32, n=93 | 69.23 [-50.0 to 350.0]
  C4, Year 4, Week 48, n=90 | 66.67 [-37.5 to 420.0]
  C4, Year 5, Week 16, n=83 | 71.43 [-33.3 to 500.0]
  C4, Year 5, Week 32, n=81 | 66.67 [-33.3 to 425.0]
  C4, Year 5, Week 48, n=81 | 80.00 [-66.7 to 460.0]
  C4, Year 6, Week 16, n=78 | 70.33 [-12.5 to 380.0]
  C4, Year 6, Week 32, n=74 | 85.71 [-12.5 to 400.0]
  C4, Year 6, Week 48, n=71 | 100.0 [-25.0 to 450.0]
  C4, Year 7, Week 16, n=66 | 79.29 [-13.3 to 350.0]
  C4, Year 7, Week 32, n=67 | 85.71 [-25.0 to 440.0]
  C4, Year 7, Week 48, n=65 | 100.0 [-50.0 to 377.8]
  C4, Year 8, Week 16, n=61 | 90.00 [-15.4 to 433.3]
  C4, Year 8, Week 32, n=62 | 81.67 [-18.2 to 575.5]
  C4, Year 8, Week 48, n=56 | 76.36 [-8.3 to 866.7]
  C4, Year 9, Week 16, n=62 | 87.86 [-57.1 to 566.7]
  C4, Year 9, Week 32, n=59 | 72.73 [-33.3 to 533.3]
  C4, Year 9, Week 48, n=55 | 71.43 [-42.9 to 566.7]
  C4, Year 10, Week 16, n=54 | 81.82 [-33.3 to 625.0]
  C4, Year 10, Week 32, n=52 | 84.52 [-57.1 to 575.0]
  C4, Year 10, Week 48, n=51 | 73.33 [-57.1 to 575.0]
  C4, Year 11, Week 16, n=50 | 75.71 [-27.3 to 500.0]
  C4, Year 11, Week 32, n=48 | 81.67 [-20.0 to 475.0]
  C4, Year 11, Week 48, n=44 | 103.33 [-33.3 to 650.0]
  C4, Year 12, Week 16, n=41 | 75.0 [-20.0 to 525.0]
  C4, Year 12, Week 32, n=37 | 100.0 [-23.1 to 340.0]
  C4, Year 12, Week 48, n=31 | 80.0 [-18.2 to 475.0]
  C4, Year 13, Week 16, n=16 | 135.0 [0.0 to 400.0]
  C4, Year 13, Week 32, n=3 | 190.0 [33.3 to 258.3]
  C4, Exit, n=93 | 78.57 [-57.1 to 575.0]

19. Secondary Outcome: Percentage of Participants With Daily Prednisone Dose Reduction at Indicated Time Points
Description: Daily prednisone dose reduction was assessed at Baseline, Week 8, 16, 24, 32, 40, and 48 during Year 1 to 12 and Week 8, 16, 24, 32, and 40 during Year 13. Percentage of participants with daily prednisone dose reduced to <=7.5 mg/day from >7.5 mg/kg at the Baseline are summarized. Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study.
Time Frame: Approximately up to 13 years
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 92
Percentage of participants
  Year 1, Week 8, n=91 | 0
  Year 1, Week 16, n=90 | 5.6
  Year 1, Week 24, n=91 | 19.8
  Year 1, Week 32, n=91 | 19.8
  Year 1, Week 40, n=87 | 23.0
  Year 1, Week 48, n=88 | 27.3
  Year 2, Week 8, n=90 | 28.9
  Year 2, Week 16, n=89 | 31.5
  Year 2, Week 24, n=90 | 28.9
  Year 2, Week 32, n=88 | 34.1
  Year 2, Week 40, n=84 | 35.7
  Year 2, Week 48, n=83 | 34.9
  Year 3, Week 8, n=81 | 35.8
  Year 3, Week 16, n=81 | 34.6
  Year 3, Week 24, n=73 | 34.2
  Year 3, Week 32, n=77 | 36.4
  Year 3, Week 40, n=78 | 33.3
  Year 3, Week 48, n=75 | 30.7
  Year 4, Week 8, n=72 | 40.3
  Year 4, Week 16, n=74 | 41.9
  Year 4, Week 24, n=71 | 45.1
  Year 4, Week 32, n=69 | 37.7
  Year 4, Week 40, n=67 | 37.3
  Year 4, Week 48, n=68 | 38.2
  Year 5, Week 8, n=67 | 41.8
  Year 5, Week 16, n=63 | 42.9
  Year 5, Week 24, n=64 | 45.3
  Year 5, Week 32, n=65 | 38.5
  Year 5, Week 40, n=58 | 48.3
  Year 5, Week 48, n=60 | 41.7
  Year 6, Week 8, n=61 | 44.3
  Year 6, Week 16, n=57 | 43.9
  Year 6, Week 24, n=58 | 48.3
  Year 6, Week 32, n=59 | 44.1
  Year 6, Week 40, n=55 | 41.8
  Year 6, Week 48, n=55 | 38.2
  Year 7, Week 8, n=52 | 46.2
  Year 7, Week 16, n=51 | 39.2
  Year 7, Week 24, n=51 | 41.2
  Year 7, Week 32, n=51 | 39.2
  Year 7, Week 40, n=51 | 39.2
  Year 7, Week 48, n=51 | 39.2
  Year 8, Week 8, n=50 | 40.0
  Year 8, Week 16, n=49 | 38.8
  Year 8, Week 24, n=50 | 38.0
  Year 8, Week 32, n=49 | 36.7
  Year 8, Week 40, n=49 | 38.8
  Year 8, Week 48, n=48 | 41.7
  Year 9, Week 8, n=48 | 39.6
  Year 9, Week 16, n=49 | 38.8
  Year 9, Week 24, n=49 | 38.8
  Year 9, Week 32, n=48 | 39.6
  Year 9, Week 40, n=48 | 35.4
  Year 9, Week 48, n=45 | 37.8
  Year 10, Week 8, n=46 | 37.0
  Year 10, Week 16, n=43 | 39.5
  Year 10, Week 24, n=44 | 31.8
  Year 10, Week 32, n=44 | 31.8
  Year 10, Week 40, n=43 | 34.9
  Year 10, Week 48, n=43 | 32.6
  Year 11, Week 8, n=44 | 36.4
  Year 11, Week 16, n=41 | 34.1
  Year 11, Week 24, n=40 | 32.5
  Year 11, Week 32, n=39 | 35.9
  Year 11, Week 40, n=40 | 40.0
  Year 11, Week 48, n=35 | 34.3
  Year 12, Week 8, n=35 | 34.3
  Year 12, Week 16, n=32 | 31.3
  Year 12, Week 24, n=29 | 34.5
  Year 12, Week 32, n=30 | 40.0
  Year 12, Week 40, n=30 | 46.7
  Year 12, Week 48, n=26 | 53.8
  Year 13, Week 8, n=19 | 47.4
  Year 13, Week 16, n=13 | 38.5
  Year 13, Week 24, n=6 | 50.0
  Year 13, Week 32, n=2 | 50.0
  Year 13, Week 40, n=1 | 0.0

20. Secondary Outcome: Absolute Serum Immunoglobulin G Values at Indicated Time Points
Description: Serum immunoglobulin G values were assessed at Baseline, Week 8, 16, 24, 32, 40, and 48 during Year 1 to 12 and Week 8, 16, 24, 32, and 40 during Year 13, Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. For Year 1, Baseline included Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with belimumab in the parent study.
Time Frame: Approximately up to 13 years
Population: as for outcome 4
Measure: Median (Full Range); unit: grams per liter
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
grams per liter
  Baseline, n=293 | 12.90 [3.3 to 39.5]
  Year 1, Week 8, n=288 | 12.10 [3.4 to 38.1]
  Year 1, Week 16, n=292 | 11.70 [3.3 to 34.3]
  Year 1, Week 24, n=293 | 11.60 [3.6 to 48.5]
  Year 1, Week 32, n=291 | 11.50 [3.8 to 32.6]
  Year 1, Week 40, n=288 | 11.40 [3.5 to 34.6]
  Year 1, Week 48, n=289 | 11.50 [3.5 to 33.8]
  Year 2, Week 8, n=286 | 11.20 [3.8 to 42.0]
  Year 2, Week 16, n=284 | 11.30 [3.2 to 41.7]
  Year 2, Week 24, n=288 | 11.55 [3.4 to 35.6]
  Year 2, Week 32, n=284 | 11.40 [3.2 to 32.2]
  Year 2, Week 40, n=269 | 11.30 [4.0 to 23.8]
  Year 2, Week 48, n=269 | 11.30 [3.1 to 24.5]
  Year 3, Week 8, n=265 | 11.40 [2.8 to 24.9]
  Year 3, Week 16, n=260 | 11.45 [3.2 to 27.2]
  Year 3, Week 24, n=244 | 11.15 [3.5 to 30.9]
  Year 3, Week 32, n=250 | 11.40 [3.2 to 27.0]
  Year 3, Week 40, n=246 | 11.70 [2.8 to 25.8]
  Year 3, Week 48, n=244 | 11.70 [3.3 to 28.3]
  Year 4, Week 8, n=240 | 11.50 [3.0 to 26.9]
  Year 4, Week 16, n=240 | 11.60 [3.0 to 28.5]
  Year 4, Week 24, n=228 | 11.35 [3.0 to 26.3]
  Year 4, Week 32, n=233 | 11.20 [3.0 to 24.0]
  Year 4, Week 40, n=220 | 11.40 [3.0 to 24.6]
  Year 4, Week 48, n=222 | 11.35 [3.0 to 26.8]
  Year 5, Week 8, n=218 | 11.45 [2.5 to 28.1]
  Year 5, Week 16, n=215 | 11.00 [2.8 to 26.7]
  Year 5, Week 24, n=212 | 10.80 [2.3 to 29.2]
  Year 5, Week 32, n=211 | 11.00 [2.8 to 27.1]
  Year 5, Week 40, n=199 | 11.10 [2.6 to 31.3]
  Year 5, Week 48, n=209 | 10.80 [2.7 to 28.2]
  Year 6, Week 8, n=207 | 10.80 [2.9 to 25.0]
  Year 6, Week 16, n=199 | 10.30 [2.7 to 23.6]
  Year 6, Week 24, n=192 | 10.20 [2.7 to 26.7]
  Year 6, Week 32, n=197 | 10.30 [2.7 to 24.9]
  Year 6, Week 40, n=186 | 10.30 [2.4 to 24.4]
  Year 6, Week 48, n=188 | 9.78 [2.1 to 23.7]
  Year 7, Week 8, n=183 | 10.10 [2.2 to 19.5]
  Year 7, Week 16, n=182 | 10.15 [2.0 to 24.6]
  Year 7, Week 24, n=176 | 10.10 [2.1 to 26.3]
  Year 7, Week 32, n=182 | 9.98 [2.0 to 23.4]
  Year 7, Week 40, n=177 | 9.85 [1.7 to 23.2]
  Year 7, Week 48, n=177 | 9.64 [1.7 to 22.6]
  Year 8, Week 8, n=173 | 9.64 [2.6 to 26.3]
  Year 8, Week 16, n=172 | 9.40 [2.0 to 22.7]
  Year 8, Week 24, n=169 | 9.67 [3.5 to 23.6]
  Year 8, Week 32, n=170 | 9.72 [2.9 to 18.8]
  Year 8, Week 40, n=163 | 9.41 [2.2 to 22.6]
  Year 8, Week 48, n=161 | 9.42 [2.3 to 22.4]
  Year 9, Week 8, n=167 | 9.41 [2.0 to 24.6]
  Year 9, Week 16, n=163 | 9.24 [4.0 to 21.7]
  Year 9, Week 24, n=163 | 9.39 [1.6 to 25.6]
  Year 9, Week 32, n=164 | 9.25 [2.0 to 24.2]
  Year 9, Week 40, n=159 | 9.06 [2.8 to 24.5]
  Year 9, Week 48, n=151 | 9.01 [3.0 to 23.9]
  Year 10, Week 8, n=153 | 9.02 [3.2 to 25.4]
  Year 10, Week 16, n=146 | 8.96 [2.7 to 27.3]
  Year 10, Week 24, n=146 | 8.98 [2.7 to 26.6]
  Year 10, Week 32, n=142 | 8.97 [2.4 to 23.1]
  Year 10, Week 40, n=138 | 9.09 [0.3 to 25.7]
  Year 10, Week 48, n=137 | 9.25 [2.6 to 26.3]
  Year 11, Week 8, n=139 | 9.54 [2.3 to 24.1]
  Year 11, Week 16, n=129 | 9.36 [2.5 to 15.3]
  Year 11, Week 24, n=131 | 9.53 [2.5 to 23.9]
  Year 11, Week 32, n=128 | 9.46 [2.5 to 23.0]
  Year 11, Week 40, n=124 | 9.68 [2.3 to 16.9]
  Year 11, Week 48, n=108 | 9.41 [2.6 to 16.8]
  Year 12, Week 8, n=111 | 8.92 [2.4 to 18.9]
  Year 12, Week 16, n=99 | 9.55 [2.2 to 17.0]
  Year 12, Week 24, n=87 | 9.33 [3.0 to 17.0]
  Year 12, Week 32, n=88 | 9.19 [2.1 to 17.1]
  Year 12, Week 40, n=84 | 8.79 [1.1 to 16.0]
  Year 12, Week 48, n=73 | 9.39 [3.2 to 15.6]
  Year 13, Week 8, n=53 | 9.62 [2.6 to 15.6]
  Year 13, Week 16, n=43 | 9.40 [2.6 to 16.4]
  Year 13, Week 24, n=20 | 9.77 [2.7 to 14.6]
  Year 13, Week 32, n=7 | 10.60 [6.8 to 11.2]
  Year 13, Week 40, n=1 | 11.50 [11.5 to 11.5]
  Exit, n=248 | 9.62 [1.8 to 23.5]
  8-Week follow-up, n=222 | 9.88 [1.8 to 30.3]
  24-Week follow-up, n=200 | 9.89 [1.3 to 29.1]

21. Secondary Outcome: Median Percent Change From Baseline in Immunoglobulin G at Indicated Time Points
Description: Serum immunoglobulin G values were assessed at Baseline, Week 8, 16, 24, 32, 40, and 48 during Year 1 to 12 and Week 8, 16, 24, 32, and 40 during Year 13, Exit visit and at follow-up (up to 8 weeks and 24 weeks post last infusion). Baseline is defined as the last available value prior to belimumab start date, for participants treated with placebo in the parent study and last pre-treatment value in the parent study for participants treated with belimumab in the parent study. For Year 1, Baseline included Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with belimumab in the parent study. Percent change from Baseline is defined as the percentage of the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and approximately up to 13 years
Population: as for outcome 4
Measure: Median (Full Range); unit: Percent change
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 296
Percent change
  Year 1, Week 8, n=285 | -6.09 [-46.4 to 116.5]
  Year 1, Week 16, n=289 | -7.69 [-47.7 to 82.4]
  Year 1, Week 24, n=290 | -8.78 [-69.6 to 165.0]
  Year 1, Week 32, n=288 | -8.84 [-47.6 to 41.6]
  Year 1, Week 40, n=285 | -10.32 [-44.4 to 32.2]
  Year 1, Week 48, n=286 | -9.34 [-46.3 to 33.8]
  Year 2, Week 8, n=283 | -11.40 [-46.0 to 43.3]
  Year 2, Week 16, n=281 | -10.76 [-50.8 to 47.3]
  Year 2, Week 24, n=285 | -11.19 [-51.7 to 66.3]
  Year 2, Week 32, n=281 | -11.40 [-52.9 to 54.0]
  Year 2, Week 40, n=266 | -10.29 [-49.9 to 93.0]
  Year 2, Week 48, n=267 | -10.54 [-58.0 to 103.0]
  Year 3, Week 8, n=263 | -10.28 [-50.4 to 62.9]
  Year 3, Week 16, n=258 | -9.92 [-53.3 to 52.9]
  Year 3, Week 24, n=242 | -9.77 [-56.6 to 60.3]
  Year 3, Week 32, n=248 | -8.93 [-52.0 to 45.7]
  Year 3, Week 40, n=244 | -8.04 [-54.9 to 46.3]
  Year 3, Week 48, n=242 | -10.40 [-52.3 to 45.0]
  Year 4, Week 8, n=238 | -10.70 [-55.3 to 46.2]
  Year 4, Week 16, n=238 | -10.77 [-54.9 to 145.1]
  Year 4, Week 24, n=226 | -11.73 [-72.6 to 37.5]
  Year 4, Week 32, n=231 | -10.99 [-53.5 to 48.2]
  Year 4, Week 40, n=218 | -10.47 [-54.9 to 47.7]
  Year 4, Week 48, n=220 | -11.69 [-59.2 to 57.3]
  Year 5, Week 8, n=216 | -13.20 [-61.8 to 45.6]
  Year 5, Week 16, n=213 | -14.62 [-64.2 to 45.5]
  Year 5, Week 24, n=210 | -14.61 [-59.9 to 89.6]
  Year 5, Week 32, n=209 | -13.24 [-54.5 to 29.7]
  Year 5, Week 40, n=197 | -15.97 [-54.8 to 42.4]
  Year 5, Week 48, n=207 | -15.47 [-57.0 to 38.6]
  Year 6, Week 8, n=205 | -17.13 [-73.7 to 40.9]
  Year 6, Week 16, n=197 | -18.16 [-75.0 to 32.6]
  Year 6, Week 24, n=190 | -18.67 [-64.5 to 36.4]
  Year 6, Week 32, n=195 | -19.83 [-65.0 to 42.4]
  Year 6, Week 40, n=184 | -19.84 [-61.9 to 26.6]
  Year 6, Week 48, n=186 | -22.36 [-79.4 to 39.2]
  Year 7, Week 8, n=181 | -21.26 [-64.4 to 29.4]
  Year 7, Week 16, n=180 | -21.22 [-68.7 to 45.0]
  Year 7, Week 24, n=175 | -21.39 [-71.5 to 39.9]
  Year 7, Week 32, n=180 | -22.03 [-71.8 to 45.5]
  Year 7, Week 40, n=175 | -22.31 [-71.7 to 24.5]
  Year 7, Week 48, n=175 | -22.20 [-69.0 to 25.4]
  Year 8, Week 8, n=171 | -24.44 [-74.3 to 46.9]
  Year 8, Week 16, n=170 | -25.51 [-76.3 to 26.6]
  Year 8, Week 24, n=167 | -24.91 [-76.6 to 32.4]
  Year 8, Week 32, n=168 | -24.48 [-76.3 to 59.9]
  Year 8, Week 40, n=161 | -25.50 [-76.8 to 87.8]
  Year 8, Week 48, n=159 | -24.58 [-76.0 to 78.9]
  Year 9, Week 8, n=165 | -25.41 [-77.8 to 100.4]
  Year 9, Week 16, n=161 | -25.44 [-80.6 to 23.7]
  Year 9, Week 24, n=161 | -27.23 [-78.8 to 155.8]
  Year 9, Week 32, n=162 | -26.92 [-79.6 to 168.3]
  Year 9, Week 40, n=157 | -27.63 [-78.9 to 164.8]
  Year 9, Week 48, n=149 | -26.48 [-79.4 to 184.4]
  Year 10, Week 8, n=151 | -28.65 [-78.7 to 125.4]
  Year 10, Week 16, n=144 | -28.45 [-74.0 to 130.8]
  Year 10, Week 24, n=144 | -28.78 [-73.8 to 211.3]
  Year 10, Week 32, n=140 | -27.98 [-74.4 to 161.2]
  Year 10, Week 40, n=137 | -28.57 [-97.6 to 98.6]
  Year 10, Week 48, n=136 | -28.86 [-72.9 to 164.8]
  Year 11, Week 8, n=138 | -28.91 [-71.9 to 61.7]
  Year 11, Week 16, n=128 | -29.34 [-69.8 to 48.1]
  Year 11, Week 24, n=130 | -29.64 [-68.0 to 180.9]
  Year 11, Week 32, n=127 | -29.50 [-67.6 to 72.5]
  Year 11, Week 40, n=123 | -27.58 [-68.9 to 202.3]
  Year 11, Week 48, n=107 | -27.13 [-67.0 to 200.5]
  Year 12, Week 8, n=110 | -29.27 [-68.5 to 220.2]
  Year 12, Week 16, n=98 | -30.30 [-70.5 to 14.4]
  Year 12, Week 24, n=86 | -30.25 [-66.0 to 28.5]
  Year 12, Week 32, n=87 | -30.72 [-72.6 to 12.2]
  Year 12, Week 40, n=83 | -32.96 [-96.4 to 9.9]
  Year 12, Week 48, n=72 | -31.72 [-65.5 to 13.2]
  Year 13, Week 8, n=52 | -32.23 [-65.7 to 5.3]
  Year 13, Week 16, n=42 | -31.91 [-67.0 to 3.5]
  Year 13, Week 24, n=20 | -28.18 [-54.9 to 5.3]
  Year 13, Week 32, n=7 | -33.06 [-58.2 to -7.8]
  Year 13, Week 40, n=1 | -12.9 [-12.9 to -12.9]
  Exit, n=245 | -23.37 [-72.0 to 200.5]
  8-Week follow-up, n=220 | -24.79 [-75.1 to 270.3]
  24-Week follow-up, n=198 | -22.09 [-77.9 to 245.3]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from Day 1 until follow-up (approximately up to 13 years).
Description: SAEs and non-serious AEs were collected in the MITT Population.
Arm/Group | Belimumab 10 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 182/296
Other Adverse Events (participants affected / at risk) | 293/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 10 mg/kg IV (N=296)
Pneumonia (Infections and infestations) | 20 (22)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 (19)
Non-cardiac chest pain (General disorders) | 12 (17)
Pyrexia (General disorders) | 11 (14)
Cellulitis (Infections and infestations) | 10 (13)
Abdominal pain (Gastrointestinal disorders) | 9 (12)
Cholelithiasis (Hepatobiliary disorders) | 8 (8)
Gastroenteritis viral (Infections and infestations) | 8 (11)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Bronchitis (Infections and infestations) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 6 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hypotension (Vascular disorders) | 6 (8)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 6 (9)
Appendicitis (Infections and infestations) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Hiatus hernia (Gastrointestinal disorders) | 5 (6)
Hypertension (Vascular disorders) | 5 (5)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 5 (6)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (5)
Lupus nephritis (Renal and urinary disorders) | 5 (6)
Syncope (Nervous system disorders) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Coronary artery disease (Cardiac disorders) | 4 (5)
Deep vein thrombosis (Vascular disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6)
Migraine (Nervous system disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (9)
Nausea (Gastrointestinal disorders) | 4 (8)
Pericarditis lupus (Cardiac disorders) | 4 (5)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (7)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Chest discomfort (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 3 (3)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Menometrorrhagia (Reproductive system and breast disorders) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (3)
Pyelonephritis (Infections and infestations) | 3 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3)
Sepsis (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2)
Arteriosclerosis (Vascular disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Asthenia (General disorders) | 2 (2)
Bacterial sepsis (Infections and infestations) | 2 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2)
Comminuted fracture (Injury, poisoning and procedural complications) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Endometriosis (Reproductive system and breast disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 2 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Lumbar radiculopathy (Nervous system disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (3)
Oesophageal candidiasis (Infections and infestations) | 2 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Pelvic adhesions (Reproductive system and breast disorders) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Renal failure (Renal and urinary disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Seizure (Nervous system disorders) | 2 (3)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Appendicitis noninfective (Gastrointestinal disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Benign intracranial hypertension (Nervous system disorders) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (3)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Central nervous system lupus (Nervous system disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (3)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colpocele (Reproductive system and breast disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (2)
Dyskinesia oesophageal (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Endometritis (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Haematocrit decreased (Investigations) | 1 (1)
Horner's syndrome (Nervous system disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1)
Idiopathic orbital inflammation (Eye disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Intervertebral discitis (Infections and infestations) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1)
Lupus enteritis (Gastrointestinal disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 1 (2)
Mouth swelling (Gastrointestinal disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Necrosis ischaemic (Vascular disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oesophageal mass (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (2)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (2)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Serositis (General disorders) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1)
Spinal epidural haemorrhage (Nervous system disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Stress at work (Social circumstances) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Surgical failure (General disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1)
Vulvar dysplasia (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
West Nile viral infection (Infections and infestations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 10 mg/kg IV (N=296)
Upper respiratory tract infection (Infections and infestations) | 217 (697)
Arthralgia (Musculoskeletal and connective tissue disorders) | 196 (703)
Headache (Nervous system disorders) | 155 (358)
Sinusitis (Infections and infestations) | 141 (409)
Nausea (Gastrointestinal disorders) | 140 (331)
Fatigue (General disorders) | 137 (277)
Urinary tract infection (Infections and infestations) | 137 (384)
Back pain (Musculoskeletal and connective tissue disorders) | 124 (225)
Cough (Respiratory, thoracic and mediastinal disorders) | 124 (246)
Diarrhoea (Gastrointestinal disorders) | 114 (231)
Bronchitis (Infections and infestations) | 110 (251)
Insomnia (Psychiatric disorders) | 110 (143)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 107 (204)
Arthritis (Musculoskeletal and connective tissue disorders) | 101 (211)
Rash (Skin and subcutaneous tissue disorders) | 98 (149)
Depression (Psychiatric disorders) | 94 (119)
Myalgia (Musculoskeletal and connective tissue disorders) | 92 (153)
Vomiting (Gastrointestinal disorders) | 86 (146)
Oedema peripheral (General disorders) | 83 (166)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 76 (121)
Hypertension (Vascular disorders) | 73 (105)
Pyrexia (General disorders) | 73 (147)
Seasonal allergy (Immune system disorders) | 73 (89)
Influenza (Infections and infestations) | 71 (96)
Nasopharyngitis (Infections and infestations) | 71 (135)
Procedural pain (Injury, poisoning and procedural complications) | 70 (117)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 68 (102)
Joint swelling (Musculoskeletal and connective tissue disorders) | 67 (113)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 67 (95)
Contusion (Injury, poisoning and procedural complications) | 66 (110)
Dizziness (Nervous system disorders) | 64 (101)
Viral upper respiratory tract infection (Infections and infestations) | 63 (115)
Migraine (Nervous system disorders) | 62 (123)
Anxiety (Psychiatric disorders) | 61 (74)
Mouth ulceration (Gastrointestinal disorders) | 60 (131)
Non-cardiac chest pain (General disorders) | 60 (88)
Gastroenteritis viral (Infections and infestations) | 59 (82)
Fall (Injury, poisoning and procedural complications) | 58 (116)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 58 (90)
Gastroenteritis (Infections and infestations) | 54 (86)
Alopecia (Skin and subcutaneous tissue disorders) | 53 (80)
Bursitis (Musculoskeletal and connective tissue disorders) | 53 (84)
Constipation (Gastrointestinal disorders) | 51 (59)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 51 (70)
Peripheral swelling (General disorders) | 49 (64)
Vulvovaginal mycotic infection (Infections and infestations) | 48 (99)
Chest X-ray (Investigations) | 47 (74)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 47 (61)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 47 (84)
Neck pain (Musculoskeletal and connective tissue disorders) | 46 (67)
Herpes zoster (Infections and infestations) | 45 (64)
Pain (General disorders) | 45 (57)
Abdominal pain (Gastrointestinal disorders) | 44 (62)
Tooth abscess (Infections and infestations) | 43 (52)
Anaemia (Blood and lymphatic system disorders) | 42 (50)
Oral candidiasis (Infections and infestations) | 42 (68)
Weight increased (Investigations) | 42 (61)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 40 (66)
Dyspepsia (Gastrointestinal disorders) | 39 (45)
Colonoscopy (Investigations) | 38 (41)
Hypoaesthesia (Nervous system disorders) | 38 (46)
Erythema (Skin and subcutaneous tissue disorders) | 37 (57)
Tendonitis (Musculoskeletal and connective tissue disorders) | 37 (56)
Hypokalaemia (Metabolism and nutrition disorders) | 36 (73)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 36 (52)
Ligament sprain (Injury, poisoning and procedural complications) | 35 (48)
Muscle strain (Injury, poisoning and procedural complications) | 35 (46)
Oral herpes (Infections and infestations) | 35 (68)
Paraesthesia (Nervous system disorders) | 35 (46)
Pruritus (Skin and subcutaneous tissue disorders) | 35 (49)
Weight decreased (Investigations) | 35 (39)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 34 (48)
Asthma (Respiratory, thoracic and mediastinal disorders) | 33 (80)
Dry eye (Eye disorders) | 33 (38)
Abdominal pain upper (Gastrointestinal disorders) | 32 (46)
Foot fracture (Injury, poisoning and procedural complications) | 32 (42)
Lymphadenopathy (Blood and lymphatic system disorders) | 32 (41)
Otitis media (Infections and infestations) | 32 (44)
Urticaria (Skin and subcutaneous tissue disorders) | 32 (56)
Dental caries (Gastrointestinal disorders) | 31 (42)
Pharyngitis (Infections and infestations) | 31 (39)
Pneumonia (Infections and infestations) | 31 (41)
Toothache (Gastrointestinal disorders) | 31 (36)
Vertigo (Ear and labyrinth disorders) | 31 (36)
Laceration (Injury, poisoning and procedural complications) | 30 (38)
Nuclear magnetic resonance imaging (Investigations) | 29 (39)
Proteinuria (Renal and urinary disorders) | 29 (42)
Arthropod bite (Injury, poisoning and procedural complications) | 28 (36)
Cellulitis (Infections and infestations) | 28 (37)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 28 (41)
Synovitis (Musculoskeletal and connective tissue disorders) | 28 (58)
Cataract (Eye disorders) | 27 (34)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 27 (40)
Leukopenia (Blood and lymphatic system disorders) | 27 (50)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 26 (27)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 26 (34)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 26 (33)
Tooth infection (Infections and infestations) | 26 (37)
X-ray limb (Investigations) | 26 (49)
Conjunctivitis (Infections and infestations) | 25 (39)
Ecchymosis (Skin and subcutaneous tissue disorders) | 25 (34)
Electrocardiogram (Investigations) | 25 (32)
Hypothyroidism (Endocrine disorders) | 25 (27)
Decreased appetite (Metabolism and nutrition disorders) | 24 (27)
Hyperlipidaemia (Metabolism and nutrition disorders) | 24 (25)
Osteopenia (Musculoskeletal and connective tissue disorders) | 24 (25)
Palpitations (Cardiac disorders) | 24 (27)
Rash erythematous (Skin and subcutaneous tissue disorders) | 24 (37)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 24 (42)
Tooth fracture (Injury, poisoning and procedural complications) | 24 (25)
Butterfly rash (Skin and subcutaneous tissue disorders) | 23 (31)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 23 (38)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 23 (24)
Bone densitometry (Investigations) | 22 (23)
Dry mouth (Gastrointestinal disorders) | 22 (24)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 22 (22)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 22 (37)
Sciatica (Nervous system disorders) | 22 (25)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 22 (31)
Upper respiratory tract infection bacterial (Infections and infestations) | 22 (31)
Abdominal discomfort (Gastrointestinal disorders) | 21 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (27)
Gastritis (Gastrointestinal disorders) | 21 (25)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 21 (28)
Rash pruritic (Skin and subcutaneous tissue disorders) | 21 (27)
Raynaud's phenomenon (Vascular disorders) | 21 (33)
Vitamin D deficiency (Metabolism and nutrition disorders) | 21 (22)
Chills (General disorders) | 20 (34)
Computerised tomogram (Investigations) | 20 (22)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 20 (47)
Dermatitis (Skin and subcutaneous tissue disorders) | 20 (28)
Ear pain (Ear and labyrinth disorders) | 20 (27)
Fungal skin infection (Infections and infestations) | 20 (30)
Haemorrhoids (Gastrointestinal disorders) | 20 (24)
Infusion site extravasation (General disorders) | 20 (25)
Mammogram (Investigations) | 20 (32)
Pharyngitis streptococcal (Infections and infestations) | 20 (25)
Rash macular (Skin and subcutaneous tissue disorders) | 20 (23)
Abdominal pain lower (Gastrointestinal disorders) | 19 (20)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 19 (25)
Eczema (Skin and subcutaneous tissue disorders) | 19 (25)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 (24)
Skin ulcer (Skin and subcutaneous tissue disorders) | 19 (24)
Trigger finger (Musculoskeletal and connective tissue disorders) | 19 (29)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 19 (24)
Creatinine renal clearance decreased (Investigations) | 18 (24)
Onychomycosis (Infections and infestations) | 18 (22)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (23)
Restless legs syndrome (Nervous system disorders) | 18 (19)
Sinus headache (Nervous system disorders) | 18 (29)
Skin abrasion (Injury, poisoning and procedural complications) | 18 (22)
X-ray of pelvis and hip (Investigations) | 18 (24)
Computerised tomogram abdomen (Investigations) | 17 (17)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 17 (19)
Dysphagia (Gastrointestinal disorders) | 17 (19)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 17 (20)
Night sweats (Skin and subcutaneous tissue disorders) | 17 (24)
Nuclear magnetic resonance imaging spinal (Investigations) | 17 (21)
Spinal X-ray (Investigations) | 17 (24)
Computerised tomogram head (Investigations) | 16 (22)
Costochondritis (Musculoskeletal and connective tissue disorders) | 16 (22)
Dysuria (Renal and urinary disorders) | 16 (18)
Flank pain (Musculoskeletal and connective tissue disorders) | 16 (21)
Haematuria (Renal and urinary disorders) | 16 (19)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (19)
Rash papular (Skin and subcutaneous tissue disorders) | 16 (19)
Skin infection (Infections and infestations) | 16 (18)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 16 (29)
Urinary tract infection bacterial (Infections and infestations) | 16 (28)
Viral infection (Infections and infestations) | 16 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (17)
Hiatus hernia (Gastrointestinal disorders) | 15 (17)
Neutropenia (Blood and lymphatic system disorders) | 15 (26)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 15 (16)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 15 (15)
Pollakiuria (Renal and urinary disorders) | 15 (16)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 15 (18)
Skin mass (Skin and subcutaneous tissue disorders) | 15 (24)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 15 (16)
Wound (Injury, poisoning and procedural complications) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.